

# SPARK 228PD201/NCT03318523

## Statistical Analysis Plan

Placebo-Controlled Period (Year 1)



Placebo-Controlled Period

V1.0

#### STATISTICAL ANALYSIS PLAN Placebo-Controlled Period

Product Studied: BIIB054 Protocol Number: 228PD201

A Multicenter, Randomized, Double-Blind, Placebo-Controlled Study, with an Active-Treatment Dose-Blinded Period, to Evaluate the Efficacy, Safety, Pharmacokinetics, and Pharmacodynamics of BIIB054 in Subjects with Parkinson's Disease

> Protocol Version: Version 8.0 Date of Protocol: 11 Aug 2020

Date of Statistical Analysis Plan: 23 Sep 2020, Final V1.0





#### **Table of Contents**

| L | IST OF ABBREVIATIONS | 5 |
|---|---|---|
| 1 | SCOPE OF WORK IN THE STATISTICAL ANAYSIS PLAN | 7 |
| 2 | DESCRIPTION OF OBJECTIVES AND ENDPOINTS | 7 |
| 3 | STUDY DESIGN | |
| | 3.1 STUDY OVERVIEW | |
| | 3.1.1 Year 1 (Placebo-Controlled Portion of the Study) | 12 |
| | 3.1.2 Years 2 Through 4 (Active-Treatment Dose-Blinded Portion of the Study) | 12 |
| | 3.2 STUDY SCHEMATIC | |
| | 3.3 SCHEDULE OF EVENTS | 15 |
| 4 | SAMPLE SIZE JUSTIFICATION | 15 |
| 5 | STATISTICAL ANALYSIS METHODS | 17 |
| | 5.1 GENERAL CONSIDERATIONS | 17 |
| | 5.1.1 End of Study (EOS) and End of Treatment (EOT) | |
| | 5.1.2 Analysis Population | |
| | 5.2 BACKGROUND CHARACTERISTICS | |
| | 5.2.1 Accounting of Subjects | |
| | 5.2.2 Demographics and Baseline Characteristics | |
| | 5.2.3 Concomitant Medications and Non-drug Therapies | |
| | 5.2.4 Protocol Deviations | |
| | 5.2.5 Study Drug Exposure and Study Drug Compliance | |
| | 5.3 EFFICACY ENDPOINTS | 21 |
| | 5.3.1 General Consideration | |
| | 5.3.2 MDS-UPDRS | |
| | 5.3.2.1 Primary efficacy endpoint | 22 |
| | 5.3.2.2 Secondary endpoints and additional MDS-UPDRS based endpoints | 23 |
| | 5.3.2.4 Early Parkinson's Regional Progression Score (EP-RPS) measure | |
| | 5.3.2.5 Time to start of PD medication, or an increase of MDS-UPDRS Part III total ≥ MCID (4.63), w | |
| | comes earlier | |
| | 5.3.2.6 Time to start of PD medication | |
| | 5.3.2.7 Time to disease progression and DCR (Disease Control Rate) | |
| | 5,3,2,9 Per-protocol analysis | |
| | 5.3.3 Other clinical efficacy endpoints | |
| | | 29 |
| | 5.3.5 Assessment of the Impact of Covid-19 on the clinical outcome analyses | |
| | 5.4 SAFETY ANALYSIS | |
| | 5.4.1 General Considerations | |
| | 5.4.2 Clinical Adverse Events | |
| | 5.4.3 Clinical Laboratory Data | |
| | 5.4.3.1 Quantitative laboratory analyses | |
| | 5.4.3.2 Qualitative laboratory analyses | |
| | 5.4.5 ECG Data | |
| | 5.4.6 Physical and Neurological Examination | |
| | 5.4.7 C-SSRS Data | |
| | 5.4.8 MRI Safety Data | |
| | 5.4.8 MKI Safety Data 5.5 PHARMACODYNAMIC -IMAGING ANALYSIS | |
| | 5.5.1 Type of imaging techniques and imaging outcomes | |
| | 5.5.1 1 pe of maging cominques and maging outcomes | , T I |



| | 5.5.2 | Analysis population | 41 |
|---|---|---|---|
| | 5.5.3 | Baseline value | |
| | 5.5.4 | Outlier of percent change from baseline | |
| | 5.5.5 | Analysis methods | |
| | 5.5.6 | Sensitivity analysis | |
| | 5.5.7 | Correlation analysis | |
| | | | 43 |
| | | | 43 |
| | | | 43 |
| | | | 43 |
| | | | 44 |
| | 5.7 | PHARMACOKINETICS ANALYSIS | 44 |
| | 5.7.1 | PK Concentration Profile | 45 |
| | 5.7.2 | Serum PK Parameters | 45 |
| | 5.8 | Immunogenicity Analysis | |
| | 5.8.1 | Analysis Methods for Immunogenicity Data | 45 |
| 6 | INTE | ERIM ANALYSIS | 46 |
| 7 | REF | ERENCES | 48 |
| 8 | APPI | ENDIX | 49 |
| | 8.1 | APPENDIX I: QUESTIONNAIRES | 49 |
| | | APPENDIX II: VISIT WINDOW MAPPING | |
| | | APPENDIX III: DESCRIPTION OF MCP-MOD METHOD | |
| | | APPENDIX IV: DEFINITION OF THE EARLY PARKINSON'S REGIONAL PROGRESSION SCOPE | |
| | | S) | |
| | | | 52 |
| | | | 52 |



Placebo-Controlled Period

#### List of Abbreviations

| O. CZ23 | Alpha expuelein |
|---|---|
| α-syn | Alpha-synuclein |
| ADA | anti dena antibodica |
| ADA | anti-drug antibodies |
| AT | a decomp accept |
| ALD | adverse event |
| ALP | alkaline phosphatase |
| ALT | alanine aminotransferase |
| ANCOVA | analysis of covariance |
| APTT | activated partial thromboplastin time |
| AST | aspartate aminotransferase |
| AUC | area under the curve |
| BL | baseline |
| BLQ | below the limit of quantification |
| BMI | body mass index |
| BPM | beats per minute |
| BRP-AUC | body region progression AUC |
| C <sub>max</sub> | observed maximum serum aducanumab concentration |
| C <sub>min</sub> | observed minimum serum aducanumab concentration |
| CI | confidence interval |
| CPP | Clinical Pharmacology and Pharmacometrics |
| C-SSRS | Columbia Suicide Severity Rating Scale |
| CTCAT | Common Toxicity Criteria for Adverse Events |
| CV | coefficient of variation |
| DaT | dopamine transporter |
| DaTscan <sup>TM</sup> | Ioflupane I123 radioligand for imaging of dopamine transporter |
| DBE | dose blinded extension |
| DBP | diastolic blood pressure |
| EC <sub>50</sub> | Concentration at 50% of maximum observed biologic effect |
| ECG | electrocardiogram |
| eCRF | electronic case report form |
| EOS | end of study |
| EOT | end of treatment |
| EP-RPS | Early Parkinson's Region Progression Score |
| ER | exposure-response |
| ICF | informed consent form |
| ICH | International Conference on Harmonisation |
| IDMC | independent data monitoring committee |
| INR | International normalized ratio |
| ITT | intent-to-treat |



Placebo-Controlled Period

| DZDC | Internation Value (WV-1- Decrees Contain |
|-----------|-------------------------------------------------------------|
| IXRS | Interactive Voice/Web Response System |
| LE | Lower Extremity |
| LOCF | last observation carried forward |
| LSmeans | least-square means |
| IV | intravenous |
| mAb | monoclonal antibody |
| MAO-B | monoamine oxidase type B |
| MCP-MOD | multiple comparison procedure – modeling |
| MDS-UPDRS | Movement Disorder Society Sponsored Revision of the Unified |
| | Parkinson's Disease Rating Scale |
| MedDRA | Medical Dictionary for Regulatory Activities |
| MMRM | mixed-model repeated measures |
| MRI | magnetic resonance imaging |
| PCS | potentially clinically significant |
| PD | Parkinson's disease |
| PIGD | Postural Instability Gait Difficulty |
| PK | pharmacokinetic(s) |
| PT | preferred term |
| PP | per-protocol |
| | per-protocor |
| RBC | red blood cell |
| RNA | ribonucleic acid |
| SAE | serious adverse event |
| SAP | statistical analysis plan |
| SBP | * * |
| SBR | systolic blood pressure<br>striatal binding ratio |
| SDK | Striatar officing ratio |
| CD | standard deriction |
| SD | standard deviation |
| SE | standard error |
| 500 | |
| SOC | system organ class |
| SPECT | single-photon emission computed tomography |
| TEAE | treatment-emergent adverse event |
| TD | Tremor Dominant |
| ULN | upper limit of normal |
| US | United States |
| WBC | white blood cell |
| WHO | World Health Organization |



#### 1 SCOPE OF WORK IN THE STATISTICAL ANAYSIS PLAN

This statistical analysis plan (SAP) only covers the analyses for the placebo-controlled portion of the study (Year 1). Hereafter, the placebo-controlled portion of the study will be referred to as "the study" in the rest of this SAP (e.g., completion of the study means completion of the placebo-controlled portion). A separate SAP will be prepared for the analyses of the dose-blinded extension period and integrated analyses across both portions of the study.

#### 2 DESCRIPTION OF OBJECTIVES AND ENDPOINTS

The objectives and endpoints of the study are listed below.

The secondary efficacy endpoints have been ranked based on the order of clinical importance.

| Primary Objective | Primary Endpoints |
|---|---|
| To evaluate the clinical efficacy of BIIB054 via dose response using the change from baseline in Movement Disorder Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Total Score | Change from baseline in MDS-UPDRS Total Score (Sum of Parts I, II, and III) at the primary timepoints of Week 52 and Week 72 |
| Secondary Objectives | Secondary Endpoints |
| To evaluate the clinical efficacy of BIIB054 based on MDS-UPDRS subparts | Change from baseline to Week 52 in MDS-UPDRS the subparts III, II and I (each part separately) |
| | Change from baseline to Week 72 and end of study in MDS-UPDRS the subparts III, II and I (each part separately) |
| To assess the PK profile of BIIB054 | Concentration of BIIB054 in the serum |
| To evaluate the dose-related safety of BIIB054 | Incidence of adverse events (AEs) and serious adverse events (SAEs) |
| To evaluate the pharmacodynamic effects of BIIB054 on the integrity of nigrostriatal dopaminergic nerve terminals | Change from baseline to Week 52 in striatal binding ratio (SBR) in the putamen, striatum, and caudate as measured by single-photon emission computed tomography (SPECT) imaging of the dopamine transporter (DaT) with ioflupane I123 (DaTscan <sup>TM</sup> ) |



Placebo-Controlled Period





Placebo-Controlled Period





Placebo-Controlled Period





Placebo-Controlled Period

V1.0



#### 3 STUDY DESIGN

#### 3.1 Study Overview

This Phase 2a, randomized, double-blind, parallel-group, placebo-controlled study (Year 1) with an active-treatment dose-blinded period (Years 2 through 4) will examine the efficacy, safety, PK, and pharmacodynamics of BIIB054, administered every 4 weeks via IV infusion



V1.0

to adult subjects with PD. Approximately 311 subjects will be enrolled at about 85 sites globally.

#### 3.1.1 Year 1 (Placebo-Controlled Portion of the Study)

Prior to the first dose in Year 1, all subjects in the study will be randomized into 4 arms, to receive 13 doses of BIIB054 (250, 1250, or 3500 mg) or placebo.

Subjects will be enrolled into 2 cohorts. Cohort A will be randomized first, in a 1:1:1:1 ratio into each of th e4 treatment arm and will include approximately 24 subjects. Randomization and dosing for Cohort B (approximately 287 planned subjects) will start after all subjects in Cohort A complete Week 12 assessments, and all available safety and PK data are reviewed by the IDMC. Randomization of subjects in Cohort B will be stratified by baseline (Day 1) MDS-UPDRS Part I + II + III total scores ( $\leq$ 35 and  $\geq$ 35) and striatum SBR ( $\leq$ 1.2 and  $\geq$ 1.2), and subjects will be randomized at Day 1 into 1 of 4 parallel dosing arms in each stratum.

After all subjects in Cohort A complete Week 12 assessments (28 days after their third infusion), and before dosing any subjects in Cohort B, all available safety and PK data will be reviewed by the IDMC. No subjects in Cohort B may be dosed until the IDMC review is complete. The study schematic is presented in Figure 1. After IDMC review is complete, subjects in Cohort B will be randomized, and dosing may begin. During the review period, subjects in Cohort A will continue to be dosed on a schedule of once every 4 weeks.

The first IDMC meeting will occur after the last subject in Cohort A completes Week 12 assessments, or approximately 6 months after the first subject has been enrolled in Cohort A, whichever comes first. Regular IDMC meetings will occur approximately every 3 months after the first meeting.

THe Week 48 infusion is the last infusion of the placebo-controlled period, and Week 52 is the first dosing of the Dose-blinded portion of the study.

#### 3.1.2 Years 2 Through 4 (Active-Treatment Dose-Blinded Portion of the Study)

Prior to Infusion 14 (the first dose of Year 2) at Week 52, subjects who received placebo in Year 1 will be randomized into 1 of the active-dosing arms for Year 2; these subjects will receive BIIB054 in Year 2. Subjects who received BIIB054 (1250 mg or 3500 mg) in Year 1 of the study will continue with the same dose regimen in Year 2. Subjects receiving the 250-mg dose in Year 1 continued on their original dose assignment.

Subjects will receive 12 additional doses of BIIB054 (250, 1250, or 3500 mg) in Year 2 and up to 16 additional doses in Years 3 and 4. Up until the last subject in the study has had his or her last dose in Year 2 of the study (Week 96 Visit), eligible subjects will be able to continue treatment once every 4 weeks.

Subjects who complete dosing through Week 96 and the Final Visit 12 weeks after the last visit will be considered Year 2 completers in the eCRF.



V1.0

See Figure 2 for a depiction of the duration of dosing in Years 3 and 4 for subjects continuing dosing past Week 96.

Figure 4 on protocol presents a flowchart for dosing and procedures from Week 96 through end of study, including how to determine which subjects are eligible to continue dosing past Week 96.

#### 3.2 Study Schematic

Figure 1: Study Design



DaT = dopamine transporter; IDMC = independent data monitoring committee; PK = pharmacokinetic(s); SPECT = single-photon emitomography

Figure 2: Overview of Study Dosing:

<sup>&</sup>lt;sup>a</sup> Prior to Infusion 14 (first dose of Year 2), subjects who received placebo in Year 1 will be randomized to 1 of the active-treatment graneeive BIIB054 in Year 2. Subjects who received BIIB054 in Year 1 will continue with the same dose regimen in Years 2 through 4. the last subject in the study has had his or her Week 96 Visit. Not all subjects will have the opportunity for dosing past Year 2/Week 9.



Placebo-Controlled Period

V1.0



Q4W = every 4 weeks.

Year 1 = Placebo-controlled period. Years 2 through 4 = Active-treatment dose-blinded period. Not all subjects will have the opportunity for dosing



V1.0

#### 3.3 Schedule of Events

See Protocol Section 4.2.

#### 4 SAMPLE SIZE JUSTIFICATION

The sample size calculation is based on changes in MDS-UPDRS Part I + II + III total score at Week 52 and at Week 72 of treatment. Based on data from the Parkinson's Progression Markers Initiative study, the placebo subject's mean and standard deviation (SD) at Week 52 and Week 72 are assumed to be 8.0 (10.64) and 9.6 (13.7) respectively. Assuming a maximum of 55% reduction in the change from baseline in the active group with maximum response relative to placebo group, the mean (SD) for this active group will be 3.2 (10.64) and 3.84 (13.7) respectively at Week 52 and Week 72, and the responses for other active groups are assumed to be somewhere between 0 and the maximum response. The primary analysis will be based on the MCP-MOD method to detect a dose-response trend while controlling for multiplicity. Optimal contrasts will be constructed to detect potential doseresponse trend under common dose-response curves (e.g., Emax, exponential, logistic, linear in log dose, and quadratic model, which are illustrated with parameters shown in Figure 4.1 which will be used for both Week 52 and Week 72). The planned enrollment is 311 subjects total (24 subjects in Cohort A and 287 subjects in Cohort B, 4.1). Actual enrollment is 357 subjects. In Cohort A, 29 subjects were randomized in a 1:1:1:1 ratio to each of the treatment groups, while in Cohort B 328 subjects were randomized in 2:1:2:2 ratio to the placebo, 250 mg, 1250 mg, and 3500 mg groups. Based on the actual enrollment, the estimated number of subjects by cohort and treatment groups are given in Table 4.4.2 below. After accounting for dropout rate of 10% and 15% at Week 52 and Week 72, respectively, the estimated sample sizes are given in Table and Table 1. With the updated sample size, the study will provide an average power of approximately 80% to detect the dose-response trend over 1 year of treatment, based on a 2-sided type I error of 0.05 and approximately 73% of power at the Week 72 analyses, based on a 2-sided type I error of 0.05. Overall, the sample size in the study will provide approximately 89% power, taking into consideration success at either Week 52 or Week 72. The final candidate models for the MCP-MOD are prespecified and described below.

With an estimated sample size of 100 subjects dosed per arm in the 1250 mg and 3500 mg arms, the study has 80% probability of detecting AEs with a rate of 1.6% or greater in these 2 arms, and a 90% probability of detecting AEs occurring with a rate of 2.3% or greater.



Placebo-Controlled Period

V1.0

Table 4.1: Estimated Sample Size Per Group (Planned)

| | Treatment Group | | | | |
|----------|-----------------|--------|---------|---------|-------|
| | | | | | Total |
| Cohort | | 250 mg | 1250 mg | 3500 mg | |
| Cohort A | 6 | 6 | 6 | 6 | 24 |
| Cohort B | 82 | 41 | 82 | 82 | 287 |
| Total | 88 | 47 | 88 | 88 | 311 |

Table 4.2: Estimated Sample Size Per Group Based on Actual Enrollment (Before Drop-Outs)

| | Treatment Group | | | | |
|---|---|---|---|---|---|
| | Placebo BIB054 BIB054 BIB054 Total | | | | |
| Cohort | | 250 mg | 1250 mg | 3500 mg | |
| Cohort A | 8 | 7 | 7 | 7 | 29 |
| Cohort B | 93 | 47 | 94 | 94 | 328 |
| Total | 101 | 54 | 101 | 101 | 357 |

Table 4.3: Estimated Sample Size Per Group Based on Actual Enrollment (After Adjusting for 10% Drop-Out At Week 52

| | Treatment Group | | | | |
|---|---|---|---|---|---|
| | Placebo BIIB054 BIIB054 Total | | | | |
| Cohort | | 250 mg | 1250 mg | 3500 mg | |
| Cohort A | 7 | 6 | 6 | 6 | 25 |
| Cohort B | 84 | 42 | 84 | 84 | 294 |
| Total | 91 | 48 | 90 | 90 | 319 |

Table 1: Estimated Sample Size Per Group Based on Actual Enrollment (After Adjusting for 15% Drop-Out At Week 72

| | Treatment Group | | | | |
|---|---|---|---|---|---|
| | Placebo BIIB054 BIIB054 Total | | | | |
| Cohort | | 250 mg | 1250 mg | 3500 mg | |
| Cohort A | 7 | 6 | 6 | 6 | 25 |
| Cohort B | 79 | 40 | 80 | 80 | 279 |
| Total | 86 | 46 | 86 | 86 | 304 |






■ EMax (EDs= 450.5) ● Exponential (ŏ = 2850.5) ▲ Logistic (EDs= 1547.5, ŏ = 510.5) ◆ Linear in log dose (off= 237.5) ■ Quadratic (ŏ = -2.2E-4) ▼ Exponential (ŏ = 860.5) ■ Linear

Figure 4.1: Candidate Models for Dose-Response

#### 5 STATISTICAL ANALYSIS METHODS

#### 5.1 General Considerations

Summary tables will be presented using descriptive summary statistics. For continuous variables, summary statistics will generally include: number of subjects with data, mean, standard deviation, median, and range (minimum and maximum). For categorical variables, this will generally include: number of subjects randomized or dosed, number with data, and the percent of those with data in each category.

Unless otherwise specified, baseline value is defined as the most recent non-missing measurement collected prior to the first dose. Change from baseline will be defined as post-baseline value minus baseline value.

Statistical testing will be performed to assess efficacy endpoints by conducting pairwise comparison between each BIIB054 group and placebo, and no multiplicity will be adjusted. Unless stated otherwise, all the statistical tests will be 2-sided with a statistical significance level of 0.05.

The statistical software, SAS® will be used for all summaries and analyses.

#### 5.1.1 End of Study (EOS) and End of Treatment (EOT)

For subjects who complete the placebo-controlled period of the study, EOS visit is defined as Week 52 visit; for subjects who are early terminated, EOS visit is defined as the scheduled



V1.0

follow-up visit after EOT visit. For subjects who complete the treatment, EOT visit is defined as Week 48.

#### 5.1.2 Analysis Population

- Intent-to-treat (ITT) population:
  - The intent-to-treat population is defined as all randomized subjects who received at least one dose of study treatment (BIIB054 or placebo).
- Per-protocol (PP) population:
  - The per-protocol population is defined as a subset of the ITT population who received at least 70% (10 doses) of study treatment (BIIB054 or placebo).
- Safety population:
  - The safety population is defined as all subjects who received at least one dose of study treatment (BIIB054 or placebo).
- PK population:
  - The PK population is defined as all subjects in the ITT population who had at least one measurable BIIB054 concentration in serum.
- Pharmacodynamic population:
  - The pharmacodynamic population is defined as all subjects in the ITT population who had at least one post-baseline pharmacodynamic measurement.
- Immunogenicity population:
  - The analysis population for immunogenicity is defined as all subjects in the safety population.



#### 5.2 Background Characteristics

The summaries in this section will be based on the ITT population. Unless otherwise specified, all the summary tables and listings will be presented by treatment group.

#### 5.2.1 Accounting of Subjects

The summary of subject disposition will include number (%) of subjects randomized, number (%) subjects randomized but not dosed, number (%) of subjects who completed the treatment/study, and number (%) of subjects who discontinued treatment and/or withdrew from study. For subjects who discontinued treatment and/or withdrew from study, the reasons for discontinuation and/or withdrawal, and days on treatment and days on study will be summarized and listed. The pattern (time and rate) of treatment discontinuation and study



V1.0

withdrawal will be displayed by Kaplan-Meier plot. The number of subjects in each analysis population will be summarized.

In addition, number of subjects dosed and number of subjects who completed the treatment/study will be summarized by country (region) and site.

The categorization of region is based not only on consideration of geography but also on type of health care system and access to health care in each country. The categories for regions will be:

- o Region 1: United States (US);
- Region 2: European countries (including Austria, France, Germany, Israel, Italy, Poland, Spain and United Kingdom) and Canada.

#### 5.2.2 Demographics and Baseline Characteristics

Demographic data, including age (in years), age category (40-50, 51-60, 61-70, 71-80 years), gender, race, ethnicity, height, weight, body mass index (BMI), country (region) and year of education at baseline will be summarized by treatment groups and overall.

Baseline PD history will be summarized by treatment groups and overall, using descriptive statistics. Time since onset of PD symptoms (in years), time since PD diagnosis (in years), subtype of PD (PIGD, TD or indeterminate), side predominately affected at disease onset, symptoms presented at PD diagnosis and immediate family with a history of Parkinson's Disease will be summarized. MDS-UPDRS total and subtotal scores, PIGD, TD, and LE subscore, Hoehn and Yahr stage,

will be

summarized. DaT/SPECT imaging outcomes,

outcomes will also be summarized. Baseline MDS-UPDRS score is defined as the Day 1 visit, if Day 1 visit score is not available, screening visit will be used. Baseline PD history data will be listed.

Number (%) of subjects with any PD treatment history will be summarized by treatment groups and overall. Total duration of previous therapies and reason for stopping therapies will be summarized. Number (%) of subjects who had taken MAO-B inhibitors, Dopamine Agonist, Levodopa and other PD medications will be displayed by treatment groups and overall. A listing of PD treatment history will be generated.

Medical history will be coded using the Medical Dictionary for Regulatory Activities (MedDRA). The number (%) of subjects with history (including both ongoing and not ongoing medical conditions) will be summarized by system organ class and preferred term, and by preferred term only. A listing of medical history will be generated.

#### 5.2.3 Concomitant Medications and Non-drug Therapies

All concomitant medications will be coded using the World Health Organization (WHO) medication dictionary. All concomitant non-drug therapies will be coded using the MedDRA dictionary. A concomitant medication/therapy will be defined as any therapy that was taken



V1.0

on or after the day of the first dose of study drug. This include therapies that start prior to the initiation of the first dose if their use continues on or after the date of first dose. To determine whether medications and/or non-drug therapies with missing start or stop dates are concomitant with study treatment, the following additional criteria will be used:

- If both the start and stop dates of a therapy are missing, then the therapy will be considered concomitant:
- If the start date is missing and the stop date of the therapy falls on/after the first dose date, then the therapy will be considered concomitant;
- If the start date is missing and the stop date of the therapy falls before the first dose date, then the therapy will be considered non-concomitant;
- If the start date of a therapy is prior to the date of the first dose and the stop date of the therapy is missing and the therapy is listed as ongoing, that therapy will be considered concomitant;
- If the start date of a therapy is prior to the date of first dose and the stop date of that therapy is missing and the therapy is not listed as ongoing, that therapy will be considered non-concomitant.
- If the start date of a therapy is on/after the date of first dose but in the treatment period (last dosing date+28 days) and the stop date of that therapy is missing, then that therapy will be considered concomitant.
- If the start date of a therapy is on/after the treatment period (last dosing date+28 days) and the stop date of that therapy is missing, then that therapy will be considered non-concomitant.

For a record with a partial start/end date, the year/month of the partial date will be compared to that of the date of first dose to determine whether it is concomitant.

The number and percent of subjects taking concomitant medication and non-drug treatments will be summarized by treatment group and overall. Concomitant PD medication will be summarized separately from the other concomitant medication.

#### **5.2.4 Protocol Deviations**

Protocol deviations identified during site monitoring will be captured in a Protocol Deviation log and categorized as major or minor deviations. The major protocol deviations will be summarized and listed. The minor protocol deviations will also be listed. Number (%) of subjects with at least one major deviation will be summarized by category. The protocol deviation related to COVID-19 will be listed.

#### 5.2.5 Study Drug Exposure and Study Drug Compliance

The number of infusions administered will be summarized as both continuous and category variables (categories as integers from 1 to 13, and 1-3, 4-6, 7-9, 10-13). The number of weeks on study drug, calculated as (date of last dose – date of first dose +1)/7, will be summarized CONFIDENTIAL



V1.0

as a categorical variable (every 8 weeks from 0 to ≥48 Weeks) as well as a continuous variable. Overall compliance, which is the percentage of drug infusions actually received over 13 planned doses, will be summarized regardless of study completion for all subjects. Percentage of study treatment taken up to the last dose, calculated as (the actual number of infusions / the number of infusions a subject is expected to take until the date of last infusion), will be summarized as a continuous variable. This table will be presented by treatment group. For subjects who completed study, the number of expected infusions is 13. For subjects who withdrew from study early, the number of expected infusions is the planned number of infusions before the time of withdrawal.

A listing of study drug administration records, including infusion start date and time, infusion stop date and time, total volume prepared, total volume administered, location of infusion, initial infusion rate, dose interruption or rate change or not, time of interruption or rate change, infusion rate after interruption or rate of change, reason for interruption or rate change will be provided.

#### 5.3 Efficacy Endpoints

#### 5.3.1 General Consideration

| Clinical efficacy (clinical function) Assessments include Movement Disorder Society Sponsor Revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS), | red |
|---|---|
| The questionnaire as well as the scor algorithm for all these clinical assessments are described in Appendix I. | ring |

Unless otherwise noted, the analysis will be performed based on all the subjects in both Cohort A and B and the common visits. For numerical outcomes, the actual value and the change from baseline will be presented by treatment group and visit. For categorical outcome, the count and frequency will be summarized by treatment group and visit.

#### Analysis population

All clinical function endpoints will be evaluated in the ITT population as defined in Section 5.1.2. MDS-UPDRS may also be analyzed in the per protocol population as defined in Section 5.1.2.

#### Baseline value

| MDS-UPDRS, | are assessed at both screening visit and Day |
|------------|----------------------------------------------|
| visit. | |



**Placebo-Controlled Period** 

V1.0

. For all of them, the baseline values are defined as the latest data collected prior to or on the first dose date.

#### Visit windows for mapping clinical function endpoint

Assessments from all scheduled visits, EOT visit and EOS visit, and unscheduled visits will be mapped to an appropriate analysis visit using a windowing scheme (Appendix II).

#### Handling missingness of itemed question score

For MDS-UPDRS, the maximum number of missing item allowable to provide a valid standard score for each part are: 2 for Part I, 2 for Part II, 9 for Part III, and 0 for Part IV. For each part, if no item is missing, the total score is the sum of all the item scores in the part. If some items are missing, the total score is the sum of all available item scores multiplied by the total number of items in the part and then divided by the number of items with available scores. MDS-UPDRS Part I+II+III (II+III) total score is the sum of all relevant part scores. As subjects were not guided to enter 0 to the Part IV questionnaire before they start symptomatic PD medication, some subjects left blank to the Part IV items at applicable visits. Therefore, we will impute the missing item in Part IV as 0. The total score is missing if and only if any relevant part score is missing (Stebbins et. al. 2015). For all other clinical endpoints, if more than half of the items are missing, then the total score is set to be missing. Otherwise, the missing item score will be imputed and used to derive the total score. In particular, if an item score is missing at a post baseline visit, it will be imputed by last observation carried forward method. And if an item score is missing at baseline, it will be imputed by the median of the item score among all the subjects of the same PD subtype (PIGD-dominant, Tremor-dominant, Indeterminate) in the study who have a baseline score in the item.

#### 5.3.2 MDS-UPDRS

#### 5.3.2.1 Primary efficacy endpoint

#### Estimand:

The estimand of the primary analysis is the mean difference of the change from baseline in MDS-UPDRS I+II+III total score at Week 52 between treatment groups in the ITT population in a hypothetical setting where subjects do not start PD medication. MDS-UPDRS data collected after the intercurrent events, i.e., subjects start PD medication will be excluded in the primary analysis. Specifically, the estimand takes the following into consideration:

- A. Population: ITT population as defined in Section 5.1.2
- B. Variable: change from baseline to Week 52 in MDS-UPDRS score
- C. Intercurrent events: had PD medication not been made available to subjects prior to Week 52
- D. Population-level summary: difference in variable means between treatment conditions.



V1.0

MMRM will be used as the primary analysis to analyze the change from baseline in MDS-UPDRS score. The model includes the fixed effects of treatment group, time (categorical), baseline PD subtype (categorical; PIGD vs TD vs indeterminate), prior use of PD medication (categorical), treatment group-by-time interaction, region (categorical), baseline MDS-UPDRS I+II+III total (continuous), baseline MDS-UPDRS I+II+III total by time interaction and baseline striatum SBR values (continuous), and baseline striatum SBR by time interaction. A random intercept and slope will be included in the model to model the random effects within subjects. If small sample size in subgroups of PD types causes lack of model convergence, the indeterminate group will be combined with the TD group. The Kenward-Roger approximation will be used to estimate the denominator degrees of freedom. Least square means (LSmeans) of each treatment group as well as treatment difference between BIIB054 groups and placebo will be displayed with 95% CI and p-value at Week 52. If the distribution of the outcome is highly skewed, p-value will be generated from the MMRM model based on ranked data. In the primary analysis, missing data are assumed to be missing at random (Rubin 1976), and MDS-UPDRS I+II+III score is impacted by PD medication.

The multiple comparison procedure-modelling (MCP-MOD) method will be used to assess the dose-response relationship while controlling for multiplicity (Pinheiro 2013). The dose-response parameter of interest for MCP-MOD are the least-squares means (LSmeans) at Week 52 for each treatment group from the MMRM model. The underlying models to be tested are specified in Figure 4.1. P-value of dose response will be presented. Details of MCP-MOD procedure are specified in Appendix III.

A multiple comparison adjustment method will be applied to control the overall type I error at 0.05 in the study, due to the primary endpoint of change from baseline in MDS-UPDRS total score being analyzed at Week 52 and Week 72, and superiority against placebo is considered reached in the study if statistically significant result is achieved at either timepoint at the respective adjusted alpha-level. This will be applied to the p-value from the MCP-MOD model. Please refer to Section 6 "Interim Analyses" for more detail.

Nominal p-values for pair-wise comparison of each active group vs placebo will be reported, no additional multiple comparison adjustment will be applied.

Item 1.6 of features of dopamine dysregulation syndrome will be excluded to calculate all the scores.

#### 5.3.2.2 Secondary endpoints and additional

MDS-UPDRS based endpoints

The analysis approach and the MMRM model as described for the primary endpoint will be performed for additional MDS-UPDRS based endpoints as listed below, except that, 1) the baseline MDS-UPDRS I+II+III total score term in the model will be replaced by the corresponding baseline value of MDS-UPDRS total or sub-part score being analyzed, 2) MCP-MOD dose-response may be performed, 3) no additional multiple comparison adjustment will be applied for secondary efficacy

- MDS-UPDRS Parts I, II, III (Secondary Efficacy Endpoints),
- MDS-UPDRS Parts II+III, Ib+II+III



Placebo-Controlled Period

V1.0

- Postural Instability -Gait Difficulty (PIGD) score (mean score of MDS-UPDRS items 2.12+2.13+3.10+3.11+3.12),
- Lower Extremity (LE) score (mean score of MDS-UPDRS items 3.10+3.11+3.12+3.13+3.3d+3.3e+3.7a+3.7b+3.8a+3.8b+3.17c+3.17d+2.12+2.13), and Tremor score (mean score of MDS-UPDRS items 2.10+3.15a+3.15b+3.16a+3.16b+3.17a+3.17b+3.17c+3.17d+3.17e+3.18).

#### 5.3.2.3 Sensitivity analysis

A sensitivity analysis will be conducted for MDS-UPDRS based endpoints, by including the data after PD medication assessed in the "OFF" status, that is, the assessment was made at least 12 hours since the last time the subject took the medication, or assessed in the "off" status by the rater, or if subject reported not taking PD medication at that visit.

The analyses will be performed based on the same MMRM model as described for the primary endpoint, except the following:

 An unstructured covariance matrix will be used to model the within-subject variancecovariance errors (instead of random intercept and slope). If the unstructured covariance structure matrix results in a lack of convergence, the heterogeneous Toeplitz covariance structure followed by the heterogeneous first-order autoregressive covariance structure will be used.

The table below summarizes the detailed information.

| | | Primary analys | ses | Sensivity analyses | |
|---|---|---|---|---|---|
| MDS-<br>UPDRS<br>endpoints | Туре | MMRM<br>model<br>covariance<br>structure | Data after PD<br>medications<br>included (Y/N) | MMRM<br>model<br>covariance<br>structure | Data after PD<br>medications<br>included (Y/N) |
| I+II+III | Primary | | N | | Y |
| I | Secondary | Based on random | N | Based on pre- | Y |
| II | Secondary | | N | specified covariance | Y |
| III | Secondary | slope and | N | structure<br>(UN if no | Y |
| | | intercept - | | convergency<br>issue | |
| | | | | occurs) | |

| Biogen | Statistical Analysis Plan<br>Placebo-Controlled Period | V1.0 |
|---|---|---|

#### 5.3.2.4 Early Parkinson's Regional Progression Score (EP-RPS) measure

The Early Parkinson's Regional Progression Score (EP-RPS) measure is a novel method of assessing disease progression based on a modified scoring algorithm for the MDS-UPDRS Part III items that is potentially more reliable and sensitive to progression in early stages of PD, as compared with change in MDS-UPDRS Part III total score. The new concept has been developed to capture the spread of the progression of disease symptoms across body regions as a reflection of the underlying topographic spread of pathology. Figure 5.1 shows a general diagram of the concept of EP-RPS and the detailed definition are provided in Appendix IV.

Figure 5.1: Diagram of the concept of EP-RPS measure



EP-RPS will be summarized and analyzed by using ANCOVA model. The model will include the endpoint as the outcome, fixed effect of treatment group (categorical) and adjust for region (categorical), baseline PD subtype (categorical), baseline MDS-UPDRS Part III total score (continuous) and baseline striatum SBR values (continuous). Least square means (LSmeans) of each treatment group as well as treatment difference between BIIB054 groups and placebo will be displayed with 95% CI and p-value at Week 52. MDS-UPDRS Data after the PD medication will be included and excluded in two separate analyses, since this endpoint is unknown, though expected to be minimally impacted by PD medications and including the data will reduce the amount of missing data.

Spearman's correlation of this endpoint with change from baseline at Week 52 in MDS-UPDRS Part III will be calculated.



Placebo-Controlled Period





**Placebo-Controlled Period** 

V1.0



#### 5.3.2.8 Subgroup analysis

Subgroup analyses will be performed for the outcomes of MDS-UPDRS part III and I+II+III respectively in the subgroups of the following baseline covariates. The MMRM model is the same as the one in the primary analyses. If the MMRM model of a specific subgroup does not converge, no results will be displayed for that subgroup. A forest plot will be generated to present the results of all subgroups together.

- Age (above v.s. below median)
- Gender (male v.s. female)
- region, (US v.s. Other)
- prior use of PD medication (Yes v.s. No)
- time since onset of PD symptoms (above v.s. below median)
- baseline type of PD (tremor-dominant v.s PIGD-dominant v.s. Indeterminate)
- baseline MDS-UPDRS III (above v.s. below median)
- baseline MDS-UPDRS I+II+III (above v.s. below median),
- baseline modified H&Y stage (<=1.5 v.s. >=2)
- •
- baseline total striatum SBR measure, occipital reference (<=mean-sd v.s >mean-sd to <=mean+sd v.s. >mean+sd)
- baseline contralateral putamen SBR measure, occipital reference (<=mean-sd v.s >mean-sd to <=mean+sd v.s. >mean+sd)
- baseline ipsilateral putamen SBR measure, occipital reference (<=mean-sd v.s >mean-sd to <=mean+sd v.s. >mean+sd)
- •
- baseline total striatum volume (above v.s. below median),
- baseline lateral ventricle volume (above v.s. below median),
- •
- baseline stride time variability (above v.s. below median),

Subgroup analysis will be performed respectively by including and excluding data after PD medication. The forest plot will be generated respectively as well. Besides, subgroup analysis of time to start of PD medication will be performed for the subgroup of regions (US v.s. Italy v.s Other)



V1.0

#### 5.3.2.9 Per-protocol analysis

The per-protocol analysis will be performed in the same fashion as the primary analysis for MDS-UPDRS I+II+III, but by applying in the per-protocol population as defined in Section 4.1. If the per-protocol population is largely the same as the ITT population, i.e.,  $\geq 90\%$  of subjects included in the ITT population are also included in the per-protocol population, then the per-protocol analysis will not be performed.

#### 5.3.3 Other clinical efficacy endpoints

Other clinical efficacy (function) and quality of life assessments are listed as below. The questionnaire as well as the scoring algorithm for these clinical assessments are described in Appendix I.



- Clinical Global Impressions Improvement (CGI-I) Scale (collected at Week 52 in the US sites only)\*,
- Patient Global Impression of Change (PGI-C) (collected at Week 52 in the US sites only)\*.

Data after PD medication will be included in the analysis for all the outcomes except

For each clinical assessments that are collected longitudinally, an MMRM model will be used to analyze the change from baseline in the continuous clinical outcome, with addition of adjustment for the corresponding baseline outcome value and its interaction with time. i.e. the model will include fixed effects of treatment group (categorical), time (categorical), region (categorical), treatment group-by-time interaction, baseline value of the corresponding outcome (continuous), baseline value of the outcome by time interaction, baseline MDS-UPDRS I+II+III total score (continuous), baseline MDS-UPDRS I+II+III total score-by-time interaction, baseline striatum SBR values (continuous), and baseline striatum SBR by time interaction. The endpoints listed with a "\*" next to them, will additionally include the baseline PD subtype (categorical) as a covariate. An unstructured covariance matrix will be used to model the within-subject variance-covariance errors. If the unstructured covariance structure matrix results in a lack of convergence, the heterogeneous Toeplitz covariance structure followed by the heterogeneous first-order autoregressive covariance structure will



V1.0

be used. Least square means (LSmeans) of each treatment group as well as treatment difference between BIIB054 groups and placebo will be displayed with 95% CI and p-value at Week 52.

For CGI-I and PGI-C that are only collected at Week 52, an ANCOVA model will be used to analyze the data and adjust for the covariates of baseline MDS-UPDRS I+II+III (continuous) and baseline straiatum SBR values (continuous), and baseline PD subtype (categorical).

The Spearman's correlation of change from baseline at Week 52 in each clinical outcome with that of the MDS-UPDRS I+II+III, EP-RPS will be computed by including and excluding data after PD medication respectively





Placebo-Controlled Period





V1.0



#### 5.3.5 Assessment of the Impact of Covid-19 on the clinical outcome analyses

As this study is on-going when the Covid-19 public health emergency (PHE) occurred, subject visits and data collection were impacted, including missing visits, missed assessments, delayed visits and/or some visits were performed via remote assessments, e.g. telephone/video visits. Every effort was made to document these impacted study activities systematically on the eCRF and othe electronic source data.

A complete listing of all visits impacted (e.g. missed visits, delayed or assessment done via remote visits) will be listed in the clinical study report.

In addition, subgroup analyses of the selected key clinical outcome MDS-UPDRS will be performed on a subset of subjects who did not have >=3 consecutive missing doses throughout the study to further evaluate the impact of Covid-19 on the study. The same MMRM model for the primary analyses will be used for the subgroup analyses.

In addition, due to Covid-19, some visits were delayed. A few subjects will have their Week 52 imaging done at later visits up to Week 72 and these will still be considered as Week 52 visit data in the analyses for Week 52. These data were not included in the Week 52 database lock in time, but will be included in the Week 72 database, and the related Week 52 imaging analyses will be updated at the time of the Week 72 interim analyses.

#### 5.4 Safety Analysis

#### 5.4.1 General Considerations

#### Analysis population

All safety endpoints will be evaluated in the safety population (all subjects dosed) as defined in Section 5.1.2.

#### Methods of analysis

All adverse events (AEs) and serious adverse events (SAEs), clinical laboratory abnormalities, vital sign measurements, physical and neurological examination findings, 12-lead ECG readings, disease activity by brain MRI metrics, body weight and Columbia Suicide Severity Rating Scale (C-SSRS) will be evaluated for safety. Safety data collected by EOS defined in Section 5.1.1 will be used for the safety analyses. The main safety analysis will include data after PD medication. Additional analyses may be performed by excluding CONFIDENTIAL



V1.0

data after PD medication. Unless mentioned otherwise, all safety data will be summarized by treatment group and overall active group.

Although treatment assignment error is not expected, if some subjects received different study treatment than the randomization allocation, the safety analyses will be based on the actual treatment allocation. Specifically, if a subject who was assigned placebo received BIIB054 at any visit at the same dose level by mistake, this subject will be included in the BIIB054 group of that dose in the safety statistical analyses; if a subject was assigned placebo or BIIB054 of certain dose level, but received BIIB054 at multiple dose level by mistake, this subject will be included in the BIIB054 group of the dose level that were taken the most frequently in the safety statistical analyses; on the other hand, if a subject who was assigned BIIB054 does receive placebo by mistake, this subject will be included under placebo group in the safety statistical analyses only when this subject received placebo at all study visits.

For the clinical laboratory assessments, vital sign measurements and 12-lead ECG readings, subjects in Cohort A have additional post-baseline visits between Day 1 and Week 12, comparing to Cohort B. The summary of numerical changes over time, i.e., the quantitative analysis will be based on the pooled data of both Cohort A and Cohort B and the common visits. All the qualitative analyses including the shift analysis, grade analysis and so on will be based on all the data of Cohort A and Cohort B of all visits. All the listings will be based on all the data of Cohort A and Cohort B of all visits.

#### Visit windows for mapping safety endpoint

For safety data that are summarized by visit, assessment from all scheduled visits, EOT visit, EOS visit and unscheduled visits will be mapped to an appropriate analysis visit using a windowing scheme (Appendix II).

#### **5.4.2** Clinical Adverse Events

For this study, any AE experienced by a subject between the time of first dose of study treatment (Day 1/Baseline) and the end of study visit is to be recorded on the CRF, regardless of the severity of the event or its relationship to study treatment. Any SAE experienced by the subject between the time the subject has signed the ICF and the end of study visit is to be recorded, regardless of the severity of the event or its relationship to study treatment.

All AEs will be coded using the MedDRA and will be analyzed based on the principle of treatment emergence. An AE will be regarded as treatment-emergent if it was present prior to the first dose and subsequently worsened in severity or was not present prior to first dose but subsequently appeared.

In order to define treatment emergence for AE with missing start or stop dates, the following additional criteria will be used:

- If both the start and stop dates for a particular event are missing, then that event is considered treatment-emergent;
- If the start date for a particular event is missing and the stop date/time falls after the first dose date/time, then that event is considered treatment-emergent;



V1.0

• If the start date is the same as the first dose date, and the start time is missing, then that event is considered treatment-emergent.

For events with a partial start date, the year/month of the event date will be compared to that of the first dosing date to determine whether the event is treatment emergent.

Only TEAEs and TESAEs will be summarized in the tables, unless otherwise specified. All SAEs (including pre-dosing SAEs) will be included in the listing of SAEs, with an indicator of pre-dosing or treatment-emergent. Only TEAEs will be included in other AE listings, if not otherwise specified.

The overall summary table of AEs will present the number of subjects with the following events for each treatment group, BIIB054 total and overall. A subject is counted only once in each category.

- Any AE;
- AE by severity as measured in CTCAE grade of version 5.0: 1 (mild), 2 (moderate), 3 (severe or medically significant), 4 (life-threatening), 5 (death)
- Study drug-related AE;
- •
- Radioligand related AE;Any SAE;
- Study drug-related SAE;
- •
- Radioligand related SAE;
- AE leading to discontinuation of study treatment; and
- AEs leading to withdrawal from study
- Death

The incidence of AEs will be summarized using the primary system organ class (SOC) or preferred term (PT) or both, sorted by decreasing frequency and alphabetical order, respectively. Additionally, AEs at least 5% higher in incidence for any active group compared to placebo group will be summarized by SOC and PT.

The incidence of AEs will also be summarized by severity as measured in CTCAE grade of version 5.0 using system organ class and preferred term. Within each system organ class or/and preferred term, the same subject will be counted only once. Under the same system organ class or/and preferred term, the occurrence of the adverse event with the greatest severity will be used in the calculation of incidence by severity.

The study drug related AEs, and radioligand related AEs will be summarized by SOC, PT and treatment group as well.

The incidence of SAEs will be summarized by primary system organ class, preferred term and treatment group. Study drug related SAEs, and radioligand related SAEs will be summarized in the same fashion as well.

Tables of AEs that led to study drug discontinuation and AEs that led to study withdrawal by SOC, PT and treatment group will be presented.



V1.0

Listings of all AEs, SAEs, AEs that led to study drug discontinuation, and AEs that led to study withdrawal will be presented. Listing of death will be provided if applicable.

In some AE/SAE listings, complete AE start and end dates are needed to calculate the relative study days of AE start and end. Therefore, any partial date will be imputed for these listings. Specifically, the partial AE start date will be imputed as the earliest possible date on or after the first dose based on the partial information, and the partial AE end date will be imputed as the latest possible date on or before the EOS.

#### AEs around the time of infusion

The incidence of AEs within 2 hours from infusion start will be summarized by preferred term and visit for each treatment group. At each visit, the same subject will be counted only once within each preferred term. Preferred terms will be ordered by decreasing frequency of AEs in the BIIB054 total column. Listings of such AEs within 2 hours from infusion start will be provided by treatment group.

#### 5.4.3 Clinical Laboratory Data

The following clinical laboratory parameters are assessed in the protocol:

- Hematology: Complete blood count with differential and platelet count, INR, prothrombin time, and APTT
- Blood chemistry: total protein, albumin, creatinine, blood urea nitrogen, uric acid, bilirubin (total and direct), alkaline phosphatase, alanine aminotransferase, aspartate aminotransferase, gamma-glutamyl transferase, glucose, calcium, phosphorus, bicarbonate, chloride, sodium, and potassium
- Urinalysis: dipstick for blood, protein, and glucose (microscopic examination may also be performed)





**Placebo-Controlled Period** 

V1.0

All the laboratory tables and listings, unless otherwise specified, will be presented by treatment group.

#### **5.4.3.1** Quantitative laboratory analyses

For numeric laboratory parameters, actual values, change and percent change from baseline will be summarized by visit. Number of evaluable subjects, mean, standard deviation, median, min and max values will be presented at each visit.

Plots of mean values (with standard deviation) for key numeric laboratory parameters by visit will be provided.

#### Visit windows for by visit summaries

For laboratory by visit summaries, the analysis visit should be defined using visit windows in Appendix II. If there is more than 1 value in the same analysis visit window (>1 value for the same analysis visit) for a certain parameter for a subject, then the closest record to the target visit day will be used for the by visit analysis. If there are 2 values in the same analysis visit window with the same distance from the target visit day for a certain parameter for a subject, then the record with the later date will be used for the by visit analysis. If there are 2 values on the same day for a certain parameter for a subject, then the record with the later time will be used for the by visit analysis. If there are 2 records on the same date and time, then use the average value for quantitative parameters and the worse value for qualitative parameters.

#### 5.4.3.2 Qualitative laboratory analyses

For all qualitative analyses, all values will be included (not just the "analyzed record" within each visit window in the quantitative analyses).

#### Shift analyses

Laboratory data will be summarized using shift tables where appropriate. Each subject's hematology, blood chemistry and urinalysis numeric values will be flagged as "low", "normal", or "high" relative to the normal ranges of the central laboratory or as "unknown" if no result is available. Each subject's urinalysis categorical values will be flagged as "positive", "negative", or "unknown" if no value is available. Shifts from baseline to high/low status will be presented for hematology, blood chemistry and urinalysis numeric parameters, and shifts from baseline to abnormal (positive) will be presented for urinalysis categorical parameters.

In the hematology, blood chemistry and urinalysis numeric values shift summary tables, entries are numbers of subjects shift to low (or high) divided by number of subjects at risk CONFIDENTIAL



Placebo-Controlled Period

V1.0

followed by corresponding percentages. Number at risk for shifting to low (or high) is the number of subjects whose baseline value was not low (or high) and who had at least one post-baseline evaluation. Shift to low includes normal to low, high to low, and unknown to low. Shift to high includes normal to high, low to high, and unknown to high.

In the urinalysis categorical values shift summary table, entries are numbers of subjects shift to abnormal (positive) divided by number of subjects at risk followed by corresponding percentages. Number at risk for shift to abnormal (positive) is the number of subjects whose baseline value was not abnormal (positive) and who had at least one post-baseline evaluation. Shift to abnormal (positive) includes normal or negative to positive and unknown to positive.

#### Potentially Clinically Significant (PCS) laboratory abnormalities analyses

For hematology, blood chemistry and urinalysis, the number of subjects with potentially clinically significant laboratory abnormalities post-baseline will be summarized for the parameters provided in Table 5.1. Subjects need to have at least one post-baseline evaluation in order to be included in the analysis.

Listings will also be presented for all subjects with any PCS laboratory abnormalities. In these listings, each subject's complete history from screening to last study visit for that specific laboratory test meeting the PCS criteria will be listed; any abnormal values based on the normal ranges of the central laboratory and abnormal values based on PCS criteria will be separately flagged in the same listing.

Table 5.1. Criteria to Determine Potentially Clinically Significant (PCS) Laboratory Abnormalities

| Clinical Labo | | | |
|---|---|---|---|
| Parameter name | PCS Low | PCS High | STANDARD UNIT in the SDTM dataset |
| HEMATOLOGY | | | |
| Basophils Absolute | N/A | >1.6 x 10 <sup>9</sup> /L | 10 <sup>9</sup> /L |
| Eosinophils | N/A | >1.6 x 10 <sup>9</sup> /L | $10^{9}/L$ |
| Erythrocytes (RBC) | $\leq 3.5 \times 10^{12}/L$ | $\geq$ 6.4 x 10 <sup>12</sup> /L | $10^{12}/L$ |
| Hematocrit - Females | ≤0.32 | ≥0.54 | L/L |
| Hematocrit - Males | ≤0.37 | ≥0.60 | L/L |
| Hemoglobin - Females | ≤95 g/L | ≥175 g/L | g/L |
| Hemoglobin - Males | ≤115 g/L | ≥190 g/L | g/L |
| Leukocytes (WBC) | <3.0 x 10 <sup>9</sup> /L | >16 x 10 <sup>9</sup> /L | $10^{9}/L$ |
| Lymphocytes | <0.8 x 10 <sup>9</sup> /L | >12 x 10 <sup>9</sup> /L | $10^{9}/L$ |
| Monocytes | N/A | >2.5 x 10 <sup>9</sup> /L | $10^{9}/L$ |
| Neutrophils | <1.5 x 10 <sup>9</sup> /L | >13.5 x 10 <sup>9</sup> /L | 10 <sup>9</sup> /L |
| Platelet count | ≤75 x 10 <sup>9</sup> /L | ≥700 x 10 <sup>9</sup> /L | 10 <sup>9</sup> /L |
| BLOOD CHEMISTRY | | | |
| Albumin | ≤25 g/L | ≥625 g/L | g/L |
| Alkaline phosphatase (ALP) | N/A | >3 x ULN | IU/L |
| Alanine aminotransferase (ALT) | N/A | >3 x ULN | U/L |
| Aspartate aminotransferase (AST) | N/A | >3 x ULN | IU/L |
| Bicarbonate | ≤16 mmol/L | ≥35 mmol/L | mmol/L |



Placebo-Controlled Period

V1.0

| Clinical Laboratory Outlier Criteria | | | |
|---|---|---|---|
| Parameter name | PCS Low | PCS High | STANDARD UNIT in the SDTM dataset |
| Bilirubin | N/A | >1.5 x ULN | umol/L |
| Calcium | ≤2 mmol/L | ≥3 mmol/L | Mmol/L |
| Chloride | ≤90 mmol/L | ≥118 mmol/L | Mmol/L |
| Creatinine | N/A | ≥176.8 umol/L | Umol/L |
| Gamma-Glutamyl Transferase | N/A | >3 x ULN | U/L |
| Glucose | ≤2.2 mmol/L | ≥9.7 mmol/L | Mmol/L |
| Potassium | ≤3 mmol/L | ≥6 mmol/L | Mmol/L |
| Phosphate | ≤0.6 mmol/L | ≥1.7 mmol/L | Mmol/L |
| Protein | ≤45 g/L | ≥100 g/L | g/L |
| Sodium | ≤126 mmol/L | ≥156 mmol/L | Mmol/L |
| Urate | N/A | >475.88 umol/L<br>(female); >594.85<br>umol/L (male) | umol/L |
| Urea Nitrogen | N/A | ≥10.7 mmol/L | Mmol/L |
| <u>URINALYSIS</u> | | | |
| Glucose | N/A | Trace or ≥ ++++ | |
| Protein | N/A | Trace or ≥ ++ | |
| Occult Blood | N/A | Trace or ≥+ | |
| ULN = upper limit of normal | | | |

#### Potential serious hepatotoxicity

Potential serious hepatotoxicity is defined as ALT or AST > 3x ULN and total bilirubin > 2x ULN at any time post-baseline, not necessarily concurrent. A scatterplot of the maximum post-baseline ALT or AST value relative to ULN and maximum post-baseline total bilirubin value relative to ULN (not necessarily concurrent) will be provided. In addition, a line plot of ALT, AST, ALP and total bilirubin values over time for each subject with potential serious hepatotoxicity will be provided.

A listing of subjects with potential serious hepatotoxicity will be provided with the concurrent records labeled. Concurrent is defined as on the same day. Subjects with ALT > 1x ULN, > 3x ULN, > 5x ULN, > 10x ULN or > 20x ULN, subjects with AST > 1x ULN, > 3x ULN, > 5x ULN, > 10x ULN or > 20x ULN, subjects with total bilirubin > 1x ULN, > 1.5x ULN or > 2x ULN, subjects with ALP > 1x ULN or > 1.5x ULN, and subjects with AST or ALT > 3x ULN post-baseline accompanied by concurrently elevated total bilirubin > 1.5x ULN or > 2x ULN will be labeled.

#### 5.4.4 Vital Sign Data

Vital sign parameters include diastolic blood pressure, systolic blood pressure, body temperature, pulse rate and respiration rate. Vital signs will be measured with the subject supine and after the subject has been resting for at least 10 minutes. The analysis of vital signs will focus on the incidence of clinically relevant abnormalities based on the following criteria in Table 5.2.



V1.0

Table 5.2. Criteria Used to Clinically Relevant Abnormalities in Vital Signs

| Variable | Low | High |
|---|---|---|
| Body temperature | <36 degrees C | >38 degrees C |
| Pulse Rate | <60 bpm | >100 bpm |
| Systolic Blood Pressure (Supine) | <90 mm Hg or a decrease from baseline of >30 mm Hg | >140 mm Hg or an increase from baseline of >40 mm Hg |
| Orthostatic Systolic Blood<br>Pressure | > 20 mm Hg decrease from supine to 3-minute standing measure | |
| Diastolic Blood Pressure | < 50 mm Hg or a decrease from<br>baseline of > 20 mm Hg | ≥90 mm Hg or an increase from basleine of >30 mm Hg |
| Orthostatic Diastolic Blood<br>Pressure | >10 mm Hg decrease from supine to 3-minute standing measure | |
| Respiration Rate | < 12 breaths per minute | >20 breaths per minute |
| Weight | ≥7% decrease from BL | ≥7 % increase from BL |
| BL= baseline; bpm = beats per | minute | l |

Note: the clinically relevant abnormality criteria will be evaluated based on the supine measure unless otherwise mentioned.

A summary table for subjects with any clinically relevant post-baseline abnormalities will be provided. In the summary table, entries are numbers of subjects with an abnormality divided by number of subjects evaluated followed by corresponding percentages. Number evaluated is the number of subjects who had a baseline assessment and at least one post-baseline assessment for that vital sign.

The descriptive statistics for actual values and change from baseline will be summarized over time for each treatment group and overall active group. The line of mean vital sign over time by treatment group will be graphed.

A subject listing will be presented for subjects with any post-baseline clinically relevant abnormalities in vital signs. In this listing, each subject's complete vital sign values from screening to last study visit will be listed with abnormalities labeled.

#### <u>Visit windows for by visit summaries</u>

For vital sign visit summaries, the analysis visit will be defined by visit window in Appendix II. For the same parameter for a subject, if there is more than 1 record in the same analysis visit window), then select the record closest to the target visit day. If there are 2 records in the same analysis visit window with the same distance from the target visit day, then select the record with the later date. If there are 2 records on the same date, then use the average value for quantitative parameters and the worse value for qualitative parameters.

#### 5.4.5 ECG Data

Actual value and change from Baseline in ECG will be summarized using descriptive statistics and presented by treatment group, overall active group and visit.

The ECG result is classified as normal or abnormal. The post baseline abnormal ECG result is further classified as abnormal AE or Abnormal but not AE. Shift table from normal or CONFIDENTIAL



V1.0

unknown ECG at baseline to abnormal post-baseline ECG will be summarized. The worst post-baseline record of each subject is selected. Subjects with abnormal post-baseline ECG status will be listed.

In addition, the number of subjects with potential QTcF interval outlier post-baseline will be summarized by treatment group. The criteria of defining QTcF interval outliers is specified in Table 5.3.

Table 5.3. Criteria used for QTcF interval outlier

| Variable | Low | High |
|-----------------------------------|-----|------------------|
| QTcF interval (msec.) | NA | >450; >480; >500 |
| Increase in QTcF interval (msec.) | NA | >30;>60 |

#### Visit windows for by visit summaries

For ECG visit summaries, the analysis visit will be defined by visit window in Appendix II. For the same subject, if there is more than 1 record in the same analysis visit window, then the record closest to the target visit day is selected. If there are 2 records in the same analysis visit window with the same distance from the target visit day, then the record with the later date is selected. If there are 2 records on the same date, then the worse record is selected.

#### 5.4.6 Physical and Neurological Examination

Abnormal findings during physical and neurological examinations are captured as adverse events and will be reflected in the summary of AEs.

#### 5.4.7 C-SSRS Data

The Columbia Suicide Severity Rating Scale (C-SSRS) is an assessment that evaluates suicidal ideation and behavior. C-SSRS measurements are collected with respect to "Lifetime: time he/she felt most suicidal" and "P3M: time he/she felt most suicidal during the past 3 month" at baseline, and with respect to "Since last visit" at post-baseline visit.

There are 11 common "Yes/No" questions at baseline and post-baseline visits. Five questions on <u>suicidal ideation</u> and five questions on <u>suicidal behavior</u> are re-ordered and follow increasing severity order respectively as shown in Table 5.4; another question on <u>self-injurious behavior without suicidal intent</u> is listed separately. In particular, only subjects who answered "Yes" to question 2 will proceed to question 3, 4 and 5, and the questions in the section of intensity of ideation. Thus, for any subjects who answered "No" to question 2, an answer "No" will also be assumed to question 3, 4, and 5. An additional "Yes/No" question is used to record if subject had committed suicide in post-baseline visits.

Table 5.4: C-SSRS re-ordered questions

| Suicidal Ideation | |
|--------------------------------------------------|-----------------|
| Question 1 | Wish to be dead |
| Question 2 Non-specific active suicidal thoughts | |



V1.0

| Question 3 | Active suicidal ideation with any methods (not plan) without intent to act |
|---|---|
| Question 4 | Active suicidal ideation with some intent to act, without specific plan |
| Question 5 | Active suicidal ideation with specific plan and intent |
| Suicidal Behavior | |
| Question 6 | Preparatory acts or behavior |
| Question 7 | Aborted attempt |
| Question 8 | Interrupted attempt |
| Question 9 | Actual attempt |
| Question 10 | Suicidal behavior |
| Question 11 (post-baseline visits | Suicide |
| only) | |
| Self-Injurious Behavior without Suicidal Intent | |
| Question 12 | Self-injurious behavior without suicidal intent |

A subject is considered to have <u>suicidal ideation</u> at the period of interest if a "Yes" is answered to any of the five suicidal ideation questions (Question 1-5). A subject is considered to have <u>suicidal behavior</u> at the period of interest if a "Yes" is answered to any of the five suicidal behavior questions (Question 6-10) at baseline or a "Yes" is answered to any of the six suicidal behavior questions (Question 6-11) at post-baseline visit.

A subject's <u>Suicidal Ideation Score</u> is defined as the maximal suicidal ideation question number (maximal of 1-5) with an answer "Yes" per visit. The score is defined as 0 if the subject answered "No" to all 5 Suicidal Ideation questions at that visit.

The following analyses on C-SSRS measurements will be conducted:

• Descriptive summary of subjects who answered "Yes" to any question 1-12 as well as subjects who had suicidal ideation or suicidal behavior at baseline and at any post-baseline visit, the denominator for summary is the number of subjects who were dosed and had a baseline assessment and at least one post-baseline assessment for each question.

Listing of subjects having a post-baseline suicidal ideation will be provided. The listing will display both baseline and post-baseline suicidal ideation scores for each subject.

#### 5.4.8 MRI Safety Data

Brain MRI safety finding (may include T1, fluid-attenuated inversion recovery, gradient echo) or other modalities and sequences (to be detailed in Imaging/MRI manual) are assessed at Screening visit, Week 24 and 52 visits.

The MRI safety result is classified as normal or abnormal. Shift table from normal or unknown MRI at baseline to abnormal post-baseline MRI will be summarized. The worst post-baseline record of each subject is selected. A listing of details for abnormal brain MRI findings will also be presented.



V1.0

#### 5.5 Pharmacodynamic - Imaging Analysis

#### 5.5.1 Type of imaging techniques and imaging outcomes

There are three types of imaging techniques used in the study:

(1) DaT/SPECT imaging,
(2)

DaT/SPECT imaging assesses the biological effects of BIIB054 on brain dopamine neurons and nerve terminals. DaT-associated outcome measures include the estimates of anterior and posterior putamen, caudate, as well as total striatum striatal binding ratio (SBR), a measure that compares signal intensity in the region of interest to that in the occipital cortex, a region relatively devoid of dopamine nerve terminals. Measurements are obtained both ipsilateral and contralateral to the side of worst motor symptoms, anterior, posterior as well as combining both sides.



#### 5.5.2 Analysis population

All pharmacodynamic imaging endpoints will be evaluated based on the Pharmacodynamics population as defined in Section 5.1.2.

#### 5.5.3 **Baseline value**

Baseline value is defined as the latest data collected at any time prior to the first dose, or if collected only after dosing the earliest data on the first dose date, given the data is collected within 1 week after first dose date.

#### 5.5.4 Outlier of percent change from baseline

If the percent change from baseline in a post-baseline value of a DaT/SPECT SBR measure is greater than 50% or less than -50%, the post-baseline value of the DaT/SPECT measures is considered as physiologically implausible, and therefore will be excluded in the analysis.

#### 5.5.5 Analysis methods

The estimand of the primary analysis for imaging outcome measure is the mean difference of the change from baseline in the imaging measure at Week 52 between treatment groups in the



V1.0

pharmacodynamics population regardless of whether start of PD medication had occurred or not. Specifically, the estimand takes the following into consideration:

- A. Population: pharmacodynamics population as defined in Section 5.1.2;
- B. Variable: change from baseline to Week 52 in the imaging measure;
- C. Intercurrent events: regardless of whether start of PD medication had occurred or not;
- D. Population-level summary: difference in variable means between each active treatment and placebo group

A set of DaT/SPECT measures and have been selected for the statistical anlayses based on literature review and clinical inputs before the DBL. Please see Appendix VI for the listed measures.

Data collected after subjects who have begun taking PD medication will be included in the primary analysis. Change and percent change from baseline will be summarized by visit and treatment groups using descriptive statistics. Change or percent change from baseline in the imaging measures will be analyzed using the mixed model for repeated measures (MMRM), which includes the fixed effect of the treatment group (categorical), time (categorical), interaction between treatment group and time, region (categorical), baseline imaging values (continuous), baseline imaging values by time interaction, baseline MDS-UPDRS I+II+III total score (continuous) and baseline MDS-UPDRS I+II+III total score by time interaction. An unstructured covariance matrix will be used to model the within-subject variancecovariance errors. If the unstructured covariance structure matrix results in a lack of convergence, the heterogeneous Toeplitz covariance structure followed by the heterogeneous first-order autoregressive covariance structure will be used. The Kenward-Roger approximation will be used to estimate the denominator degrees of freedom. Least square means (LSmeans) of each treatment group as well as treatment difference between each BIIB054 groups and placebo will be displayed with 95% CI and p-value at Week 52. If the distribution of the outcome is highly skewed, p-value will be generated from the MMRM model based on the rank data. In the primary analysis, missing data are assumed to be missing at random (Rubin 1976), and the PD medication is assumed to have minimal impact on the imaging measures.

The same MCP-MOD method as used in the primary analyses of MDS-UPDRS I+II+III may be used to assess and model dose-response relationship of the imaging outcomes.

#### 5.5.6 Sensitivity analysis

A sensitivity analysis will be performed using the same MMRM model in the primary analysis, but by excluding DaT/SPECT values that are collected after subjects starting PD medications.

The sensitivity analysis will be performed only for the key DaT/SPECT measures as specified in the Appendix VI.



Placebo-Controlled Period

V1.0

#### 5.5.7 Correlation analysis

Spearman's correlation of change from baseline to Week 52 will be computed for the following imaging and MDS-UPDRS parameters. For the pairs with MDS-UPDRS III, I+II+III and EP-RPS correlation will be computed respectively by including and excluding data after PD medication. For the other pairs, correlation will be computed by including the data after PD medication only.

- DaT-SPECT Striatum total SBR (25. STR SBR) x MDS-UPDRS III
- DaT-SPECT Striatum total SBR (25. STR SBR) x MDS-UPDRS I+II+III
- DaT-SPECT Striatum total SBR (25. STR\_SBR) x Early Parkinson's Regional Progression Score (EP-RPS)
- DaT-SPECT Striatum total SBR (25. STR\_SBR) x structural MRI Striatum total volume (13. STR\_VOL)
- DaT-SPECT Striatum total SBR (25. STR\_SBR) x SNc total volume via GRE (23. GRE NM VOL)
- DaT-SPECT Striatum total SBR (25. STR\_SBR) x SNc total intensity ref 4 via GRE (98. GRE NM NMSIG R4)
- NM-MRI SNc total volume via GRE (23. GRE\_NM\_VOL) x NM-MRI SNc total volume via TSE (9. TSE NM VOL)
- NM-MRI SNc total intensity ref 4 via GRE (98. GRE\_NM\_NMSIG\_R4) x NM-MRI SNc total intensity ref 4 via TSE (37. TSE\_NM\_NMSIG\_R4)





V1.0



#### 5.7 Pharmacokinetics Analysis

The PK analysis population as defined in Section 5.1.2 will be used for the description of the concentration-time profiles and for the estimation of PK parameters.

A serum drug concentration that is deemed inconsistent with dosing (very low or very high) will be excluded from the analysis if no apparent explanation exists. Concentration observations may also be removed from the data set if corresponding dosing or sampling times are missing or cannot be imputed. Concentration data with below limit of quantification value will be excluded. All exclusions of data points or subjects from the analysis will be appropriately documented.

In addition, a detailed listing of sampling time (actual and nominal) and corresponding concentration at each time point for all subjects in the PK population will be provided. Presence of anti-BIIB054 antibody will also be listed and summarized. Additional listings may be generated as deemed necessary.



Placebo-Controlled Period

V1.0

#### 5.7.1 PK Concentration Profile

Descriptive statistics (N, arithmetic mean, standard deviation, geometric mean, CV, median, minimum, maximum, 25<sup>th</sup> and 75<sup>th</sup> percentiles) will be used to summarize concentration of BIIB054 in serum and by visit and treatment groups.

Mean serum concentrations of BIIB054 versus time will be plotted by treatment group on both a linear and a logarithmic scale for Cohort A (doses 1 and 3 only). Dose proportionality will be assessed for Cohort A (doses 1 and 3 only) as deemed appropriate.

Additional listings or plots may be generated as deemed necessary.

#### 5.7.2 Serum PK Parameters

All listed PK parameters below will be computed by non-compartmental methods, as data permits, from serum concentration-time data for cohort A. For cohort B, only C<sub>trough</sub> will be reported, due to sparse PK collection.

| Parameter | Definition/Calculation |
|---|---|
| C <sub>max</sub> | Observed maximum concentration |
| Ctrough | Observed concentration at the end of the dosing interval |
| T <sub>max</sub> | Time to reach maximum concentration |
| AUCtau | area under the concentration-time curve within a dosing |
| | interval tau |
| Accumulation | Using C <sub>max</sub> , C <sub>trough</sub> , and AUC <sub>tau</sub> |
| ratio | |

Individual subject PK parameter data will be listed. Descriptive statistics (N, mean, standard deviation, geometric mean, CV, median, minimum, maximum, 25<sup>th</sup> and 75<sup>th</sup> percentiles) will be used to summarize the PK parameters.

Population PK analysis will be conducted to estimate BIIB054 population PK parameters and to identify potential covariates (e.g., demographics, body weight, anti-BIIB054 mAb etc.) on the variability of BIIB054 PK. In addition, an exposure-response (ER) analysis will be conducted to detect any ER relationship trend and potential covariate using any primary or secondary endpoint and BIIB054 exposure metrics as deemed appropriate. Other tables and figures based on the population PK and ER analyses will be generated by Clinical Pharmacology and Pharmacometrics (CPP) team and will be included in a separate report from CPP.

#### 5.8 Immunogenicity Analysis

#### 5.8.1 Analysis Methods for Immunogenicity Data

Immunogenicity population as defined in Section 5.1.2 will be used to analyze immunogenicity data.



V1.0

For immunogenicity, baseline value is defined as the latest data collected at any time prior to the first dose, or if collected only after dosing the earliest data on the first dose date. More specifically, if samples are only available prior to the first dose, or samples are available both prior to first dose date and on the first dose date, baseline is the latest sample prior to the first dose date. However, if samples are only available on the first dose date but not prior to the first date, baseline is the earliest sample on the first dose date.

A study subject will be given "antibody positive" status if they have at least one confirmed positive sample result at any time during the treatment or post-treatment evaluation periods. A study subject will be given "antibody negative" status if all evaluated antibody sample results are antibody negative.

Anti-BIIB054 antibody responses in antibody-positive subjects are defined as treatment emergent if a subject is:

- ADA-negative at baseline and ADA-positive post-baseline, or
- ADA-positive at baseline and had a greater than 2-fold increase in antibody titer post-baseline.

Summary table of the number and percentage of treatment-emergent anti- BIIB054-positive and -negative antibody events by visit will be displayed for each active treatment groups. A listing of all anti- BIIB054 antibody results will also be provided.

#### **6 INTERIM ANALYSIS**

Safety and PK data only will be reviewed by the IDMC after subjects in Cohort A have completed Week 12 Visit assessments, and before dosing any subjects in Cohort B.

After subjects in Cohort A complete the Week 24 Visit, , all available serum PK,

from Cohort A will be analyzed by a statistical/PK team independent of the study. The grouped level summary statistics will be reviewed only by a limited number of individuals at Biogen who are not involved in the management of the subjects or subject-level data for the study. No changes to the study design are expected based on this review.

For the purpose of planning for future studies, an administrative interim analysis may be performed when approximately 60% of the subjects have completed the Week 52 Visit. A small unblinded team from Biogen, separate from the study management team, will have access to the unblinded interim analysis results. As of the finalization of protocol Version 8 and all subjects have completed Week 52 visits, this analyses was not conducted

A full analysis of the 1-year data will be performed after all subjects have completed the Week 52 Visit. A small unblinded team from Biogen, separate from the study management team, will have access to the unblinded 1-year analysis results. All efficacy endpoints will be analyzed at the Week 52 analyses. All available safety data will also be summarized.

An interim analysis when all subjects have completed the Week 72 Visit is planned to be conducted. A small unblinded team from Biogen, separate from the study management team, will have access to the unblinded interim analysis results. All efficacy endpoints and available will be analyzed at the Week 72 analyses. Selected key safety data (e.g. summary of AE and SAE, summary of MRI safety findings and incidence of anti-drug



V1.0

antibodies) will be summarized, as this is only a snapshort of the safety profile at the time of the Week 72 interim analysis, and the comprehensive safety profile will be presented at the End of Study

A multiple comparison adjustment method will be applied to control the overall type I error at 0.05 in the study, due to the primary endpoint of change from baseline in MDS-UPDRS total score being analyzed at Week 52 and Week 72, and superiority against placebo is considered reached in the study if statistically significant result is achieved at either timepoint at the respective adjusted alpha-level.

An improved fall-back procedure will be used to control the overall type I error at 0.05 level due to multiple-testing. An alpha of 0.04 will be allocated to the Week 52 primary endpoint analyses and an alpha of 0.01 will be allocated to the Week 72 primary endpoint analysis.

- If the Week 52 analysis is statistically significant at the 0.04 level (i.e. p-value ≤0.04), the alpha of 0.04 will be transferred (recycled) to the Week 72 analysis, and Week 72 will have alpha=0.05.
- If the Week 52 analysis is not statistically significant at the 0.04 level, alpha of 0.01 will be used for the Week 72 analysis. Statistically significance is considered achieved if the p-value is ≤0.01 at Week 72.
- If statistically significance is achieved at the Week 72, in either scenarios above, then the alpha of 0.01 will be transferred (recycled) back to Week 52, and the Week 52 primary analysis will be re-evaluated for statistically signifiance at the 0.05 level. This will only change the conclusion of the Week 52 results if the initial p-value is greater than 0.04 and ≤0.05.

No additional multiplicity adjustments will be made for secondary or analyses.

A blinded sample size re-estimation may be conducted when approximately 10% of subjects have completed the Week 52 Visit or approximately 1 month before enrollment is projected to be completed, whichever is earlier (description of method is below). The study sample size may be increased based on this blinded data review. There may be small adjustments to the percentage depending on actual enrollment rate. As of the finaliation of protocol Version 8 (Aug 2020), all subjects have completed Week 52 visits, this analyses was not conducted.

#### Blind sample size re-estimation

The sample size for this study may be reassessed in a blinded manner in a cutoff date of February 2020, by which time approximately 78/311 (25%) of subjects will complete the Week 52 visit.

The standard deviation (SD) of the change from baseline to Week 52 in the putamen ipsilateral side SBR will be estimated based on the blinded data using a modified version of Gould-Shih simple adjustment on sample variance (Zucker et al. 1999):

$$s_{adj}^2 = s_{os}^2 - \frac{2N}{9(N-1)}\delta^2,$$




V1.0

where N denotes the number of subjects included in the analysis for blinded sample size reestimation (subjects with both baseline and Week 52 data of the putamen ipsilateral side SBR available at the time of sample size re-estimation),  $\delta$  is the assumed true treatment effect (same treatment effect assumed for high, medium and low dose group in this analysis), and  $S_{os}^2$  is the unadjusted one sample variance of the estimate of the change from baseline to Week 52 in the putamen ipsilateral side SBR from the pooled blinded data.

The recommendation of sample size increase depends on the comparison of  $s_{adj}^2$  with 0.156, the assumed value of SD for the current sample size (see Section 4). If  $s_{adj}^2$  is less than or equal to 0.156, the value used for sample size calculation when planning the study, the study will continue with the original planned sample size 311. If  $s_{adj}^2$  is greater than 0.156, the study will continue with an increased sample size. The increased sample size will be calculated by using the same MCP-MOD method as specified in Protocol 16.9, subject to a maximum of 413, which is a 30% increase on the original sample size.

#### 7 References

Donald B.Rubin. Inference and missing data. Biometrika. 1976;63: 581-592.

Jose Pinheiro, Bjorn Bornkamp, Ekkehard Glimm and Frank Bretz. Model-based dose finding under model uncertainty using general parametric models. *Statistics in Medicine*. 2013;33: 1646–1661.

Stacy M, Hauser R (2007) Development of a Patient Questionnaire to facilitate recognition of motor and non-motor wearing-off in Parkinson's disease. *J Neural Transm* 114:211–217

Washburn RA, Smith KW, Jette AM, Janney CA. The physical activity scale for the elderly (PASE): Development and evaluation. *Journal of Clinical Epidemiology*. 1993 Feb 1;46(2):153–62.

Christopher G. Goetz, Sheng Luo, Lu Wang, Barbara C. Tilley, Nancy R. LaPelle, Glenn T. Stebbins. Handling Missing Values in the MDS-UPDRS. *Mov Disord. 2015 October; 30(12): 1632-1638*.

K. Horvath, Z. Aschermann, P. Acs, G. Deli, J. Janszky, S. Komoly, E. Balazs, K. Takacs, K. Karadi, N. Kovacs. Minimal clinically important difference on the Motor Examination part of MDS-UPDRS. *Parkinsonism and Related Disorders* 2015. 21: 1421-1426.

K. Horvath, Z. Aschermann, M. Kovacs, A. Makkos, M. Harmat, J. Janszky, S. Komoly, K. Karadi, N. Kovacs. Minimal clinically important difference on the Experiences of Daily Living Parts of Movement Disorder Society-Sponsored Unified Parkinson's Disease Rating Scale. *Movement Disorders* 2017. Vol. 32, No. 5.

L. M. Shulman, A. L. Gruber-Baldini, K. E. Anderson, P. S. Fishman, S. G. Reich, W. J. Weiner. The Clinically Important Difference on the Unified Parkinson's Disease Rating Scale. *Arch Neurol.* 2010; 67 (1): 64-70



V1.0

Zucker, D. M., Wittes, J. T., Schabenberger, O. and Brittain, E. Internal pilot studies II: comparison of various procedures. *Statistics in Medicine*. 1999;18: 3493–3509.

#### 8 Appendix

#### 8.1 Appendix I: Questionnaires

Please refer to the separate Appendix document for the details of the questionnaire as well as the corresponding scoring algorithm.

#### 8.2 Appendix II: Visit Window Mapping

Please refer to the separate Appendix document for the details of the visit window mapping rule for all the study endpoints.

#### 8.3 Appendix III: Description of MCP-MOD method

MCP-MOD method works in the following steps.

#### Step 1: Set of candidate models

Candidate models include Emax (ED50=450.5), Exponential ( $\delta$ =2850.5), logistic (ED50=1547.5,  $\delta$ =510.5), linear-log (off=237.5), quadratic ( $\delta$ =-0.0002), Exponential ( $\delta$ =860.5) and Linear. The response shapes are displayed in Figure 4.1 in the SAP.

#### **Step 2: Optimal model contrast**

The LSmeans at Week 52 and the covariance matrix of the LSmeans will be estimated from the MMRM model and used to determine the optimal contrasts. The coefficients of the contrasts are pre-specified during the design stage once the candidate models are selected in Step 1.

#### **Step 3: Testing for dose response signal**

A multiple contrast test will be used to test the overall dose response signal and to identify all contrasts that have adjusted p-values less than or equal to the pre-specified alpha controlling for multiplicity at Week 52 and Week 72. As a result, the significance of the dose response signal will be established.

#### **Step 4: Model selection**

Value of AIC will be presented together with the p-values for the dose response models in Step 3.



# 8.4 Appendix IV: Definition of the Early Parkinson's Regional Progression Score (EP-RPS)

EP-RPS is derived in the following steps based on MDS-UPDRS Part III motor assessments.

**Step 1:** group the 30 MDS-UPDRS Part III items into 7 body regions as below (item 3.11 of freezing of gait, item of 3.13 of posture and item 3.18 of constancy of rest are excluded.)

| Body region | Question items in UPDRS Part III | Variable names in |
|-------------|--------------------------------------|-------------------|
| | questionnaire | SAS data set |
| Right hand | 3.3b Rigidity-RUE | 3.3b NP3RIGRU |
| | 3.4a Finger Tapping-Right hand | 3.4a NP3FTAPR |
| | 3.5a Hand movements-Right hand | 3.5a NP3HMOVR |
| | 3.6a Pronation-supination movements- | 3.6a NP3PRSPR |
| | Right hand | 3.15a NP3PTRMR |
| | 3.15a Postural tremor-Right hand | 3.16a NP3KTRMR |
| | 3.16a Kinetic tremor-Right hand | 3.17a NP3RTARU |
| | 3.17a Rest tremor amplitude-RUE | |
| Left hand | 3.3c Rigidity-LUE | 3.3c NP3RIGLU |
| | 3.4b Finger Tapping-Left hand | 3.4b NP3FTAPL |
| | 3.5b Hand movements-Left hand | 3.5b NP3HMOVL |
| | 3.6b Pronation-supination movements- | 3.6b NP3PRSPL |
| | Left hand | 3.15b NP3PTRML |
| | 3.15b Postural tremor-Left hand | 3.16b NP3KTRML |
| | 3.16b Kinetic tremor-Left hand | 3.17b NP3RTALU |
| | 3.17b Rest tremor amplitude-LUE | |
| Right leg | 3.3d Rigidity-RLE | 3.3d PN3RIGRL |
| | 3.7a Toe tapping-Right foot | 3.7a NP3TTAPR |
| | 3.8a Leg agility-Right leg | 3.8a NP3LGAGR |
| | 3.17c Rest tremor amplitude-RLE | 3.17c NP3RTARL |
| Left leg | 3.3e Rigidity-LLE | 3.3e NP3RIGLL |
| | 3.7b Toe tapping-Left foot | 3.7b NP3TTAPL |
| | 3.8b Leg agility-Left leg | 3.8b NP3LGAGL |
| | 3.17d Rest tremor amplitude-LLE | 3.17d NP3RTALL |
| Trunk | 3.3a Rigidity-Neck | 3.3a NP3RIGN |
| | 3.9 Arising from chair | 3.9 NP3RISNG |
| | 3.10 Gait | 3.10 NP3GAIT |
| | 3.12 Postural Stability | 3.12 NP3PSTBL |
| | 3.13 Posture | 3.13 NP3POSTR |
| Speech | 3.1 Speech | 3.1 NP3SPCH |
| Face | 3.2 Facial expression | 3.2 NP3FACXP |
| | 3.17e Rest tremor amplitude-Lip/jaw | 3.17e NP3RTALJ |



**Step 2:** For each body region, derive the region score as the maximum score of all the items included in the region. As a result, a score will be derived per subject per visit per body region.

**Step 3:** For each subject at each visit, count the total number of progressed body region. A body region is progressed at visit t if and only if the change from baseline in the body region score is greater than or equal to 1 at visit t, and the change is confirmed by the next visit after visit t. A body region is progressed by visit s, if and only if the body region is progressed prior to or at visit s.

**Step 4:** For each subject at each visit, derive the body region progression AUC as the weighted average of the number of progressed body regions of all the visits before the current visit. The weight of each visit is proportional to the time elapsed from the previous visit to the current visit. Alternatively, the body region progression AUC at visit t can be computed as the area from baseline to visit t under the trajectory curve of the number of progressed body regions by time, divided by the total number of years elapsed from baseline to visit t. Missing data will be imputed by linear interpolation for the intermediate missing visits and by linear extrapolation for the trailing missing visits.

For illustration purpose, suppose a subject had 0, 1, 2, 2, 3, 3 and 4 body regions with progression at Week 8, 16, 24, 32, 40, 48 and 54 visits respectively, then the subject's progression AUC value is as shown in the following plot.

#### Number of progressed body regions over time for a hypothetical patient





V1.0









Placebo-Controlled Period

V1.0





V1.0







#### **Certificate Of Completion**

Envelope Id: 484DE3E88EAA4C7A85354F1CA7E50C1C

Subject: Please DocuSign: 228PD201\_SAP\_Year 1\_v1.0 \_clean.docx

Vendor Name: Source Envelope:

Document Pages: 54 Signatures: 4 Initials: 0 Certificate Pages: 5

AutoNav: Enabled

**Envelopeld Stamping: Disabled** 

Time Zone: (UTC-05:00) Eastern Time (US & Canada)

Status: Completed

**Envelope Originator:** 

#### **Record Tracking**

Status: Original

9/23/2020 5:31:35 PM

Holder:

Location: DocuSign

#### Signer Events

Security Level: Email, Account Authentication

(None)

Signature



Signature Adoption: Pre-selected Style Using IP Address

#### Timestamp

Sent: 9/23/2020 5:35:47 PM Viewed: 9/24/2020 7:45:29 AM Signed: 9/24/2020 7:45:49 AM

#### Electronic Record and Signature Disclosure:

Accepted: 9/24/2020 7:45:29 AM ID: 784a50be-df21-43fb-8f2e-2dd2446fdc86



Biogen

Security Level: Email, Account Authentication

(None)



Signature Adoption: Pre-selected Style

Using IP Address:

Sent: 9/23/2020 5:35:47 PM Viewed: 9/23/2020 5:36:04 PM Signed: 9/23/2020 5:36:10 PM

#### Electronic Record and Signature Disclosure:

Not Offered via DocuSign



Security Level: Email, Account Authentication

(None)



Signature Adoption: Pre-selected Style

Using IP Address:

Sent: 9/23/2020 5:35:48 PM Viewed: 9/24/2020 9:34:00 AM Signed: 9/24/2020 9:34:09 AM

#### **Electronic Record and Signature Disclosure:**

Accepted: 9/24/2020 9:34:00 AM

ID: 1d693b9f-e866-4173-a57c-11d43045c917



Biogen

Security Level: Email, Account Authentication

(None)

Signature Adoption: Pre-selected Style

Using IP Address:

Sent: 9/23/2020 5:35:47 PM Viewed: 9/25/2020 12:27:11 PM Signed: 9/25/2020 12:27:47 PM

## **Electronic Record and Signature Disclosure:**

Not Offered via DocuSign

| In Person Signer Events | Signature | Timestamp |
|---|---|---|
| Editor Delivery Events | Status | Timestamp |
| Agent Delivery Events | Status | Timestamp |
| Intermediary Delivery Events | Status | Timestamp |
| Certified Delivery Events | Status | Timestamp |
| Carbon Copy Events | Status | Timestamp |
| Witness Events | Signature | Timestamp |
| Notary Events | Signature | Timestamp |
| Envelope Summary Events | Status | Timestamps |
| Envelope Sent Certified Delivered Signing Complete Completed | Hashed/Encrypted Security Checked Security Checked Security Checked | 9/23/2020 5:35:48 PM<br>9/25/2020 12:27:11 PM<br>9/25/2020 12:27:47 PM<br>9/25/2020 12:27:47 PM |
| Payment Events | Status | Timestamps |
| <b>Electronic Record and Signature Discl</b> | | |

#### ELECTRONIC RECORD AND SIGNATURE DISCLOSURE

From time to time, Biogen (we, us or Company) may be required by law to provide to you certain written notices or disclosures. Described below are the terms and conditions for providing to you such notices and disclosures electronically through your DocuSign, Inc. (DocuSign) Express user account. Please read the information below carefully and thoroughly, and if you can access this information electronically to your satisfaction and agree to these terms and conditions, please confirm your agreement by clicking the 'I agree' button at the bottom of this document.

#### Getting paper copies

At any time, you may request from us a paper copy of any record provided or made available electronically to you by us. For such copies, as long as you are an authorized user of the DocuSign system you will have the ability to download and print any documents we send to you through your DocuSign user account for a limited period of time (usually 30 days) after such documents are first sent to you. After such time, if you wish for us to send you paper copies of any such documents from our office to you, you will be charged a \$0.00 per-page fee. You may request delivery of such paper copies from us by following the procedure described below.

#### Withdrawing your consent

If you decide to receive notices and disclosures from us electronically, you may at any time change your mind and tell us that thereafter you want to receive required notices and disclosures only in paper format. How you must inform us of your decision to receive future notices and disclosure in paper format and withdraw your consent to receive notices and disclosures electronically is described below.

#### Consequences of changing your mind

If you elect to receive required notices and disclosures only in paper format, it will slow the speed at which we can complete certain steps in transactions with you and delivering services to you because we will need first to send the required notices or disclosures to you in paper format, and then wait until we receive back from you your acknowledgment of your receipt of such paper notices or disclosures. To indicate to us that you are changing your mind, you must withdraw your consent using the DocuSign 'Withdraw Consent' form on the signing page of your DocuSign account. This will indicate to us that you have withdrawn your consent to receive required notices and disclosures electronically from us and you will no longer be able to use your DocuSign Express user account to receive required notices and consents electronically from us or to sign electronically documents from us.

#### All notices and disclosures will be sent to you electronically

Unless you tell us otherwise in accordance with the procedures described herein, we will provide electronically to you through your DocuSign user account all required notices, disclosures, authorizations, acknowledgements, and other documents that are required to be provided or made available to you during the course of our relationship with you. To reduce the chance of you inadvertently not receiving any notice or disclosure, we prefer to provide all of the required notices and disclosures to you by the same method and to the same address that you have given us. Thus, you can receive all the disclosures and notices electronically or in paper format through the paper mail delivery system. If you do not agree with this process, please let us know as described below. Please also see the paragraph immediately above that describes the consequences of your electing not to receive delivery of the notices and disclosures electronically from us.

#### How to contact Biogen:

You may contact us to let us know of your changes as to how we may contact you electronically, to request paper copies of certain information from us, and to withdraw your prior consent to receive notices and disclosures electronically as follows:

To contact us by email send messages to: DL-eSignature@biogen.com

#### To advise Biogen of your new e-mail address

To let us know of a change in your e-mail address where we should send notices and disclosures electronically to you, you must send an email message to us at DL-eSignature@biogen.com and in the body of such request you must state: your previous e-mail address, your new e-mail address. We do not require any other information from you to change your email address.. In addition, you must notify DocuSign, Inc to arrange for your new email address to be reflected in your DocuSign account by following the process for changing e-mail in DocuSign.

#### To request paper copies from Biogen

To request delivery from us of paper copies of the notices and disclosures previously provided by us to you electronically, you must send us an e-mail to DL-eSignature@biogen.com and in the body of such request you must state your e-mail address, full name, Postal address, and telephone number. We will bill you for any fees at that time, if any.

#### To withdraw your consent with Biogen

To inform us that you no longer want to receive future notices and disclosures in electronic format you may:

i. decline to sign a document from within your DocuSign account, and on the subsequent page, select the check-box indicating you wish to withdraw your consent, or you may; ii. send us an e-mail to DL-eSignature@biogen.com and in the body of such request you must state your e-mail, full name, IS Postal Address, telephone number, and account number. We do not need any other information from you to withdraw consent.. The consequences of your withdrawing consent for online documents will be that transactions may take a longer time to process..

#### Required hardware and software

| Here and a final and sold final a | |
|---|---|
| Operating Systems: | Windows2000? or WindowsXP? |
| Browsers (for SENDERS): | Internet Explorer 6.0? or above |
| Browsers (for SIGNERS): | Internet Explorer 6.0?, Mozilla FireFox 1.0, |
| | NetScape 7.2 (or above) |
| Email: | Access to a valid email account |
| Screen Resolution: | 800 x 600 minimum |
| Enabled Security Settings: | •Allow per session cookies |
| | •Users accessing the internet behind a Proxy<br>Server must enable HTTP 1.1 settings via<br>proxy connection |

<sup>\*\*</sup> These minimum requirements are subject to change. If these requirements change, we will provide you with an email message at the email address we have on file for you at that time providing you with the revised hardware and software requirements, at which time you will have the right to withdraw your consent.

#### Acknowledging your access and consent to receive materials electronically

To confirm to us that you can access this information electronically, which will be similar to other electronic notices and disclosures that we will provide to you, please verify that you were able to read this electronic disclosure and that you also were able to print on paper or electronically save this page for your future reference and access or that you were able to e-mail this disclosure and consent to an address where you will be able to print on paper or save it for your future reference and access. Further, if you consent to receiving notices and disclosures exclusively in electronic format on the terms and conditions described above, please let us know by clicking the 'I agree' button below.

By checking the 'I Agree' box, I confirm that:

- I can access and read this Electronic CONSENT TO ELECTRONIC RECEIPT OF ELECTRONIC RECORD AND SIGNATURE DISCLOSURES document; and
- I can print on paper the disclosure or save or send the disclosure to a place where I can print it, for future reference and access; and
- Until or unless I notify Biogen as described above, I consent to receive from exclusively through electronic means all notices, disclosures, authorizations, acknowledgements, and other documents that are required to be provided or made available to me by Biogen during the course of my relationship with you.



Statistical Analysis Plan Dose Blinded Extension Period

V2.0

# **SPARK**228PD201

## Statistical Analysis Plan

**Dose Blinded Extension Period** 



Dose Blinded Extension Period

V2.0

#### STATISTICAL ANALYSIS PLAN **Dose Blinded Extension Period**

**Product Studied: BIIB054** Protocol Number: 228PD201

A Multicenter, Randomized, Double-Blind, Placebo-Controlled Study, with an Active-Treatment Dose-Blinded Period, to Evaluate the Safety, Pharmacokinetics, and Pharmacodynamics of BIIB054 in Subjects with Parkinson's Disease

> **Protocol Version: Version 8.0** Date of Protocol: 11 Aug 2020

Date of Statistical Analysis Plan: 23 June 2021, Final V2.0





#### Statistical Analysis Plan Dose Blinded Extension Period

**V2.0** 

#### **VERSION HISTORY**

| SAP Version | Date | Primary Reasons for<br>Amendment |
|-------------|--------------|-----------------------------------------|
| 1.0 | 25-SEP-2020 | First version of the SAP |
| 2.0 | 23-JUNE-2021 | Update links within sample size section |
| | | Update SMT job titles |



**Dose Blinded Extension Period** 

**V2.0** 

#### **Table of Contents**

| 1 | 1 DESCRIPTION OF OVERALL STUDY (INCLUDING DOSE-BLINDED EXTENSION (DBE)) OBJECTIVES AND ENDPOINTS | |
|---|---|---|
| 2 | STUDY DESIGN | 12 |
| | 2.1 Study Overview | |
| | 2.1.1 Year 1 (Placebo-Controlled Portion of the Study) | |
| | 2.1.2 Years 2-4 (Active-Treatment Dose-Blinded Portion of the Study) | |
| | 2.2 STUDY SCHEMATIC | |
| | 2.3 SCHEDULE OF EVENTS | |
| 3 | SAMPLE SIZE JUSTIFICATION | 15 |
| 4 | STATISTICAL ANALYSIS METHODS | 18 |
| | 4.1 GENERAL CONSIDERATIONS | 18 |
| | 4.1.1 Analysis Population | 20 |
| | 4.1.2 Analyses period | |
| | 4.2 BACKGROUND CHARACTERISTICS | 21 |
| | 4.2.1 Accounting of Subject | 21 |
| | 4.2.2 Demographics and Baseline Characteristics | |
| | 4.2.3 Concomitant Medications and Non-Drug Therapies | |
| | 4.2.4 Protocol Deviations | |
| | 4.2.5 Study Drug Exposure and Study Drug Compliance | |
| | 4.3 EFFICACY ANALYSES | |
| | 4.3.1 General Consideration | |
| | 4.3.2 Primary efficacy endpoint analysis | |
| | 4.3.3 Secondary efficacy endpoints and additional endpoints analysis | 26 |
| | 4.3.3.1 MDS-UPDRS based endpoints | |
| | 4.3.3.2 Other clinical efficacy measures | |
| | 4.5 SAFETY ANALYSES | |
| | 4.5.1 General Considerations. | |
| | 4.5.2 Clinical Adverse Events | |
| | 4,5,2,1 Summary and incidence analysis | |
| | 4.5.2.2 Incidence and incidence rate analysis for active treatment (placebo-controlled and DBE | |
| | 4.5.3 Clinical Laboratory Data | |
| | 4.5.3.1 Quantitative analyses | 32 |
| | 4.5.3.2 Qualitative analyses | |
| | 4.5.4 Vital Sign Data | |
| | 4.5.5 ECG Data | |
| | 4.5.6 Physical and Neurological Examination | |
| | 4.5.7 C-SSRS Data | |
| | 4.5.8 MRI Safety Data | |
| | 4.6 PHARMACODYNAMIC -IMAGING ANALYSIS | |
| | 4.6.1 General Consideration | |
| | 4.6.2 By Visit Summary and MMRM Model | / 3<br>وو |
| | 4.0.3 Additional analyses of placeoo-controlled period due to COVID-19 | 38 |
| | | 38 |
| | 4.8 PHARMACOKINETICS ANALYSIS | |
| | 4.9 IMMUNOGENICITY ANALYSIS | |
| | 4.9.1 Analysis population. | |
| | 4.9.2 Method of analysis | |
| | 4.10 Interim Analyses | |
| _ | ACCECOMENT OF THE IMPACT OF COVID 10 ON STATISTICAL ANALYSES | 40 |



Dose Blinded Extension Period

V2.0

#### LIST OF ABBREVIATIONS

| SI OF ABBREVIAL | |
|---|---|
| 470.4 | |
| ADA | anti-drug antibodies |
| AE | adverse event |
| ALP | alkaline phosphatase |
| ALT | alanine aminotransferase |
| ANCOVA | analysis of covariance |
| APTT | activated partial thromboplastin time |
| AST | aspartate aminotransferase |
| AUC | area under the curve |
| BL | baseline |
| BLQ | below the limit of quantification |
| BMI | body mass index |
| BPM | beats per minute |
| BRP-AUC | body region progression AUC |
| C <sub>max</sub> | observed maximum serum BIIB054 concentration |
| C <sub>min</sub> | observed minimum serum BIIB054 concentration |
| CI | confidence interval |
| CPP | Clinical Pharmacology and Pharmacometrics |
| C-SSRS | Columbia Suicide Severity Rating Scale |
| CTCAT | Common Toxicity Criteria for Adverse Events |
| CV | coefficient of variation |
| DaT | dopamine transporter |
| DaTscan <sup>TM</sup> | Ioflupane I123 radioligand for imaging of dopamine transporter |
| DBE | dose blinded extension |
| DBP | diastolic blood pressure |
| EC <sub>50</sub> | Concentration at 50% of maximum observed biologic effect |
| ECG | electrocardiogram |
| eCRF | electronic case report form |
| EOS | end of study |
| EOT | end of treatment |
| EP-RPS | Early Parkinson's Region Progression Score |
| ER | exposure-response |
| ICF | informed consent form |
| ICH | International Conference on Harmonisation |
| IDMC | independent data monitoring committee |
| INR | International normalized ratio |
| ITT | intent-to-treat |
| IXRS | Interactive Voice/Web Response System |
| LOCF | last observation carried forward |
| Loci | Last coservation earlies forward |



Dose Blinded Extension Period

| T. G | |
|-----------|-------------------------------------------------------------|
| LSmeans | least-square means |
| DBE | Dose-blinded extension |
| IV | intravenous |
| mAb | monoclonal antibody |
| MAO-B | monoamine oxidase type B |
| MCP-MOD | multiple comparison procedure – modeling |
| MDS-UPDRS | Movement Disorder Society Sponsored Revision of the Unified |
| | Parkinson's Disease Rating Scale |
| MedDRA | Medical Dictionary for Regulatory Activities |
| MMRM | mixed-model repeated measures |
| MRI | magnetic resonance imaging |
| PCS | potentially clinically significant |
| PD | Parkinson's disease |
| PK | pharmacokinetic(s) |
| PT | preferred term |
| PP | per-protocol |
| RBC | red blood cell |
| RNA | ribonucleic acid |
| SAE | serious adverse event |
| SAP | statistical analysis plan |
| SBP | systolic blood pressure |
| SBR | striatal binding ratio |
| SD | standard deviation |
| SE | standard error |
| SOC | system organ class |
| SPECT | single-photon emission computed tomography |
| TEAE | treatment-emergent adverse event |
| ULN | upper limit of normal |
| US | United States |
| WBC | white blood cell |
| .,,,,, | |
| WHO | World Health Organization |



## Statistical Analysis Plan Dose Blinded Extension Period

V2.0

Note: This statistical analysis plan (SAP) covers the analyses of the dose-blinded extension (i.e., long terms extension) period (Years 2-4) and the analyses across both the placebo-controlled period and the DBE period (analyses integrating the data for Years 1-4) for study 228PD201. Please refer to the separate SAP for the analyses methods and approaches for placebo-controlled Year 1 period.

#### 1 DESCRIPTION OF OVERALL STUDY (INCLUDING DOSE-BLINDED EXTENSION (DBE)) OBJECTIVES AND ENDPOINTS

The objectives and endpoints of the study are listed below.

The secondary efficacy endpoints have been ranked based on the order of clinical importance.

| Primary Objective | Primary Endpoints |
|---|---|
| To evaluate the clinical efficacy of BIIB054 via dose response using the change from baseline in Movement Disorder Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Total Score | Change from baseline in MDS-UPDRS Total Score (Sum of Parts I, II, and III) at the primary timepoints of Week 52 and Week 72 |
| Secondary Objectives | Secondary Endpoints |
| To evaluate the clinical efficacy of BIIB054 based on MDS-UPDRS subparts | Change from baseline to Week 52 in MDS-UPDRS the subparts III, II and I (each part separately) |
| | Change from baseline to Week 72 and end of study in MDS-UPDRS the subparts III, II and I (each part separately) |
| To assess the PK profile of BIIB054 | Concentration of BIIB054 in the serum |
| To evaluate the dose-related safety of BIIB054 | Incidence of adverse events (AEs) and serious adverse events (SAEs) |
| To evaluate the pharmacodynamic effects of BIIB054 on the integrity of nigrostriatal dopaminergic nerve terminals | Change from baseline to Week 52 in striatal binding ratio (SBR) in the putamen, striatum, and caudate as measured by single-photon emission computed tomography (SPECT) imaging of the dopamine transporter (DaT) with ioflupane I123 (DaTscan <sup>TM</sup> ) |
| To evaluate the immunogenicity of BIIB054 | Incidence and titer of anti-BIIB054 antibodies in the serum |



Dose Blinded Extension Period

| <b>Exploratory Objectives</b> | <b>Exploratory Endpoints</b> |
|-------------------------------|------------------------------|
| Exploratory Objectives | Exploratory Enupoints |
| | • |
| | • |
| | • |
| | ≥ |
| | - |
| | _ |
| | - |
| | • |



Dose Blinded Extension Period





Dose Blinded Extension Period





Dose Blinded Extension Period





## Statistical Analysis Plan Dose Blinded Extension Period

V2.0

#### 2 STUDY DESIGN

#### 2.1 Study Overview

This Phase 2a, randomized, double-blind, parallel-group, placebo-controlled study (Year 1) with an active-treatment dose-blinded period (Year 2 through 4) will examine the efficacy, safety, PK, and pharmacodynamics of BIIB054, administered every 4 weeks via IV infusion to adult subjects with PD. Approximately 311 subjects will be enrolled at about 85 sites globally.

#### 2.1.1 Year 1 (Placebo-Controlled Portion of the Study)

Prior to the first dose in Year 1, all subjects in the study will be randomized into 4 arms, to receive 13 doses of BIIB054 (250, 1250, or 3500 mg) or placebo.

Subjects will be enrolled into 2 cohorts. Cohort A will be randomized first, in a 1:1:1:1 ratio into each of the 4 treatment arm and will include approximately 24 subjects. Randomization and dosing for Cohort B (approximately 287 planned subjects) will start after all subjects in Cohort A complete Week 12 assessments, and all available safety and PK data are reviewed by the IDMC. Randomization of subjects in Cohort B will be stratified by baseline (Day 1) MDS-UPDRS Part I + II + III total scores (≤35 and >35) and striatum SBR (≤1.2 and >1.2), and subjects will be randomized at Day 1 into 1 of 4 parallel dosing arms in each stratum. After all subjects in Cohort A complete Week 12 assessments (28 days after their third infusion), and before dosing any subjects in Cohort B, all available safety and PK data will be reviewed by the IDMC. No subjects in Cohort B may be dosed until the IDMC review is complete. The study schematic is presented in Figure 1. After IDMC review is complete, subjects in Cohort B will be randomized, and dosing may begin. During the review period, subjects in Cohort A will continue to be dosed on a schedule of once every 4 weeks.

The first IDMC meeting will occur after the last subject in Cohort A completes Week 12 assessments, or approximately 6 months after the first subject has been enrolled in Cohort A, whichever comes first. Regular IDMC meetings will occur approximately every 3 months after the first meeting.



Any changes will be documented in a protocol amendment.

#### 2.1.2 Years 2-4 (Active-Treatment Dose-Blinded Portion of the Study)

Prior to Infusion 14 (the first dose of Year 2) at Week 52, subjects who received placebo in Year 1 will be randomized into 1 of the active-dosing arms for Year 2; these subjects will receive BIIB054 in Year 2. Subjects who received BIIB054 (250mg, 1250 mg or 3500 mg) in Year 1 of the study will continue with the same dose regimen in Year 2. Subjects receiving the 250-mg dose in Year 1 continued on their original dose assignment.



## Statistical Analysis Plan Dose Blinded Extension Period

V2.0

Subjects will receive 12 additional doses of BIIB054 (250, 1250, or 3500 mg) in Year 2 and up to 16 additional doses in Years 3 and 4. Up until the last subject in the study has had his or her last dose in Year 2 of the study (Week 96 Visit), eligible subjects will be able to continue treatment once every 4 weeks.

Subjects who complete dosing through Week 96 and the Final Visit 12 weeks after the last visit will be considered Year 2 completers in the eCRF.

See Figure 2 for a depiction of the duration of dosing in Years 3 and 4 for subjects continuing dosing past Week 96.

Figure 4 in the protocol presents a flowchart for dosing and procedures from Week 96 through end of study, including how to determine which subjects are eligible to continue dosing past Week 96.

#### 2.2 Study Schematic

Figure 1: Study Design



DaT = dopamine transporter; IDMC = independent data monitoring committee; PK = pharmacokinetic(s); SPECT = single-photon emission computed tomography

<sup>&</sup>lt;sup>a</sup> Prior to Infusion 14 (first dose of Year 2), subjects who received placebo in Year 1 will be randomized to 1 of the active-treatment groups; these subjects will receive BIIB054 in Year 2. Subjects who received BIIB054 in Year 1 will continue with the same dose regimen in Years 2 through 4. Dosing will continue until the last subject in the study has had his or her Week 96 Visit. Not all subjects will have the opportunity for dosing past Year 2/Week 96.


Figure 2: Overview of Study Dosing:



Q4W = every 4 weeks.

Year 1 = Placebo-controlled period. Years 2 through 4 = Active-treatment dose-blinded period. Not all subjects will have the opportunity for dosing past Year 2/Week 96.



V2.0

#### 2.3 Schedule of Events

See Protocol Section 4.2.

#### 3 SAMPLE SIZE JUSTIFICATION

The sample size calculation is based on changes in MDS-UPDRS Part I + II + III total score at Week 52 and at Week 72 of treatment. Based on data from the Parkinson's Progression Markers Initiative study, the placebo subject's mean and standard deviation (SD) at Week 52 and Week 72 are assumed to be 8.0 (10.64) and 9.6 (13.7) respectively. Assuming a maximum of 55% reduction in the change from baseline in the active group with maximum response relative to placebo group, the mean (SD) for this active group will be 3.2 (10.64) and 3.84 (13.7) respectively at Week 52 and Week 72, and the responses for other active groups are assumed to be somewhere between 0 and the maximum response. The primary analysis will be based on the MCP-MOD method to detect a dose-response trend while controlling for multiplicity. Optimal contrasts will be constructed to detect potential doseresponse trend under common dose-response curves (e.g., E<sub>max</sub>, exponential, logistic, linear in log dose, and quadratic model, which are illustrated with parameters shown in Figure 3.1 which will be used for both Week 52 and Week 72). The planned enrollment is 311 subjects total (24 subjects in Cohort A and 287 subjects in Cohort B, 3.1). Actual enrollment is 357 subjects. In Cohort A, 29 subjects were randomized in a 1:1:1:1 ratio to each of the treatment groups, while in Cohort B 328 subjects were randomized in 2:1:2:2 ratio to the placebo, 250 mg, 1250 mg, and 3500 mg groups. Based on the actual enrollment, the estimated number of subjects by cohort and treatment groups are given in Table 3.2 below. After accounting for dropout rate of 10% and 15% at Week 52 and Week 72, respectively, the estimated sample sizes are given in Table 3.3 and Table 3.4. With the updated sample size, the study will provide an average power of approximately 80% to detect the dose-response trend over 1 year of treatment, based on a 2-sided type I error of 0.05 and approximately 73% of power at the Week 72 analyses, based on a 2-sided type I error of 0.05. Overall, the sample size in the study will provide approximately 89% power, taking into consideration success at either Week 52 or Week 72.

With an estimated sample size of 100 subjects dosed per arm in the 1250 mg and 3500 mg arms, the study has 80% probability of detecting AEs with a rate of 1.6% or greater in these 2 arms, and a 90% probability of detecting AEs occurring with a rate of 2.3% or greater.



V2.0

Figure 3.1: Candidate Models for Dose-Response





## Statistical Analysis Plan

**Dose Blinded Extension Period** 

V2.0

**Table 3.1: Estimated Sample Size Per Group (Planned)** 

| | Treatment Group | | | | |
|----------|-----------------|--------|---------|---------|-----|
| | Placebo | | | | |
| Cohort | | 250 mg | 1250 mg | 3500 mg | |
| Cohort A | 6 | 6 | 6 | 6 | 24 |
| Cohort B | 82 | 41 | 82 | 82 | 287 |
| Total | 88 | 47 | 88 | 88 | 311 |

**Table 3.2: Estimated Sample Size Per Group Based on Actual Enrollment** (Before Drop-Outs)

| | Treatment Group | | | | |
|----------|-----------------|--------|---------|---------|-----|
| | Placebo | | | | |
| Cohort | | 250 mg | 1250 mg | 3500 mg | |
| Cohort A | 8 | 7 | 7 | 7 | 29 |
| Cohort B | 93 | 47 | 94 | 94 | 328 |
| Total | 101 | 54 | 101 | 101 | 357 |

**Table 3.3:** Estimated Sample Size Per Group Based on Actual Enrollment (After Adjusting for 10% Drop-Out At Week 52

| | Treatment Group | | | | |
|----------|-----------------|--------|---------|---------|-----|
| | Placebo | | | | |
| Cohort | | 250 mg | 1250 mg | 3500 mg | |
| Cohort A | 7 | 6 | 6 | 6 | 25 |
| Cohort B | 84 | 42 | 84 | 84 | 294 |
| Total | 91 | 48 | 90 | 90 | 319 |

**Table 3.4:** Estimated Sample Size Per Group Based on Actual Enrollment (After Adjusting for 15% Drop-Out At Week 72

| | Treatment Group | | | | |
|----------|-----------------|--------|---------|---------|-----|
| | Placebo | | | | |
| Cohort | | 250 mg | 1250 mg | 3500 mg | |
| Cohort A | 7 | 6 | 6 | 6 | 25 |
| Cohort B | 79 | 40 | 80 | 80 | 279 |
| Total | 86 | 46 | 86 | 86 | 304 |




V2.0

#### 4 STATISTICAL ANALYSIS METHODS

#### 4.1 General Considerations

This statistical analysis plan (SAP) covers the analyses of the dose-blinded extension (i.e., long term extension) period (Years 2-4) and the analyses across both the placebo-controlled period and the DBE period (analyses integrating the data for Years 1-4).

Summary tables will be presented using descriptive summary statistics. For continuous variables, summary statistics will generally include number of subjects with data, mean, standard deviation, median, 25% percentile, 75% percentile, minimum and maximum. For categorical variables, this will generally include number of subjects randomized or dosed, number with data, and the percent of those with data in each category. Pharmacokinetics (PK) summaries will also include Geometric mean and geometric CV.

Statistical testing will be performed to assess efficacy endpoints by conducting pairwise comparison between each BIIB054 group and the delayed-start group (i.e. subjects who were randomized to placebo in Year-1),. Dose-response relationship may also be tested. Unless stated otherwise, all the statistical tests will be 2-sided with a statistical significance level of 0.05.

The statistical software, SAS® will be used for all summaries and analyses.

#### Analysis displays

Unless otherwise specified, the analysis of the DBE period and the analyses across both the placebo-controlled period and the DBE period will be displayed by DBE treatment groups as shown below, separate for early and delayed start treatment group) including tables, listings and figures, unless otherwise specified.

Unless otherwise specified, analyses for efficacy data (e.g., pharmacodynamics of imaging, clinical efficacy, displayed by the following treatment groups according to randomization assignment at the start of the placebo-controlled period:

- BIIB054 early start: subjects who are assigned to (1) receive BIIB054 in the placebo-controlled period and (2) continue receiving BIIB054 in the DBE period
- BIIB054 late start: subjects who are assigned to (1) receive placebo in the placebo-controlled period and (2) switch to BIIB054 in the DBE period

Unless otherwise specified, analyses for safety, PK, and ADA data will be displayed by the following treatment groups according to dose received:

• BIIB054 early start: subjects who receive BIIB054 in the placebo-controlled period (regardless of randomization assignment)



V2.0

- BIIB054 late start: subjects who receive only placebo in the placebo-controlled period (regardless of randomization assignment) and switch to receive BIIB054 in the DBE period
- BIIB054 total: subjects in either BIIB054 early or late start treatment groups

.

If all subjects received study treatment according to their randomization assignments during the placebo-controlled period (i.e. no subject assigned to placebo received BIIB054, and no subject assigned to BIIB054 received only placebo), then the assignment of subjects to treatment groups in efficacy related tables will be the same as those in safety related tables.

For efficacy, pharmacodynamic of imaging, and PK and ADA outcomes. Each BIIB054 early start dose group may be compared with the corresponding delay-start dose group, as well as the pooled delay-start group. Outputs will be presented in the following two ways:

| | BIIB054 delayed start | | | BIIB054 early start | |
|---|---|---|---|---|---|
| (N = xx) | | (N = xx) | | | |
| Placebo to $250 \text{ mg}$ $(N = xx)$ | Placebo to $1250 \text{mg}$ $(N = xx)$ | Placebo to $3500 \text{ mg}$ $(N = xx)$ | 250 mg $(N = xx)$ | 1250 mg $(N = xx)$ | 3500 mg $(N = xx)$ |

| BIIB054 delayed start | BIIB054 early start | | |
|-----------------------|---------------------|----------|----------|
| (N = xx) | (N = xx) | | |
| Placebo to BIIB054 | 250 mg | 1250 mg | 3500 mg |
| (N = xx) | (N = xx) | (N = xx) | (N = xx) |

#### For baseline and safety related outputs:

| BIIB054 delayed start | | BIIB054 early start | | | | BIIB054 | |
|---|---|---|---|---|---|---|---|
| (N = xx) | | (N = xx) | | | | Total | |
| Placebo Placebo to 250 to mg 1250mg $(N = xx)$ $(N = xx)$ | Placebo<br>to 3500<br>mg<br>(N = xx) | Total<br>(N=xx) | 250 mg $(N = xx)$ | 1250 mg $(N = xx)$ | 3500 mg $(N = xx)$ | Total<br>(N=xx) | (N=xx) |

For all listings the start and stop day in the listing will be computed based on the placebocontrolled baseline.

Baseline for all the analyses across the SAP

Unless otherwise specified, baseline refers to the baseline value for the placebo-controlled period and is defined as the most recent non-missing measurement collected prior to the first CONFIDENTIAL



V2.0

dose in Year 1. DBE baseline is defined as the last non-missing measurement collected prior to the first dose of the DBE period in Year 2.

For analyses on the DBE period or on the active treatment (placebo-controlled and DBE) period, DBE baseline will be used for delayed start subjects who are assigned to receiving BIIB054 in the DBE period. Change from baseline will be defined as post-baseline value minus baseline value.

#### 4.1.1 Analysis Population

- Intent-to-treat (ITT) population:
  The Intent-to-treat population is defined as all randomized subjects who received at least one dose of study treatment (BIIB054 or placebo).
- Safety population:
   The safety population is defined as all subjects who received at least one dose of study treatment (BIIB054 or placebo).
- Pharmacodynamic analysis population:
  The pharmacodynamic population is defined as a subset of the ITT population with at least 1 post-baseline pharmacodynamic measurement.
- PK analysis population:
   The PK population is defined as a subset of the ITT population who have at least 1 measurable BIIB054 concentration in serum
- Immunogenicity population:
   Immunogenicity analysis will be performed for all subjects in the safety population.

#### 4.1.2 Analyses period

Depending on the purpose, different analyses will be conducted on the following study periods:

- 1. DBE period. Only data in the DBE period will be included in these analyses. For example, incidence table of adverse events in the DBE period.
- Placebo-controlled and DBE period. All the data in the placebo-controlled and DBE periods will be included in these analyses. For example, mean plot of actual laboratory values in the placebo-controlled and DBE period.



V2.0

3. Active treatment (placebo-controlled and DBE) period (i.e., Total BIIB054 experience) period. Active treatment period is defined as the study period(s) that a subject is assigned to BIIB054. For early start subjects – subjects who are assigned to BIIB054 in both placebo-controlled and DBE period, all the data (placebo-controlled and DBE periods) will be included in the analyses. For delayed start subjects – subjects who are assigned to placebo in Year 1 and BIIB054 in the DBE period, only data in the DBE period will be included. For example, incidence table of adverse events in the active treatment (placebo-controlled and DBE) period will not include the AEs started on placebo treatment in year 1.

Subjects to be included in a certain output is determined by both the analysis population and the analysis period. For example, the incidence table of adverse events in the DBE period will include subjects in the safety population for the DBE period, i.e., all randomized subjects who received at least one dose of study treatment in the DBE period. The incidence table of adverse events in the active treatment (placebo-controlled and DBE) period will include subjects in the safety population for the active treatment period, i.e., all randomized subjects who received at least one dose of study treatment in the active treatment period. In this SAP we do not separately define the analysis population in each analysis period.

#### 4.2 Background Characteristics

The summaries in this section will be based on the ITT population. Analysis period will be specified for each table or figure. Unless otherwise specified, summary tables will be presented by DBE treatment group. Listings will include all data in the placebo-controlled and DBE periods (all data in the study), with an indicator of the study period in a column (pre-dosing, placebo-controlled, or DBE) for each record to indicate when the event occurred. Listings will be presented by DBE treatment group.

#### 4.2.1 Accounting of Subject

Disposition in the DBE period will be summarized for subjects enrolled in DBE. The summary data will include number (%) of subjects dosed in the DBE period, number (%) of subjects who completed the first year of treatment/study of DBE (i.e., year 2 of the study), number (%) of subject who discontinued treatment and/or withdrew from study in the first year of DBE (i.e., year 2 of the study), the reason for treatment discontinuation and/or study withdrawal for in the first year of DBE (i.e., year 2 of the study), number (%) of subjects who completed the treatment/study in DBE (i.e., year 2-4 of the study), and number (%) of subjects who discontinued treatment and/or withdrew from study in DBE (i.e., year 2-4 of the study), the reason for treatment discontinuation and/or study withdrawal in DBE (i.e., year 2-4 of the study).

For subject who discontinued treatment and/or withdrew from the study in the first year of DBE (i.e., year 2 of the study), days on treatment and days on study will be summarized.

For subjects who discontinued treatment and/or withdrew from study in DBE (i.e., year 2-4 of the study), days on treatment and days on study will be summarized and listed. In the listing, the subjects who discontinued treatment and/or withdrew from study in the first year




V2.0

of DBE will be flagged. Time to treatment discontinuation and time to study withdrawal in the DBE period may be displayed by Kaplan-Meier plot (presented by DBE treatment group).

Disposition in the placebo-controlled and DBE period will be also summarized in the same fashion. Number (%) of subjects dosed in the placebo-controlled period, number (%) subject who completed the placebo-controlled period, number (%) of subjects who entered the DBE period, number (%) of subjects who completed the first year of DBE period, number (%) of subjects who completed the whole study will be displayed. Number of subjects who discontinued treatment or study and reason of discontinuation will be summarized for each period and for the whole study.

#### 4.2.2 Demographics and Baseline Characteristics

Demographics, baseline characteristics, medical history and PD treatment history will be summarized for subjects enrolled in the DBE period and subjects not enrolled in the DBE period, respectively. Please refer to the SAP of placebo-controlled period for more details.

#### 4.2.3 Concomitant Medications and Non-Drug Therapies

All medications will be coded using the World Health Organization Drug (WHODrug March 2020 B3 or higher) dictionary. All non-drug therapies (defined as diagnostic procedures or medical treatment procedures) will be coded using the MedDRA dictionary version 23.0 or higher.

The number (%) of subjects taking concomitant general medication (excluding PD medications) and non-drug therapies in the DBE period will be summarized by DBE treatment group for subjects enrolled in the DBE period. In addition, number of subjects in the ITT population that have taken any concomitant medications in the active treatment (placebo-controlled and DBE) period will be summarized. Concomitant non-PD medications and non-drug therapies will be listed in the placebo-controlled and DBE treatment period. Start and stop day in the listing will be computed based on the placebo-controlled baseline.

For subjects enrolled in the DBE period, the number (%) of subjects taking any concomitant PD symptomatic medications, number of subjects taking Dopamine, MAO-B inhibitor, Dopamine Agonist at the baseline of the placebo-controlled period and at the baseline of DBE period will be summarized respectively by DBE treatment group. The placebo-controlled and DBE period data will be summarized in the same fashion. Concomitant PD symptomatic medication will be listed for all subjects in the placebo-controlled and DBE periods. Start and stop day in the listing will be computed based on the placebo-controlled baseline. Please refer to the placebo-controlled SAP for definitions of concomitant therapies and PD symptomatic medication use at baseline.

#### 4.2.4 Protocol Deviations

Protocol deviations identified during site monitoring will be captured in a Protocol Deviation log and categorized as major or minor deviations. The major protocol deviations occurred in CONFIDENTIAL



V2.0

the DBE period will be summarized for subjects enrolled in DBE. The major protocol deviations for all ITT subjects in the combined placebo-controlled and DBE periods will also be summarized. Major and minor protocol deviations for all ITT subjects will be listed, respectively, across the placebo-controlled period and the DBE period. All summaries for protocol deviations will be presented by DBE treatment group. A separate Covid-19 related protocol deviation category will be shown in the protocol deviation listings.

#### 4.2.5 Study Drug Exposure and Study Drug Compliance

A summary table of study drug exposure and compliance in the DBE period will be provided. Number of infusions of BIIB054 received will be summarized as a continuous variable as well as a categorical variable (categories as 1-5, 6-10 and 11-15, 16-20, 20-25, >=26) as well as a continuous variable. Number of weeks on study treatment, calculated as (date of last dose – date of first dose +1)/7, will be summarized as a categorical variable (categories as <0.5 years, >=0.5 years, >=1 year, >=2 years, >=3 years) as well as a continuous variable. Percentage of study treatment taken up to the last dose, calculated as (the actual number of infusions / the number of infusions a subject is expected to take until the date of last infusion)\*100, will be summarized as a continuous variable. This table will be presented by DBE treatment group. A similar table will also be provided on the active treatment (placebocontrolled and DBE) period in order to summarize the exposure data while subjects are on BIIB054.

A listing of study drug administration records, including infusion start date and time, infusion stop date and time, total volume prepared, total volume administered, location of infusion, initial infusion rate, dose interruption or rate change or not, time of interruption or rate change, infusion rate after interruption or rate change, reason for interruption or rate change will be provided for the placebo-controlled and DBE period. A listing of subjects who received the wrong treatment compared to what they were randomized to will be provided for the placebo-controlled and DBE period.

#### 4.3 Efficacy analyses

#### 4.3.1 General Consideration

The analysis population for the efficacy analyses are defined in Section 4.2.1. The analysis period includes data from both placebo-controlled and DBE period combined. That is, data from both the placebo-controlled and DBE periods will be included in the analysis.

The following three comparisons will be evaluated for the long-term efficacy analyses of BIIB054:

- The early start 250 mg compared with the pooled delayed start group;
- The early start 1250 mg compared with the pooled delayed start group;
- The early start 3500 mg compared with the pooled delayed start group

The following comparisons may also be evaluated:

• The early start 250 mg compared with the delayed start 250 mg;



V2.0

- The early start 1250 mg compared with the delayed start 1250 mg.
- The early start 3500 mg compared with the delayed start 3500 mg.

The pooled delayed start group contains all the subjects who were randomized to placebo treatment in the placebo-controlled period including those who did and who did not enter into the DBE period. There will be no multiple comparison adjustments. Data after subjects start PD symptomatic treatment will be included in the analyses, since the majority of subjects are expected to take PD medication after Week 52.

Subjects who were randomized to placebo group but accidentally received one or more doses of the active treatment during the placebo-controlled period will be classified as delayed start for all the efficacy, pharmacodynamic, and analyses.

#### Visit Windows for by visit analyses

For the by visit summaries and MMRM models, the analysis visit should be defined using visit windows (see Tables 6-16 in the Appendix). If there is more than 1 value in the same analysis visit window (>1 value for the same analysis visit) for a certain parameter for a subject, then the closest record to the target visit day will be used for the by visit analysis. If they are with the same distance from the target visit day, then the record with the later time will be used for the by visit analysis.

#### Handling of missing items for scales

Please refer to the placebo-controlled SAP for the imputation method. The same method will be applied to efficacy endpoints collected in the DBE period.

#### 4.3.2 Primary efficacy endpoint analysis

The estimand of the primary analysis for MDS-UPDRS Part I+II+III total score at Week 72 is the mean difference of the change from baseline at Week 72 between treatment groups in the ITT population regardless of whether start of PD medication had occurred or not. Specifically, the estimand takes the following into consideration:

- A. Population: ITT population as defined in Section 4.1.1;
- B. Variable: change from baseline to Week 72 in the MDS-UPDRS Part I+II+III total score:
- C. Intercurrent events: regardless of whether start of PD medication had occurred or not;
- D. Population-level summary: difference in variable means between each early start group and delayed start group

Change from baseline in the MDS-UPDRS Part I+II+III total score at Week 72 will be analyzed using an MMRM model for all the visits in the placebo-controlled and DBE period.

Data after subjects start PD medication will be included in the primary analyses.

For details on the model to be used please refer back to the Year 1 SAP, for the analyses of MDS-UPDRS including data after PD medication. Adjusted means for each treatment group, CONFIDENTIAL



V2.0

pairwise adjusted differences for the comparisons, 95% confidence intervals for the differences will be presented at each visit, and p-values will be presented for the key visits of week 24, 52, and 72. Dose-response testing will be done using the adjusted mean with the pre-specified MCP-MOD procedure with pre-specified candidate models (refer to Year 1 SAP Sample Size Consideration section). If the distribution of the outcome is highly skewed, p-value will be generated from the MMRM model based on the rank data. Missing data are assumed to be missing at random behind the MMRM model.

A multiple comparison adjustment method (graphical procedure) will be applied to control the overall type I error at 0.05 in the study, due to the primary endpoint of MDS-UPDRS total score being analyzed at Week 52 and Week 72, and superiority against placebo is considered reached in study if statistically significant result is achieved at either timepoint. Please refer to the "Interim Analysis" section for this method. Pairwise comparison of each active group versus delayed-start group(s) will also be conducted, however, no additional multiplicity adjustment will be made, and nominal p-values will be reported. The primary comparison is between each of the early-start BIIB054 dose group, with the pooled delayed-start BIIB054 group.

The following three comparisons will be evaluated for the long-term efficacy analyses of BIIB054:

- The early start 250 mg compared with the pooled delayed start group;
- The early start 1250 mg compared with the pooled delayed start group;
- The early start 3500 mg compared with the pooled delayed start group

The following comparisons may also be evaluated:

- The early start 250 mg compared with the delayed start 250 mg;
- The early start 1250 mg compared with the delayed start 1250 mg.
- The early start 3500 mg compared with the delayed start 3500 mg.

Per design, a subset of subjects will enter year 3 and 4 for a limited time. There will be some visits with too few data in year 3 and 4. If this is the case, the visits with too few data will be excluded from the MMRM analyses, Otherwise, the MMRM model will not converge. In addition, since most patients will start PD medication by year 1, most data in year 2-4 will be after PD medication. Therefore, data after subject start PD medication will be included in the MMRM analyses. Otherwise, the MMRM model will not converge.

Data at the common visits of cohort A and cohort B will be included in the by visit summary and MMRM model. Data at all visits will be listed.



V2.0

#### 4.3.3 Secondary efficacy endpoints and additional endpoints analysis

Secondary endpoints, e.g., change from baseline in the MDS-UPDRS subscores (e.g., Part I, II, or III score, Part II and III total score) will be analyzed in a similar model, but no additional multiplicity adjustment will be made or for other secondary endpoints.

#### 4.3.3.1 MDS-UPDRS based endpoints

The analysis approaches and the MMRM model described will be performed for additional MDS-UPDRS based endpoints as listed below, except that, 1) the baseline MDS-UPDRS total score term in the model will be replaced by the corresponding baseline value of MDS-UPDRS total or sub-part score being analyzed, 2) MCP-MOD dose-response may be performed, 3) no additional multiple comparison adjustment will be applied for secondary efficacy and exploratory efficacy endpoints

- MDS-UPDRS Parts I, II, III (Secondary Efficacy Endpoints),
- MDS-UPDRS Total Score (I+II+III) at the end of the study
- MDS-UPDRS Parts II+III, Ib+II+III
- MDS-UPDRS Part IV
- Postural Instability -Gait Difficulty (PIGD) score (mean score of MDS-UPDRS items 2.12+2.13+3.10+3.11+3.12),
- Lower Extremity (LE) score (mean score of MDS-UPDRS items 3.10+3.11+3.12+3.13+3.3d+3.3e+3.7a+3.7b +3.8a+3.8b+3.17c+3.17d+2.12+2.13), and Tremor score (mean score of MDS-UPDRS items 2.10+3.15a+3.15b+3.16a+3.16b+3.17a+3.17b+3.17c+3.17d+3.17e+3.18).

#### 4.3.3.2 Other clinical efficacy measures





V2.0



#### 4.4 Pharmacodynamics analyses

There are three types of imaging outcomes in the study: DaT/SPECT imaging,

Please refer to the placebo-controlled SAP for details.

The analysis population for pharmacodynamic analyses is defined in Section 3.1.1. The analysis period is placebo-controlled and DBE period combined. That is, data from both the placebo-controlled and DBE periods will be included in the analyses.

Similar analyses will be conducted for the pharmacodynamic analyses as for the clinical outcome analysis. The main comparison will be between the early and delayed-start groups. The pooled delayed start group contains all the subjects who were randomized to placebo treatment in the placebo-controlled period including those who did and who did not enter to the DBE period. There will be no multiple comparison adjustments. Data after subjects start PD symptomatic treatment will be included in the analyses.

Visit Windows for by visit analyses



V2.0

For the by visit summaries and MMRM models, the analysis visit should be defined using visit windows (see Table 3 in the Appendix). If there is more than 1 value in the same analysis visit window (>1 value for the same analysis visit) for a certain parameter for a subject, then the closest record to the target visit day will be used for the by visit analysis. If they are with the same distance from the target visit day, then the record with the later time will be used for the by visit analysis.

A prespecified set of imaging measures as well as the change from baseline will be summarized by DBE treatment groups by visit for all the visits in the placebo-controlled and DBE period.

#### MMRM model analyses:

Similar MMRM model will be used to conduct the pharmacodynamic analyses as for the clinical outcome analysis, with the same terms included in the model.

#### 4.5 Safety Analyses

#### 4.5.1 General Considerations

#### Analysis population

Safety population will be used for safety analyses of AEs, clinical laboratory data, vital sign data, ECG data, physical and neurological examination findings, Columbia Suicide Severity Rating Scale (C-SSRS) data and MRI safety data.

#### DBE safety treatment groups

Please refer to Section 3.1 for the safety treatment groups. Subjects who were randomized to placebo group but accidentally received one or more doses of BIIB054 during the placebo-controlled period will be classified as early start for all the safety analyses that involves DBE, and their applicable safety data in the placebo-controlled period will be included in the analysis for active treatment (placebo-controlled and DBE) period.

#### Safety analysis period

Analysis period will be specified for each output. Analyses periods in this SAP are

- Long-term extension period for AE analyses
- Active treatment (placebo-controlled and DBE) period for AE analyses and analyses of hematology/blood chemistry/urinalysis, hepatotoxicity, vital sign, ECG, MRI.

Safety data in the specified analysis period will be included in the analysis. Listings will include all data in the placebo-controlled and DBE period, unless otherwise specified.

#### Incidence, incidence proportion and incidence rate

• Incidence and incidence proportion will be provided in incidence tables. Incidence is defined as the number of subjects who experienced an event. Incidence proportion is CONFIDENTIAL



V2.0

defined as the number of subjects who experienced an event divided by the total number of subjects in the analysis population, i.e., percentage. Each subject will be counted only once within each category.

• Incidence and incidence rate will be provided in incidence rate tables. Incidence rate is defined as the number of subjects who experienced an event divided by the total follow-up time among the subjects in the analysis population (e.g., incidence rate per 100 subject-years). The total follow-up time is the sum of all subjects' follow-up time. The follow-up time for a subject is defined as the number of days (inclusive) from the first dose of treatment until the last day on study divided by 365.25. For active treatment (placebo-controlled and DBE) period analyses, the first dose of treatment is considered as the first dose received in the study period (PC or OLE) in which a subject first receives BIIB054. Each subject will be counted only once within each category.

#### 4.5.2 Clinical Adverse Events

Treatment emergent AEs (TEAEs)

All AEs will be coded using the MedDRA dictionary version 23.0 or higher.

All AEs will be analyzed based on the principle of treatment emergence. A treatment emergent AE is defined as an AE that started or worsened after the start of first infusion of study treatment.

To define treatment emergence for AEs with missing start or stop date or time the following additional criteria will be used:

- if both the start and stop dates for a particular AE are missing, then that AE is considered treatment emergent.
- if the start date for a particular AE is missing and the stop date/time falls after the first dose date/time, then that AE is considered treatment emergent.
- if the start date for a particular AE was the same as the first dose date, and the start time was missing, then that event is considered treatment emergent.

For AEs with a partial start date, the year/month of the event date will be compared to that of the first dosing date to determine whether the event is treatment emergent.

In addition, SAEs that occurred since a subject was screened in the study and prior to the first infusion of study treatment, which by definition are not treatment emergent, will be analyzed separately.

Only TEAEs will be included in the AE tables, unless otherwise specified. Listings of AEs will include all events, whether treatment emergent or not.

#### 4.5.2.1 Summary and incidence analysis

Overall summary of AE table will be done for the following periods, by DBE treatment groups:

• DBE period, and,



V2.0

• the active treatment (placebo-controlled and DBE) period

The following information will be summarized: the number of subjects with any AE, with any AE by maximum severity, with any related AE (related to study drug as assessed by investigator), with radioligand rated AE, with SAE, with related SAE, with radioligand rated SAE, with AE leading to study drug discontinuation, with AE leading to study withdrawal and the number of deaths.

The sorting order of AE incidence tables, unless otherwise specified, will be by decreasing frequency order of "BIIB054 total" column within each category in the tables presented by DBE treatment group. A subject is counted only once within each category in each table. For example, for the table of AEs by system organ class and preferred terms sorted by decreasing frequency presented by DBE treatment group, system organ class will be presented in decreasing frequency order of BIIB054 total column, and within each system organ class, preferred terms will be presented in decreasing frequency order of BIIB054 total column. A subject is counted only once within each system organ class and preferred term.

The severity of AEs and SAEs is graded using the CTCAE grade, version 5.0. The categorisation of severity is as follows: grade 1 (mild), 2 (moderate), 3 (severe or medically significant), 4 (life-threatening) and 5 (death), Severe AEs and SAEs are classed as CTCAE grade >=3.

The following AE incidence tables will be provided for the DBE period:

- 1. AEs by system organ class and preferred term sorted by decreasing frequency
- 2. AEs by preferred term
- 3. Severe AEs by system organ class and preferred term
- 4. Severe AEs by preferred term
- 5. Study drug related AEs by system organ class and preferred term
- 6. SAEs by system organ class and preferred term sorted by decreasing frequency
- 7. SAEs by preferred term
- 8. Study drug related SAEs by system organ class and preferred term
- 9. AEs that led to discontinuation of study treatment by system organ class and preferred term
- 10. AEs that led to withdrawal from study by system organ class and preferred term

## 4.5.2.2 Incidence and incidence rate analysis for active treatment (placebo-controlled and DBE) period

Due to the different length of active treatment (placebo-controlled and DBE) period in early start versus delayed start subjects, both incidence (proportion) tables and incidence rate tables will be used for AE analyses in this period. The entire follow-up time is from the first dose in



V2.0

active treatment period (first dose in placebo-controlled period for early start subjects and first dose in DBE period for delayed start subjects) until the last day in the study.

The following incidence (proportion) will be provided for the active treatment (placebo-controlled and DBE) period. The follow-up adjusted incidence rate table will be provided for 1, 10, 12, 14, 16 and 17.

- 1. AEs by system organ class and preferred term sorted by decreasing frequency
- 2. AEs by system organ class and preferred term sorted by alphabetical order analysis
- 3. AEs by system organ class
- 4. AEs by preferred term
- 5. AEs with an incidence of 5% or more in any treatment group by preferred term
- 6. Severe AEs by system organ class and preferred term
- 7. Severe AEs by preferred term
- 8. AEs by maximum severity by system organ class and preferred term (System organ class will be presented alphabetically. Preferred term will be presented in decreasing frequency order.
- 9. AEs by maximum severity by preferred term (Preferred term will be presented in decreasing frequency order)
- 10. Study drug related AEs by system organ class and preferred term
- 11. Radioligand related AEs by system organ class and preferred term
- 12. SAEs by system organ class and preferred term
- 13. SAEs by preferred term
- 14. Study drug related SAEs by system organ class and preferred term
- 15. Radioligand related SAEs by system organ class and preferred term
- 16. AEs that led to discontinuation of study treatment by system organ class and preferred term
- 17. AEs that led to withdrawal from study by system organ class and preferred term
- 18. AEs that occurred within 2 hours from infusion start by system organ class and preferred term

The following listings will be provided for the placebo-controlled and DBE period:

- 1. Listing of AEs
- 2. Listing of SAEs
- 3. Listing of AEs that led to discontinuation of study treatment
- 4. Listing of AEs that led to withdrawal from study
- 5. Listing of AEs that occurred within 2 hours from infusion start
- 6. Listing of study drug related AEs
- 7. Listing of radioligand related AEs

#### CONFIDENTIAL



V2.0

8. Listing of deaths

#### 4.5.3 Clinical Laboratory Data

The following laboratory assessments will be performed in Year 2-4 to evaluate the safety profile of BIIB054:

- Hematology: Complete blood count with differential and platelet count, INR, PT, and APTT
- Blood chemistry: total protein, albumin, creatinine, blood urea nitrogen, uric acid, bilirubin (total and direct), alkaline phosphatase, alanine aminotransferase, aspartate aminotransferase, gamma-glutamyl transferase, glucose, calcium, phosphorus, bicarbonate, chloride, sodium, and potassium
- Urinalysis: dipstick for blood, protein, and glucose (microscopic examination may also be performed)

#### 4.5.3.1 Quantitative analyses

For quantitative analyses, analysis period is active treatment (placebo-controlled and DBE) period. For numeric laboratory parameters, actual values will be summarized by visit for all the common visits in both Cohort A and B in the active treatment (placebo-controlled and DBE) period. Number of evaluable subjects, mean, standard deviation, median, 25% and 75% quartiles, minimum and maximum values will be presented at each visit. Plots of mean actual values (with standard error) for key numeric laboratory parameters at each visit for all the visits in the active treatment (placebo-controlled and DBE) period will be provided.

Plots of mean actual values (with standard error) for numeric laboratory parameters at each visit for all the visits in the active treatment (placebo-controlled and DBE) period may be provided.

Change from baseline and percent change from baseline for numeric laboratory parameters will be summarized in the active treatment (placebo-controlled and DBE) period. Placebo-controlled baseline will be used for early start subjects and DBE baseline will be used for delayed start subjects. Change and percent change from baseline will be calculated based on the DBE baseline for delayed start subjects. Number of evaluable subjects, mean, standard deviation, median, 25% and 75% quartiles, minimum and maximum values will be presented at each visit.

Listings of individual laboratory measurements by patients for all the parameters will be provided for placebo-controlled and DBE period.



V2.0

Visit windows for by visit summaries

For laboratory by visit summaries, the analysis visit should be defined using visit windows (see Table 1 in the Appendix). Visit windows are generally from mid-points between the visit before to the current, and the midpoint from the current visit to the next visit. If there is more than 1 value in the same analysis visit window for a certain parameter for a subject, then the closest record to the target visit day will be used for the by visit analysis. If there are 2 values in the same analysis visit window with the same distance from the target visit day for a certain parameter for a subject, then the record with the later date will be used for the by visit analysis. If there are 2 values on the same day for a certain parameter for a subject, then the record with the later time will be used for the by visit analysis.

#### 4.5.3.2 Qualitative analyses

For qualitative analyses, all available values will be included (not just the "analyzed record" within each visit window in the quantitative analyses). Analysis period is active treatment (placebo-controlled and DBE) period.

#### Shift analyses

Laboratory data will be summarized using shift tables where appropriate for the active treatment (placebo-controlled and DBE) period. Each subject's hematology, blood chemistry and urinalysis numeric values will be flagged as "low", "normal", or "high" relative to the normal ranges of the central laboratory or as "unknown" if no result is available. Each subject's urinalysis categorical values will be flagged as "positive" or "negative", or "unknown" if no value is available.

Shifts from baseline to high/low status will be presented for hematology, blood chemistry and urinalysis numeric parameters, and shifts from baseline to abnormal (positive) will be presented for urinalysis categorical parameters. Shift to low includes normal to low, high to low, and unknown to low; Shift to high includes normal to high, low to high, and unknown to high. Subjects need to have at least one post-baseline evaluation and a baseline value not low or high or positive (including missing) in order to be included in the analysis.

For early start subjects, the placebo-controlled baseline will be used and shifts that occurred in either placebo-controlled or DBE period will be included. For delayed start subjects, the DBE baseline will be used and shifts that occurred in the DBE period based on DBE baseline will be included.

Potentially Clinically Significant (PCS) laboratory abnormalities analyses

Please refer to the placebo-controlled SAP for the parameters and criteria for potentially clinically significant laboratory abnormalities analyses.

The number of subjects with potentially clinically significant laboratory abnormalities post-baseline will be summarized for the active treatment (placebo-controlled and DBE) period.



V2.0

Subjects need to have at least one post-baseline evaluation in the active treatment period in order to be included in the analysis. For early start subjects, the placebo-controlled baseline will be used and abnormalities that occurred in either placebo-controlled or DBE period will be included. For delayed start subjects, the DBE baseline will be used and PCS abnormalities that occurred in the DBE period based on DBE baseline will be included.

A listing of subjects with PCS laboratory abnormalities in the active treatment (placebo-controlled and DBE) period will also be provided, with all the data in the placebo-controlled and DBE period will be listed.

#### Potential serious hepatotoxicity

Potential serious hepatotoxicity is defined as ALT or AST > 3x ULN and total bilirubin > 2x ULN at any time post-baseline, not necessarily concurrent, in the active treatment (placebo-controlled and DBE) period. A scatterplot of the maximum post-baseline ALT or AST value relative to ULN and maximum post-baseline total bilirubin value relative to ULN (not necessarily concurrent) will be provided. In addition, a line plot of ALT, AST, ALP and total bilirubin values over time for each subject with potential serious hepatotoxicity will be provided.

A listing of subjects with potential serious hepatotoxicity in the active treatment (placebo-controlled and DBE) period will be provided with the concurrent records labeled. All the data in the placebo-controlled and DBE period will be listed. Concurrent is defined as on the same day. Subjects with ALT > 1x ULN, > 3x ULN, > 5x ULN, > 10x ULN or > 20x ULN, subjects with AST > 1x ULN, > 3x ULN, > 5x ULN, > 10x ULN or > 20x ULN, subjects with total bilirubin > 1x ULN, > 1.5x ULN or > 2x ULN, subjects with ALP > 1x ULN or > 1.5x ULN and subjects with AST or ALT > 3x ULN post-baseline accompanied by concurrently elevated total bilirubin > 1.5x ULN or > 2x ULN will be labeled.

#### 4.5.4 Vital Sign Data

For vital sign data analyses, the analysis period is active treatment (placebo-controlled and DBE) period. Vital sign parameters include body temperature, systolic blood pressure, diastolic blood pressure, heart rate, respiration rate and weight. Vital signs will be measured with the subject supine and after the subject has been resting for at least 10 minutes. The descriptive statistics for actual values will be summarized at each visit in the active treatment (placebo-controlled and DBE) period. Plot of mean vital sign values in the active treatment (placebo-controlled and DBE period) may be provided.

Summary of change from baseline including number of evaluable subjects, mean, standard deviation, median, 25% and 75% quartiles, minimum, and maximum values will be summarized at each visit in the active treatment (placebo-controlled and DBE) period. Placebo-controlled baseline will be used for early start subjects and DBE baseline will be used for delayed start analysis.

The analysis of vital signs will also focus on the incidence of clinically relevant abnormalities at any post-baseline visit in the active treatment (placebo-controlled and DBE) period. Please refer to the placebo-controlled SAP for the criteria to assess potential clinically relevant abnormalities in vital sign. The incidence and percentage of clinically relevant abnormalities



V2.0

determined by each criterion will be summarized in the active treatment (placebo-controlled and DBE) period.

A listing of subjects with clinically relevant abnormalities at any post-baseline visit in the active treatment (placebo-controlled and DBE) period will also be provided. All the data in the placebo-controlled and DBE period will be listed.

Visit windows for by visit summaries

For vital sign by visit summaries, the analysis visit should be defined using windows (see Table 2 in the Appendix). For the same parameter for a subject, if there is more than 1 record in the same analysis visit window, then select the record closest to the target visit day. If there are 2 records in the same analysis visit window with the same distance from the target visit day, then select the record with the later date.

#### **4.5.5** ECG Data

For ECG data analyses, the analysis period is active treatment (placebo-controlled and DBE) period. The descriptive statistics for actual values will be summarized at each visit in the active treatment (placebo-controlled and DBE) period. Plot of mean ECG values in the active treatment (placebo-controlled and DBE) period may be provided.

Shift from normal or unknown ECG at baseline to abnormal post-baseline ECG, will be summarized in the active treatment (placebo-controlled and DBE) group. The number of subjects with potential QTcF interval outlier post-baseline will also be summarized in the active treatment (placebo-controlled and DBE) period. The criteria of defining QTcF interval outliers is specified in the placebo-controlled SAP. For early start subjects, the placebo-controlled baseline will be used. For delayed start subjects, the DBE baseline will be used.

A listing of subjects with abnormal ECG status post-baseline in the active treatment (placebo-controlled and DBE) period will be provided. All data in the placebo-controlled and DBE period will be listed.

#### 4.5.6 Physical and Neurological Examination

Abnormal findings during physical and neurological examinations are captured as adverse events and will be reflected in the summary of AEs.

#### 4.5.7 C-SSRS Data

The Columbia Suicide Severity Rating Scale (C-SSRS) is an assessment that evaluates suicidal ideation and behavior. There are 5 "Yes/No" questions on suicidal ideation following the increasing severity order: (1) Wish to be dead, (2) Non-specific active suicidal thoughts, (3) Active suicidal ideation with any methods (not plan) without intent to act, (4) Active suicidal ideation with some intent to act, without specific plan, (5) Active suicidal ideation with specific plan and intent, and 6 "Yes/No" questions on suicidal behavior



V2.0

following the increasing severity order: (6) Preparatory acts or behavior, (7) Aborted attempt, (8) Interrupted attempt, (9) Actual attempt, (10) Suicidal behavior, (11) Suicide (only at post-baseline visits). Another "Yes/No" question of whether the subject has engaged in non-suicidal self-injurious behavior is also collected.

The summary table for C-SSRS will be conducted for the active treatment (placebo-controlled and DBE) period. Number of subjects who answered "Yes" to each of the 11 questions post-baseline, subjects who answered "Yes" to at least one question for suicidal ideation, subjects who answered "Yes" to at least one question for suicidal behavior, and subjects who have engaged in non-suicidal self-injurious behavior will be presented.

A listing of subjects with any suicidal ideation or behavior at baseline or post-baseline will be provided for the placebo-controlled and DBE period.

#### 4.5.8 MRI Safety Data

Brain MRI safety finding are assessed at Screening visit, Week 24, 52, 96, 148 and 4 weeks after last dose/ET visits.

The MRI safety result is classified as normal or abnormal. Shift table from normal or unknown MRI at baseline to abnormal post-baseline MRI will be summarized in the active treatment (placebo-controlled and DBE) period. The worst post-baseline record of each subject is selected. A listing of details for abnormal brain MRI findings will be presented for placebo-controlled and DBE period.

#### 4.6 Pharmacodynamic - Imaging analysis

#### 4.6.1 General Consideration

There are three types of imaging outcomes in the study: DaT/SPECT imaging, Neuromelanin MRI imaging and Structural MRI imaging. Please refer to the placebo-controlled SAP for details.

The analysis population for pharmacodynamic analysis is defined in Section 3.1.1. The analysis period is placebo-controlled and DBE period. That is, data from both the placebo-controlled and DBE periods will be included in the analysis. All pharmacodynamic analyses will be presented by DBE treatment group.

The following three comparisons will be evaluated for the long-term pharmacodynamic analyses of BIIB054:

- The early start 250 mg compared with the delayed start 250 mg;
- The early start 1250 mg compared with the delayed start 1250 mg.
- The early start 3500 mg compared with the delayed start 3500 mg.

The following comparisons may also be evaluated:

• The early start 250 mg compared with the pooled delayed start group;



V2.0

- The early start 1250 mg compared with the pooled delayed start group;
- The early start 3500 mg compared with the pooled delayed start group

The pooled delayed start group contains all the subjects who were randomized to placebo treatment in the placebo-controlled period including those who did and who did not enter to the DBE period. There will be no multiple comparison adjustments. Data after subjects start PD symptomatic treatment will be included in the analyses.

#### Visit Windows for by visit analyses

For the by visit summaries and MMRM models, the analysis visit should be defined using visit windows (see Table 3 in the Appendix). If there is more than 1 value in the same analysis visit window (>1 value for the same analysis visit) for a certain parameter for a subject, then the closest record to the target visit day will be used for the by visit analysis. If they are with the same distance from the target visit day, then the record with the later time will be used for the by visit analysis.

#### 4.6.2 By Visit Summary and MMRM Model

A prespecified set of imaging measures as well as the change from baseline will be summarized by DBE treatment groups by visit for all the visits in the placebo-controlled and DBE period.

Change or percent change from baseline in the imaging measures will be analyzed using an MMRM model for all the visits in the placebo-controlled and DBE period. For details of the model to be used please see the 1 year SAP. Adjusted means for each treatment group, pairwise adjusted differences for the comparisons, 95% confidence intervals for the differences will be presented at each visit, and p-values will be presented for the key visits of week 24, 52, 96 and 148. If the distribution of the outcome is highly skewed, p-value will be generated from the MMRM model based on the rank data. Missing data are assumed to be missing at random behind the MMRM model.

Per design, a subset of subjects will enter year 3 and 4 for a limited time. There will be some visits with too few data in year 3 and 4. If this is the case, the visits with too few data will be excluded from the MMRM analyses, Otherwise, the MMRM model will not converge. In addition, since most patients will start PD medication by year 1, most data in year 2-4 will be after PD medication. Therefore, data after subject start PD medication will be included in the MMRM analyses. Otherwise, the MMRM model will not converge.

Data at the common visits of cohort A and cohort B will be included in the by visit summary and MMRM model. Data at all visits will be listed.

#### 4.6.3 Additional analyses of placebo-controlled period due to COVID-19

Due to COVID-19 public health emergency, considerations were made to allow week 52 assessments to be delayed up to 4 weeks. If this occurs, some of the data may not be included in the all patient week 52 analyses, as they may miss the timeline of the corresponding CONFIDENTIAL



V2.0

interim database lock. However, these data are still considered in the placebo-controlled period because they are before the first dose of DBE period. Depending how much data are missing in the all patient week 52 analyses database lock, the MMRM analyses in the placebo-controlled period may be repeated by including all the available data in the placebo-controlled period.



#### 4.8 Pharmacokinetics Analysis

Per protocol, sparse PK data are collected in the DBE period. Therefore, the PK analyses will be focused on summarizing the PK concentration over time. The PK analysis population as defined in Section 3.1.1 and data from both placebo-controlled and DBE periods will be included. All the PK analyses will be presented by DBE treatment group. In addition, an exposure-response (ER) analysis from both placebo-controlled and DBE periods will be conducted, to detect any ER relationship trend and potential covariate using any primary or secondary endpoint and BIIB054 exposure metrics as deemed appropriate. Other tables and figures based on the population PK and ER analyses will be generated by Clinical Pharmacology and Pharmacometrics (CPP) team and will be included in a separate report from CPP.

#### 4.9 Immunogenicity Analysis

#### 4.9.1 Analysis population

All immunogenicity data will be analyzed based on the immunogenicity population, which is same as the safety population as defined in Section 3.1.1.



V2.0

#### 4.9.2 Method of analysis

A summary table of subjects with treatment-emergent positive anti-BIB054 antibody responses in the placebo-controlled and DBE active treatment period will be displayed by DBE treatment group and by visit. Please refer to the placebo-controlled SAP for the definition of treatment-emergent positive anti-BIB054 antibody responses. In this summary, DBE baseline will be used for delayed start subjects who are assigned to receiving BIB054 in the DBE period. A listing of immunogenicity data in the placebo-controlled and DBE period for subjects with anti-BIB054 antibody positive responses will be provided.

#### Visit Windows for by visit analyses

For immunogenicity by visit summaries, the analysis visit should be defined using visit windows (see Table 12 in the Appendix). If there is more than 1 value in the same analysis visit window for a subject, then the closest record to the target visit day will be used for the by visit analysis. If there are 2 values in the same analysis visit window with the same distance from the target visit day for a certain parameter for a subject, then the record with the later date will be used for the by visit analysis. If there are 2 values on the same day for a certain parameter for a subject, then the record with the later time will be used for the by visit analysis.

#### 4.10 Interim Analyses

Safety and PK data only will be reviewed by the IDMC after subjects in Cohort A have completed Week 12 Visit assessments, and before dosing any subjects in Cohort B.

After subjects in Cohort A complete the Week 24 Visit, all available serum PK, and biomarker data (specifically the α-syn levels and complex formation data, if available) from Cohort A will be analyzed by a statistical/PK team independent of the study. The grouped level summary statistics will be reviewed only by a limited number of individuals at Biogen who are not involved in the management of the subjects or subject-level data for the study. No changes to the study design are expected based on this review.

For the purpose of planning for future studies, an administrative interim analysis may be

For the purpose of planning for future studies, an administrative interim analysis may be performed when approximately 60% of the subjects have completed the Week 52 Visit. A small unblinded team from Biogen, separate from the study management team, will have access to the unblinded interim analysis results. As of the finalization of protocol Version 8 and all subjects have completed Week 52 visits, this analyses was not conducted.

A full analysis of the 1-year data will be performed after all subjects have completed the Week 52 Visit. A small unblinded team from Biogen, separate from the study management team, will have access to the unblinded 1-year analysis results.

An interim analysis when all subjects have completed the Week 72 Visit is planned to be conducted. A small unblinded team from Biogen, separate from the study management team, will have access to the unblinded interim analysis results. All efficacy endpoints will be analyzed at the Week 72 analyses. Selected key safety data (e.g. summary of AE and SAE, summary of MRI safety findings and incidence of anti-drug antibodies) will be summarized, as this is only a snapshort of the safety profile at the time of CONFIDENTIAL



V2.0

the Week 72 interim analysis, and the comprehensive safety profile will be presented at the End of Study

A multiple comparison adjustment method will be applied to control the overall type I error at 0.05 in the study, due to the primary endpoint of change from baseline in MDS-UPDRS total score being analyzed at Week 52 and Week 72, and superiority against placebo is considered reached in the study if statistically significant result is achieved at either timepoint at the respective adjusted alpha-level.

A graphical procedure will be used to control the overall type I error at 0.05 level due to multiple-testing. An alpha of 0.04 will be allocated to the Week 52 primary endpoint analyses and an alpha of 0.01 will be allocated to the Week 72 primary endpoint analysis.

- If the Week 52 analysis is statistically significant at the 0.04 level (i.e. p-value ≤ 0.04), the alpha of 0.04 will be transferred (recycled) to the Week 72 analysis, and Week 72 will have alpha=0.05.
- If the Week 52 analysis is not statistically significant at the 0.04 level, alpha of 0.01 will be used for the Week 72 analysis. Statistically significance is considered achieved if the p-value is ≤0.01 at Week 72.
- If statistical significance is achieved at the Week 72, in either scenarios above, then the alpha of 0.01 will be transferred (recycled) back to Week 52, and the Week 52 primary analysis will be re-evaluated for statistically signifiance at the 0.05 level. This will only change the conclusion of the Week 52 results if the initial p-value is greater than 0.04 and ≤0.05.

No additional multiplicity adjustments will be made for secondary or exploratory endpoint analyses.

A blinded sample size re-estimation may be conducted when approximately 10% of subjects have completed the Week 52 Visit or approximately 1 month before enrollment is projected to be completed, whichever is earlier. The study sample size may be increased based on this blinded data review. There may be small adjustments to the percentage depending on actual enrollment rate. As of the finalization of protocol Version 8 and all subjects have completed Week 52 visits, this analyses was not conducted.

#### 5 Assessment of the impact of Covid-19 on statistical analyses

As this study is on-going when the Covid-19 public health emergency (PHE) occurred, subject visits and data collection were impacted, including missing visits, delayed visits, missed assessments and/or some visits were performed via remote assessments, e.g. telephone/video visits. Every effort was made to document these impacted study activities systematically on the eCRF and other electronic source data.



V2.0

A complete listing of all visits impacted (e.g. missed visits, delayed or assessment done via remote visits) will be listed in the clinical study report. Missing data due to Covid-19 is considered as missing at random.

#### Impact of COVID-19 on the clinical outcome analyses

In addition, subgroup analyses of the selected key clinical outcome MDS-UPDRS will be performed on a subset of subjects who did not have >=3 consecutive missing doses throughout the study to further evaluate the impact of Covid-19 on the study. The same MMRM model for the primary analyses will be used for the subgroup analyses.

In addition, due to Covid-19, some visits were delayed. A few subjects will have their Week 52 imaging done at later visits up to Week 72 and these will still be considered as Week 52 visit data in the analyses for Week 52. These data were not included in the Week 52 database lock in time, but will be included in the Week 72 database, and the related Week 52 imaging analyses will be updated at the time of the Week 72 interim analyses.

#### Impact of COVID-19 on the safety analyses

During the COVID-19 pandemic period, subjects may be prone to a high risk of getting depressed or anxiety. As a result, the analyses below will be performed to evaluate the impact of the COVID-19 pandemic on the safety analyses.

- 1. An overall summary of AE in DBE period based on data after March 7<sup>th</sup>, 2020, the start date when subjects in SPARK get impacted by COVID-19
- 2. An overall summary of AE in the active treatment (placebo-controlled and DBE) period based on data after March 7<sup>th</sup>, 2020, the start date when subjects in SPARK get impacted by COVID-19
- 3. AEs by system organ class and preferred term sorted by decreasing frequency in DBE period based on data after March 7<sup>th</sup>, 2020, the start date when subjects in SPARK get impacted by COVID-19
- 4. AEs by system organ class and preferred term sorted by decreasing frequency in active treatment (placebo-controlled and DBE) period based on data after March 7<sup>th</sup>, 2020, the start date when subjects in SPARK get impacted by COVID-19
- 5. C-SSRS data summary based on data after March 7<sup>th</sup>, 2020, the start date when subjects in SPARK get impacted by COVID-19

#### **Certificate Of Completion**

Envelope Id: ECF3A588273348DCBA7D0E61E7899330

Subject: Please DocuSign: 228PD201\_SAP\_DBE\_final\_v2.0\_clean\_23June2021.docx

Vendor Name: Source Envelope:

Document Pages: 41 Certificate Pages: 5

AutoNav: Enabled

**Envelopeld Stamping: Enabled** 

Time Zone: (UTC-05:00) Eastern Time (US & Canada)

Status: Completed

**Envelope Originator:** 



#### Record Tracking

Status: Original

6/23/2021 1:48:56 PM

Location: DocuSign

#### Signer Events

Biogen

Security Level: Email, Account Authentication

(None)

#### Signature

Signatures: 5

Initials: 0



Signature Adoption: Pre-selected Style Using IP Address:

#### **Timestamp**

Sent: 6/23/2021 1:51:14 PM Viewed: 6/23/2021 2:42:37 PM Signed: 6/23/2021 2:42:55 PM

#### **Electronic Record and Signature Disclosure:**

Not Offered via DocuSign



Biogen

Security Level: Email, Account Authentication (None)

Signature Adoption: Pre-selected Style Using IP Address:

Sent: 6/23/2021 1:51:14 PM Viewed: 6/23/2021 2:05:35 PM Signed: 6/23/2021 2:05:49 PM

#### **Electronic Record and Signature Disclosure:**

Not Offered via DocuSign



Security Level: Email, Account Authentication (None)



Signature Adoption: Pre-selected Style Using IP Address:

Sent: 6/23/2021 1:51:15 PM Viewed: 6/23/2021 2:08:11 PM Signed: 6/23/2021 2:08:17 PM

#### **Electronic Record and Signature Disclosure:**

Accepted: 6/23/2021 2:08:11 PM

ID: 520189fa-b9b6-4e49-9c27-538c44833496



Biogen

Security Level: Email, Account Authentication (None)

**Electronic Record and Signature Disclosure:** 

Not Offered via DocuSign



Signature Adoption: Pre-selected Style Using IP Address:

Sent: 6/23/2021 1:51:14 PM Viewed: 6/23/2021 2:54:33 PM Signed: 6/23/2021 2:54:52 PM

## Signer Events

Biogen

Security Level: Email, Account Authentication

#### Signature



Signature Adoption: Pre-selected Style Using IP Address:

#### **Timestamp**

Sent: 6/23/2021 1:51:14 PM Viewed: 6/23/2021 1:51:32 PM Signed: 6/23/2021 1:51:42 PM

## Electronic Record and Signature Disclosure: Not Offered via DocuSign

| In Person Signer Events | Signature | Timestamp |
|---|---|---|
| Editor Delivery Events | Status | Timestamp |
| Agent Delivery Events | Status | Timestamp |
| Intermediary Delivery Events | Status | Timestamp |
| Certified Delivery Events | Status | Timestamp |
| Carbon Copy Events | Status | Timestamp |
| Witness Events | Signature | Timestamp |
| Notary Events | Signature | Timestamp |
| Envelope Summary Events | Status | Timestamps |
| Envelope Sent Certified Delivered Signing Complete Completed | Hashed/Encrypted Security Checked Security Checked Security Checked | 6/23/2021 1:51:15 PM<br>6/23/2021 1:51:32 PM<br>6/23/2021 1:51:42 PM<br>6/23/2021 2:54:52 PM |
| Payment Events | Status | Timestamps |
| Electronic Record and Signature Disclosure | | |

#### ELECTRONIC RECORD AND SIGNATURE DISCLOSURE

From time to time, Biogen (we, us or Company) may be required by law to provide to you certain written notices or disclosures. Described below are the terms and conditions for providing to you such notices and disclosures electronically through your DocuSign, Inc. (DocuSign) Express user account. Please read the information below carefully and thoroughly, and if you can access this information electronically to your satisfaction and agree to these terms and conditions, please confirm your agreement by clicking the 'I agree' button at the bottom of this document.

#### Getting paper copies

At any time, you may request from us a paper copy of any record provided or made available electronically to you by us. For such copies, as long as you are an authorized user of the DocuSign system you will have the ability to download and print any documents we send to you through your DocuSign user account for a limited period of time (usually 30 days) after such documents are first sent to you. After such time, if you wish for us to send you paper copies of any such documents from our office to you, you will be charged a \$0.00 per-page fee. You may request delivery of such paper copies from us by following the procedure described below.

#### Withdrawing your consent

If you decide to receive notices and disclosures from us electronically, you may at any time change your mind and tell us that thereafter you want to receive required notices and disclosures only in paper format. How you must inform us of your decision to receive future notices and disclosure in paper format and withdraw your consent to receive notices and disclosures electronically is described below.

### Consequences of changing your mind

If you elect to receive required notices and disclosures only in paper format, it will slow the speed at which we can complete certain steps in transactions with you and delivering services to you because we will need first to send the required notices or disclosures to you in paper format, and then wait until we receive back from you your acknowledgment of your receipt of such paper notices or disclosures. To indicate to us that you are changing your mind, you must withdraw your consent using the DocuSign 'Withdraw Consent' form on the signing page of your DocuSign account. This will indicate to us that you have withdrawn your consent to receive required notices and disclosures electronically from us and you will no longer be able to use your DocuSign Express user account to receive required notices and consents electronically from us or to sign electronically documents from us.

#### All notices and disclosures will be sent to you electronically

Unless you tell us otherwise in accordance with the procedures described herein, we will provide electronically to you through your DocuSign user account all required notices, disclosures, authorizations, acknowledgements, and other documents that are required to be provided or made available to you during the course of our relationship with you. To reduce the chance of you inadvertently not receiving any notice or disclosure, we prefer to provide all of the required notices and disclosures to you by the same method and to the same address that you have given us. Thus, you can receive all the disclosures and notices electronically or in paper format through the paper mail delivery system. If you do not agree with this process, please let us know as described below. Please also see the paragraph immediately above that describes the consequences of your electing not to receive delivery of the notices and disclosures electronically from us.

#### How to contact Biogen:

You may contact us to let us know of your changes as to how we may contact you electronically, to request paper copies of certain information from us, and to withdraw your prior consent to receive notices and disclosures electronically as follows:

To contact us by email send messages to: DL-eSignature@biogen.com

#### To advise Biogen of your new e-mail address

To let us know of a change in your e-mail address where we should send notices and disclosures electronically to you, you must send an email message to us at DL-eSignature@biogen.com and in the body of such request you must state: your previous e-mail address, your new e-mail address. We do not require any other information from you to change your email address.. In addition, you must notify DocuSign, Inc to arrange for your new email address to be reflected in your DocuSign account by following the process for changing e-mail in DocuSign.

#### To request paper copies from Biogen

To request delivery from us of paper copies of the notices and disclosures previously provided by us to you electronically, you must send us an e-mail to DL-eSignature@biogen.com and in the body of such request you must state your e-mail address, full name, Postal address, and telephone number. We will bill you for any fees at that time, if any.

#### To withdraw your consent with Biogen

To inform us that you no longer want to receive future notices and disclosures in electronic format you may:

i. decline to sign a document from within your DocuSign account, and on the subsequent page, select the check-box indicating you wish to withdraw your consent, or you may; ii. send us an e-mail to DL-eSignature@biogen.com and in the body of such request you must state your e-mail, full name, IS Postal Address, telephone number, and account number. We do not need any other information from you to withdraw consent.. The consequences of your withdrawing consent for online documents will be that transactions may take a longer time to process..

#### Required hardware and software

| Operating Systems: | Windows2000? or WindowsXP? |
|---|---|
| Browsers (for SENDERS): | Internet Explorer 6.0? or above |
| Browsers (for SIGNERS): | Internet Explorer 6.0?, Mozilla FireFox 1.0, |
| | NetScape 7.2 (or above) |
| Email: | Access to a valid email account |
| Screen Resolution: | 800 x 600 minimum |
| Enabled Security Settings: | •Allow per session cookies |
| | •Users accessing the internet behind a Proxy<br>Server must enable HTTP 1.1 settings via<br>proxy connection |

<sup>\*\*</sup> These minimum requirements are subject to change. If these requirements change, we will provide you with an email message at the email address we have on file for you at that time providing you with the revised hardware and software requirements, at which time you will have the right to withdraw your consent.

#### Acknowledging your access and consent to receive materials electronically

To confirm to us that you can access this information electronically, which will be similar to other electronic notices and disclosures that we will provide to you, please verify that you were able to read this electronic disclosure and that you also were able to print on paper or electronically save this page for your future reference and access or that you were able to e-mail this disclosure and consent to an address where you will be able to print on paper or save it for your future reference and access. Further, if you consent to receiving notices and disclosures exclusively in electronic format on the terms and conditions described above, please let us know by clicking the 'I agree' button below.

By checking the 'I Agree' box, I confirm that:

- I can access and read this Electronic CONSENT TO ELECTRONIC RECEIPT OF ELECTRONIC RECORD AND SIGNATURE DISCLOSURES document; and
- I can print on paper the disclosure or save or send the disclosure to a place where I can print it, for future reference and access; and
- Until or unless I notify Biogen as described above, I consent to receive from exclusively through electronic means all notices, disclosures, authorizations, acknowledgements, and other documents that are required to be provided or made available to me by Biogen during the course of my relationship with you.



V2.0

# **SPARK**228PD201

# Statistical Analysis Plan

**Dose Blinded Extension Period** 



## Statistical Analysis Plan

**Dose Blinded Extension Period** 

V2.0

#### STATISTICAL ANALYSIS PLAN **Dose Blinded Extension Period**

**Product Studied: BIIB054** Protocol Number: 228PD201

A Multicenter, Randomized, Double-Blind, Placebo-Controlled Study, with an Active-Treatment Dose-Blinded Period, to Evaluate the Safety, Pharmacokinetics, and Pharmacodynamics of BIIB054 in Subjects with Parkinson's Disease

> **Protocol Version: Version 8.0** Date of Protocol: 11 Aug 2020

Date of Statistical Analysis Plan: 23 June 2021, Final V2.0





**V2.0** 

## **VERSION HISTORY**

| SAP Version | Date | Primary Reasons for<br>Amendment |
|-------------|--------------|-----------------------------------------|
| 1.0 | 25-SEP-2020 | First version of the SAP |
| 2.0 | 23-JUNE-2021 | Update links within sample size section |
| | | Update SMT job titles |


**Dose Blinded Extension Period** 

**V2.0** 

#### **Table of Contents**

| 1 | DESCRIPTION OF OVERALL STUDY (INCLUDING DOSE-BLINDED EXTENS) DBJECTIVES AND ENDPOINTS | |
|---|---|---|
| 2 | STUDY DESIGN | 12 |
| | 2.1 Study Overview | |
| | 2.1.1 Year 1 (Placebo-Controlled Portion of the Study) | |
| | 2.1.2 Years 2-4 (Active-Treatment Dose-Blinded Portion of the Study) | |
| | 2.2 STUDY SCHEMATIC | |
| | 2.3 SCHEDULE OF EVENTS | |
| 3 | SAMPLE SIZE JUSTIFICATION | 15 |
| 4 | STATISTICAL ANALYSIS METHODS | 18 |
| | 4.1 GENERAL CONSIDERATIONS | 18 |
| | 4.1.1 Analysis Population | 20 |
| | 4.1.2 Analyses period | |
| | 4.2 BACKGROUND CHARACTERISTICS | 21 |
| | 4.2.1 Accounting of Subject | 21 |
| | 4.2.2 Demographics and Baseline Characteristics | |
| | 4.2.3 Concomitant Medications and Non-Drug Therapies | |
| | 4.2.4 Protocol Deviations | |
| | 4.2.5 Study Drug Exposure and Study Drug Compliance | |
| | 4.3 EFFICACY ANALYSES | |
| | 4.3.1 General Consideration | |
| | 4.3.2 Primary efficacy endpoint analysis | |
| | 4.3.3 Secondary efficacy endpoints and additional endpoints analysis | 26 |
| | 4.3.3.1 MDS-UPDRS based endpoints | |
| | 4.3.3.2 Other clinical efficacy measures | |
| | 4.5 SAFETY ANALYSES | |
| | 4.5.1 General Considerations. | |
| | 4.5.2 Clinical Adverse Events | |
| | 4,5,2,1 Summary and incidence analysis | |
| | 4.5.2.2 Incidence and incidence rate analysis for active treatment (placebo-controlled and DBE | |
| | 4.5.3 Clinical Laboratory Data | |
| | 4.5.3.1 Quantitative analyses | 32 |
| | 4.5.3.2 Qualitative analyses | |
| | 4.5.4 Vital Sign Data | |
| | 4.5.5 ECG Data | |
| | 4.5.6 Physical and Neurological Examination | |
| | 4.5.7 C-SSRS Data | |
| | 4.5.8 MRI Safety Data | |
| | 4.6 PHARMACODYNAMIC -IMAGING ANALYSIS | |
| | 4.6.1 General Consideration | |
| | 4.6.2 By Visit Summary and MMRM Model | / 3<br>وو |
| | 4.0.3 Additional analyses of placeoo-controlled period due to COVID-19 | 38 |
| | | 38 |
| | 4.8 PHARMACOKINETICS ANALYSIS | |
| | 4.9 IMMUNOGENICITY ANALYSIS | |
| | 4.9.1 Analysis population. | |
| | 4.9.2 Method of analysis | |
| | 4.10 Interim Analyses | |
| _ | ACCECOMENT OF THE IMPACT OF COVID-10 ON STATISTICAL ANALYSES | 40 |



Dose Blinded Extension Period

V2.0

#### LIST OF ABBREVIATIONS

| SI OF ABBREVIAL | |
|---|---|
| 470.4 | |
| ADA | anti-drug antibodies |
| AE | adverse event |
| ALP | alkaline phosphatase |
| ALT | alanine aminotransferase |
| ANCOVA | analysis of covariance |
| APTT | activated partial thromboplastin time |
| AST | aspartate aminotransferase |
| AUC | area under the curve |
| BL | baseline |
| BLQ | below the limit of quantification |
| BMI | body mass index |
| BPM | beats per minute |
| BRP-AUC | body region progression AUC |
| C <sub>max</sub> | observed maximum serum BIIB054 concentration |
| C <sub>min</sub> | observed minimum serum BIIB054 concentration |
| CI | confidence interval |
| CPP | Clinical Pharmacology and Pharmacometrics |
| C-SSRS | Columbia Suicide Severity Rating Scale |
| CTCAT | Common Toxicity Criteria for Adverse Events |
| CV | coefficient of variation |
| DaT | dopamine transporter |
| DaTscan <sup>TM</sup> | Ioflupane I123 radioligand for imaging of dopamine transporter |
| DBE | dose blinded extension |
| DBP | diastolic blood pressure |
| EC <sub>50</sub> | Concentration at 50% of maximum observed biologic effect |
| ECG | electrocardiogram |
| eCRF | electronic case report form |
| EOS | end of study |
| EOT | end of treatment |
| EP-RPS | Early Parkinson's Region Progression Score |
| ER | exposure-response |
| ICF | informed consent form |
| ICH | International Conference on Harmonisation |
| IDMC | independent data monitoring committee |
| INR | International normalized ratio |
| ITT | intent-to-treat |
| IXRS | Interactive Voice/Web Response System |
| LOCF | last observation carried forward |
| Loci | I hast coset varion carried for walla |



Dose Blinded Extension Period

| T. C | |
|-----------|-------------------------------------------------------------|
| LSmeans | least-square means |
| DBE | Dose-blinded extension |
| IV | intravenous |
| mAb | monoclonal antibody |
| MAO-B | monoamine oxidase type B |
| MCP-MOD | multiple comparison procedure – modeling |
| MDS-UPDRS | Movement Disorder Society Sponsored Revision of the Unified |
| | Parkinson's Disease Rating Scale |
| MedDRA | Medical Dictionary for Regulatory Activities |
| MMRM | mixed-model repeated measures |
| MRI | magnetic resonance imaging |
| PCS | potentially clinically significant |
| PD | Parkinson's disease |
| PK | pharmacokinetic(s) |
| PT | preferred term |
| PP | per-protocol |
| RBC | red blood cell |
| RNA | ribonucleic acid |
| SAE | serious adverse event |
| SAP | statistical analysis plan |
| SBP | systolic blood pressure |
| SBR | striatal binding ratio |
| SD | standard deviation |
| SE | standard error |
| SOC | system organ class |
| SPECT | single-photon emission computed tomography |
| TEAE | treatment-emergent adverse event |
| ULN | upper limit of normal |
| US | United States |
| WBC | white blood cell |
| WHO | World Health Organization |



V2.0

Note: This statistical analysis plan (SAP) covers the analyses of the dose-blinded extension (i.e., long terms extension) period (Years 2-4) and the analyses across both the placebo-controlled period and the DBE period (analyses integrating the data for Years 1-4) for study 228PD201. Please refer to the separate SAP for the analyses methods and approaches for placebo-controlled Year 1 period.

### 1 DESCRIPTION OF OVERALL STUDY (INCLUDING DOSE-BLINDED EXTENSION (DBE)) OBJECTIVES AND ENDPOINTS

The objectives and endpoints of the study are listed below.

The secondary efficacy endpoints have been ranked based on the order of clinical importance.

| Primary Objective | Primary Endpoints |
|---|---|
| To evaluate the clinical efficacy of BIIB054 via dose response using the change from baseline in Movement Disorder Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Total Score | Change from baseline in MDS-UPDRS Total Score (Sum of Parts I, II, and III) at the primary timepoints of Week 52 and Week 72 |
| Secondary Objectives | Secondary Endpoints |
| To evaluate the clinical efficacy of BIIB054 based on MDS-UPDRS subparts | Change from baseline to Week 52 in MDS-UPDRS the subparts III, II and I (each part separately) |
| | Change from baseline to Week 72 and end of study in MDS-UPDRS the subparts III, II and I (each part separately) |
| To assess the PK profile of BIIB054 | Concentration of BIIB054 in the serum |
| To evaluate the dose-related safety of BIIB054 | Incidence of adverse events (AEs) and serious adverse events (SAEs) |
| To evaluate the pharmacodynamic effects of BIIB054 on the integrity of nigrostriatal dopaminergic nerve terminals | Change from baseline to Week 52 in striatal binding ratio (SBR) in the putamen, striatum, and caudate as measured by single-photon emission computed tomography (SPECT) imaging of the dopamine transporter (DaT) with ioflupane I123 (DaTscan <sup>TM</sup> ) |
| To evaluate the immunogenicity of BIIB054 | Incidence and titer of anti-BIIB054 antibodies in the serum |



Dose Blinded Extension Period

| <b>Exploratory Objectives</b> | Exploratory Endpoints |
|-------------------------------|-----------------------|
| Exploratory Objectives | Exploratory Endpoints |
| | • |
| | • |
| | • |
| | ≥ |
| | - |
| | _ |
| | - |
| | • |



Dose Blinded Extension Period





Dose Blinded Extension Period





Dose Blinded Extension Period





V2.0

#### 2 STUDY DESIGN

#### 2.1 Study Overview

This Phase 2a, randomized, double-blind, parallel-group, placebo-controlled study (Year 1) with an active-treatment dose-blinded period (Year 2 through 4) will examine the efficacy, safety, PK, and pharmacodynamics of BIIB054, administered every 4 weeks via IV infusion to adult subjects with PD. Approximately 311 subjects will be enrolled at about 85 sites globally.

#### 2.1.1 Year 1 (Placebo-Controlled Portion of the Study)

Prior to the first dose in Year 1, all subjects in the study will be randomized into 4 arms, to receive 13 doses of BIIB054 (250, 1250, or 3500 mg) or placebo.

Subjects will be enrolled into 2 cohorts. Cohort A will be randomized first, in a 1:1:1:1 ratio into each of the 4 treatment arm and will include approximately 24 subjects. Randomization and dosing for Cohort B (approximately 287 planned subjects) will start after all subjects in Cohort A complete Week 12 assessments, and all available safety and PK data are reviewed by the IDMC. Randomization of subjects in Cohort B will be stratified by baseline (Day 1) MDS-UPDRS Part I + II + III total scores (≤35 and >35) and striatum SBR (≤1.2 and >1.2), and subjects will be randomized at Day 1 into 1 of 4 parallel dosing arms in each stratum. After all subjects in Cohort A complete Week 12 assessments (28 days after their third infusion), and before dosing any subjects in Cohort B, all available safety and PK data will be reviewed by the IDMC. No subjects in Cohort B may be dosed until the IDMC review is complete. The study schematic is presented in Figure 1. After IDMC review is complete, subjects in Cohort B will be randomized, and dosing may begin. During the review period, subjects in Cohort A will continue to be dosed on a schedule of once every 4 weeks.

The first IDMC meeting will occur after the last subject in Cohort A completes Week 12 assessments, or approximately 6 months after the first subject has been enrolled in Cohort A, whichever comes first. Regular IDMC meetings will occur approximately every 3 months after the first meeting.



Any changes will be documented in a protocol amendment.

#### 2.1.2 Years 2-4 (Active-Treatment Dose-Blinded Portion of the Study)

Prior to Infusion 14 (the first dose of Year 2) at Week 52, subjects who received placebo in Year 1 will be randomized into 1 of the active-dosing arms for Year 2; these subjects will receive BIIB054 in Year 2. Subjects who received BIIB054 (250mg, 1250 mg or 3500 mg) in Year 1 of the study will continue with the same dose regimen in Year 2. Subjects receiving the 250-mg dose in Year 1 continued on their original dose assignment.



V2.0

Subjects will receive 12 additional doses of BIIB054 (250, 1250, or 3500 mg) in Year 2 and up to 16 additional doses in Years 3 and 4. Up until the last subject in the study has had his or her last dose in Year 2 of the study (Week 96 Visit), eligible subjects will be able to continue treatment once every 4 weeks.

Subjects who complete dosing through Week 96 and the Final Visit 12 weeks after the last visit will be considered Year 2 completers in the eCRF.

See Figure 2 for a depiction of the duration of dosing in Years 3 and 4 for subjects continuing dosing past Week 96.

Figure 4 in the protocol presents a flowchart for dosing and procedures from Week 96 through end of study, including how to determine which subjects are eligible to continue dosing past Week 96.

#### 2.2 Study Schematic

Figure 1: Study Design



DaT = dopamine transporter; IDMC = independent data monitoring committee; PK = pharmacokinetic(s); SPECT = single-photon emission computed tomography

<sup>&</sup>lt;sup>a</sup> Prior to Infusion 14 (first dose of Year 2), subjects who received placebo in Year 1 will be randomized to 1 of the active-treatment groups; these subjects will receive BIIB054 in Year 2. Subjects who received BIIB054 in Year 1 will continue with the same dose regimen in Years 2 through 4. Dosing will continue until the last subject in the study has had his or her Week 96 Visit. Not all subjects will have the opportunity for dosing past Year 2/Week 96.



Figure 2: Overview of Study Dosing:



Q4W = every 4 weeks.

Year 1 = Placebo-controlled period. Years 2 through 4 = Active-treatment dose-blinded period. Not all subjects will have the opportunity for dosing past Year 2/Week 96.



V2.0

#### 2.3 Schedule of Events

See Protocol Section 4.2.

#### 3 SAMPLE SIZE JUSTIFICATION

The sample size calculation is based on changes in MDS-UPDRS Part I + II + III total score at Week 52 and at Week 72 of treatment. Based on data from the Parkinson's Progression Markers Initiative study, the placebo subject's mean and standard deviation (SD) at Week 52 and Week 72 are assumed to be 8.0 (10.64) and 9.6 (13.7) respectively. Assuming a maximum of 55% reduction in the change from baseline in the active group with maximum response relative to placebo group, the mean (SD) for this active group will be 3.2 (10.64) and 3.84 (13.7) respectively at Week 52 and Week 72, and the responses for other active groups are assumed to be somewhere between 0 and the maximum response. The primary analysis will be based on the MCP-MOD method to detect a dose-response trend while controlling for multiplicity. Optimal contrasts will be constructed to detect potential doseresponse trend under common dose-response curves (e.g., E<sub>max</sub>, exponential, logistic, linear in log dose, and quadratic model, which are illustrated with parameters shown in Figure 3.1 which will be used for both Week 52 and Week 72). The planned enrollment is 311 subjects total (24 subjects in Cohort A and 287 subjects in Cohort B, 3.1). Actual enrollment is 357 subjects. In Cohort A, 29 subjects were randomized in a 1:1:1:1 ratio to each of the treatment groups, while in Cohort B 328 subjects were randomized in 2:1:2:2 ratio to the placebo, 250 mg, 1250 mg, and 3500 mg groups. Based on the actual enrollment, the estimated number of subjects by cohort and treatment groups are given in Table 3.2 below. After accounting for dropout rate of 10% and 15% at Week 52 and Week 72, respectively, the estimated sample sizes are given in Table 3.3 and Table 3.4. With the updated sample size, the study will provide an average power of approximately 80% to detect the dose-response trend over 1 year of treatment, based on a 2-sided type I error of 0.05 and approximately 73% of power at the Week 72 analyses, based on a 2-sided type I error of 0.05. Overall, the sample size in the study will provide approximately 89% power, taking into consideration success at either Week 52 or Week 72.

With an estimated sample size of 100 subjects dosed per arm in the 1250 mg and 3500 mg arms, the study has 80% probability of detecting AEs with a rate of 1.6% or greater in these 2 arms, and a 90% probability of detecting AEs occurring with a rate of 2.3% or greater.



Figure 3.1: Candidate Models for Dose-Response





**Dose Blinded Extension Period** 

V2.0

**Table 3.1: Estimated Sample Size Per Group (Planned)** 

| | | Treatment Group | | | |
|----------|---------|-----------------|---------|---------|-----|
| | Placebo | | | | |
| Cohort | | 250 mg | 1250 mg | 3500 mg | |
| Cohort A | 6 | 6 | 6 | 6 | 24 |
| Cohort B | 82 | 41 | 82 | 82 | 287 |
| Total | 88 | 47 | 88 | 88 | 311 |

**Table 3.2: Estimated Sample Size Per Group Based on Actual Enrollment** (Before Drop-Outs)

| | Treatment Group | | | | |
|----------|-----------------|--------|---------|---------|-----|
| | Placebo | | | | |
| Cohort | | 250 mg | 1250 mg | 3500 mg | |
| Cohort A | 8 | 7 | 7 | 7 | 29 |
| Cohort B | 93 | 47 | 94 | 94 | 328 |
| Total | 101 | 54 | 101 | 101 | 357 |

**Table 3.3:** Estimated Sample Size Per Group Based on Actual Enrollment (After Adjusting for 10% Drop-Out At Week 52

| | Treatment Group | | | | |
|----------|-----------------|--------|---------|---------|-----|
| | Placebo | | | | |
| Cohort | | 250 mg | 1250 mg | 3500 mg | |
| Cohort A | 7 | 6 | 6 | 6 | 25 |
| Cohort B | 84 | 42 | 84 | 84 | 294 |
| Total | 91 | 48 | 90 | 90 | 319 |

**Table 3.4:** Estimated Sample Size Per Group Based on Actual Enrollment (After Adjusting for 15% Drop-Out At Week 72

| | Treatment Group | | | | |
|----------|-----------------|--------|---------|---------|-----|
| | Placebo | | | | |
| Cohort | | 250 mg | 1250 mg | 3500 mg | |
| Cohort A | 7 | 6 | 6 | 6 | 25 |
| Cohort B | 79 | 40 | 80 | 80 | 279 |
| Total | 86 | 46 | 86 | 86 | 304 |




V2.0

#### 4 STATISTICAL ANALYSIS METHODS

#### 4.1 General Considerations

This statistical analysis plan (SAP) covers the analyses of the dose-blinded extension (i.e., long term extension) period (Years 2-4) and the analyses across both the placebo-controlled period and the DBE period (analyses integrating the data for Years 1-4).

Summary tables will be presented using descriptive summary statistics. For continuous variables, summary statistics will generally include number of subjects with data, mean, standard deviation, median, 25% percentile, 75% percentile, minimum and maximum. For categorical variables, this will generally include number of subjects randomized or dosed, number with data, and the percent of those with data in each category. Pharmacokinetics (PK) summaries will also include Geometric mean and geometric CV.

Statistical testing will be performed to assess efficacy endpoints by conducting pairwise comparison between each BIIB054 group and the delayed-start group (i.e. subjects who were randomized to placebo in Year-1),. Dose-response relationship may also be tested. Unless stated otherwise, all the statistical tests will be 2-sided with a statistical significance level of 0.05.

The statistical software, SAS® will be used for all summaries and analyses.

#### Analysis displays

Unless otherwise specified, the analysis of the DBE period and the analyses across both the placebo-controlled period and the DBE period will be displayed by DBE treatment groups as shown below, separate for early and delayed start treatment group) including tables, listings and figures, unless otherwise specified.

Unless otherwise specified, analyses for efficacy data (e.g., pharmacodynamics of imaging, clinical efficacy, displayed by the following treatment groups according to randomization assignment at the start of the placebo-controlled period:

- BIIB054 early start: subjects who are assigned to (1) receive BIIB054 in the placebo-controlled period and (2) continue receiving BIIB054 in the DBE period
- BIIB054 late start: subjects who are assigned to (1) receive placebo in the placebo-controlled period and (2) switch to BIIB054 in the DBE period

Unless otherwise specified, analyses for safety, PK, and ADA data will be displayed by the following treatment groups according to dose received:

• BIIB054 early start: subjects who receive BIIB054 in the placebo-controlled period (regardless of randomization assignment)



V2.0

- BIIB054 late start: subjects who receive only placebo in the placebo-controlled period (regardless of randomization assignment) and switch to receive BIIB054 in the DBE period
- BIIB054 total: subjects in either BIIB054 early or late start treatment groups

.

If all subjects received study treatment according to their randomization assignments during the placebo-controlled period (i.e. no subject assigned to placebo received BIIB054, and no subject assigned to BIIB054 received only placebo), then the assignment of subjects to treatment groups in efficacy related tables will be the same as those in safety related tables.

For efficacy, pharmacodynamic of imaging, and PK and ADA outcomes. Each BIIB054 early start dose group may be compared with the corresponding delay-start dose group, as well as the pooled delay-start group. Outputs will be presented in the following two ways:

| BIIB054 delayed start | | | I | BIIB054 early start | |
|---|---|---|---|---|---|
| (N = xx) | | | <u></u> | (N = xx) | |
| Placebo to $250 \text{ mg}$ $(N = xx)$ | Placebo to $1250 \text{mg}$ $(N = xx)$ | Placebo to $3500 \text{ mg}$ $(N = xx)$ | 250 mg $(N = xx)$ | 1250 mg $(N = xx)$ | 3500 mg $(N = xx)$ |

| BIIB054 delayed start | Е | BIIB054 early s | tart |
|-----------------------|----------|-----------------|----------|
| (N = xx) | (N = xx) | | |
| Placebo to BIIB054 | 250 mg | 1250 mg | 3500 mg |
| (N = xx) | (N = xx) | (N = xx) | (N = xx) |

#### For baseline and safety related outputs:

| BIIB054 delayed start | | | BIIB054 early start | | | | BIIB054 |
|---|---|---|---|---|---|---|---|
| (N = xx) | | | (N = xx) | | | | Total |
| Placebo Placebo to 250 to mg 1250mg $(N = xx)$ $(N = xx)$ | Placebo<br>to 3500<br>mg<br>(N = xx) | Total<br>(N=xx) | 250 mg $(N = xx)$ | 1250 mg $(N = xx)$ | 3500 mg $(N = xx)$ | Total<br>(N=xx) | (N=xx) |

For all listings the start and stop day in the listing will be computed based on the placebocontrolled baseline.

Baseline for all the analyses across the SAP

Unless otherwise specified, baseline refers to the baseline value for the placebo-controlled period and is defined as the most recent non-missing measurement collected prior to the first CONFIDENTIAL



V2.0

dose in Year 1. DBE baseline is defined as the last non-missing measurement collected prior to the first dose of the DBE period in Year 2.

For analyses on the DBE period or on the active treatment (placebo-controlled and DBE) period, DBE baseline will be used for delayed start subjects who are assigned to receiving BIIB054 in the DBE period. Change from baseline will be defined as post-baseline value minus baseline value.

#### 4.1.1 Analysis Population

- Intent-to-treat (ITT) population:
  The Intent-to-treat population is defined as all randomized subjects who received at least one dose of study treatment (BIIB054 or placebo).
- Safety population:
   The safety population is defined as all subjects who received at least one dose of study treatment (BIIB054 or placebo).
- Pharmacodynamic analysis population:
  The pharmacodynamic population is defined as a subset of the ITT population with at least 1 post-baseline pharmacodynamic measurement.
- PK analysis population:
   The PK population is defined as a subset of the ITT population who have at least 1 measurable BIIB054 concentration in serum
- Immunogenicity population:
   Immunogenicity analysis will be performed for all subjects in the safety population.

#### 4.1.2 Analyses period

Depending on the purpose, different analyses will be conducted on the following study periods:

- 1. DBE period. Only data in the DBE period will be included in these analyses. For example, incidence table of adverse events in the DBE period.
- Placebo-controlled and DBE period. All the data in the placebo-controlled and DBE periods will be included in these analyses. For example, mean plot of actual laboratory values in the placebo-controlled and DBE period.



V2.0

3. Active treatment (placebo-controlled and DBE) period (i.e., Total BIIB054 experience) period. Active treatment period is defined as the study period(s) that a subject is assigned to BIIB054. For early start subjects – subjects who are assigned to BIIB054 in both placebo-controlled and DBE period, all the data (placebo-controlled and DBE periods) will be included in the analyses. For delayed start subjects – subjects who are assigned to placebo in Year 1 and BIIB054 in the DBE period, only data in the DBE period will be included. For example, incidence table of adverse events in the active treatment (placebo-controlled and DBE) period will not include the AEs started on placebo treatment in year 1.

Subjects to be included in a certain output is determined by both the analysis population and the analysis period. For example, the incidence table of adverse events in the DBE period will include subjects in the safety population for the DBE period, i.e., all randomized subjects who received at least one dose of study treatment in the DBE period. The incidence table of adverse events in the active treatment (placebo-controlled and DBE) period will include subjects in the safety population for the active treatment period, i.e., all randomized subjects who received at least one dose of study treatment in the active treatment period. In this SAP we do not separately define the analysis population in each analysis period.

#### 4.2 Background Characteristics

The summaries in this section will be based on the ITT population. Analysis period will be specified for each table or figure. Unless otherwise specified, summary tables will be presented by DBE treatment group. Listings will include all data in the placebo-controlled and DBE periods (all data in the study), with an indicator of the study period in a column (pre-dosing, placebo-controlled, or DBE) for each record to indicate when the event occurred. Listings will be presented by DBE treatment group.

#### 4.2.1 Accounting of Subject

Disposition in the DBE period will be summarized for subjects enrolled in DBE. The summary data will include number (%) of subjects dosed in the DBE period, number (%) of subjects who completed the first year of treatment/study of DBE (i.e., year 2 of the study), number (%) of subject who discontinued treatment and/or withdrew from study in the first year of DBE (i.e., year 2 of the study), the reason for treatment discontinuation and/or study withdrawal for in the first year of DBE (i.e., year 2 of the study), number (%) of subjects who completed the treatment/study in DBE (i.e., year 2-4 of the study), and number (%) of subjects who discontinued treatment and/or withdrew from study in DBE (i.e., year 2-4 of the study), the reason for treatment discontinuation and/or study withdrawal in DBE (i.e., year 2-4 of the study).

For subject who discontinued treatment and/or withdrew from the study in the first year of DBE (i.e., year 2 of the study), days on treatment and days on study will be summarized.

For subjects who discontinued treatment and/or withdrew from study in DBE (i.e., year 2-4 of the study), days on treatment and days on study will be summarized and listed. In the listing, the subjects who discontinued treatment and/or withdrew from study in the first year




V2.0

of DBE will be flagged. Time to treatment discontinuation and time to study withdrawal in the DBE period may be displayed by Kaplan-Meier plot (presented by DBE treatment group).

Disposition in the placebo-controlled and DBE period will be also summarized in the same fashion. Number (%) of subjects dosed in the placebo-controlled period, number (%) subject who completed the placebo-controlled period, number (%) of subjects who entered the DBE period, number (%) of subjects who completed the first year of DBE period, number (%) of subjects who completed the whole study will be displayed. Number of subjects who discontinued treatment or study and reason of discontinuation will be summarized for each period and for the whole study.

#### 4.2.2 Demographics and Baseline Characteristics

Demographics, baseline characteristics, medical history and PD treatment history will be summarized for subjects enrolled in the DBE period and subjects not enrolled in the DBE period, respectively. Please refer to the SAP of placebo-controlled period for more details.

#### 4.2.3 Concomitant Medications and Non-Drug Therapies

All medications will be coded using the World Health Organization Drug (WHODrug March 2020 B3 or higher) dictionary. All non-drug therapies (defined as diagnostic procedures or medical treatment procedures) will be coded using the MedDRA dictionary version 23.0 or higher.

The number (%) of subjects taking concomitant general medication (excluding PD medications) and non-drug therapies in the DBE period will be summarized by DBE treatment group for subjects enrolled in the DBE period. In addition, number of subjects in the ITT population that have taken any concomitant medications in the active treatment (placebo-controlled and DBE) period will be summarized. Concomitant non-PD medications and non-drug therapies will be listed in the placebo-controlled and DBE treatment period. Start and stop day in the listing will be computed based on the placebo-controlled baseline.

For subjects enrolled in the DBE period, the number (%) of subjects taking any concomitant PD symptomatic medications, number of subjects taking Dopamine, MAO-B inhibitor, Dopamine Agonist at the baseline of the placebo-controlled period and at the baseline of DBE period will be summarized respectively by DBE treatment group. The placebo-controlled and DBE period data will be summarized in the same fashion. Concomitant PD symptomatic medication will be listed for all subjects in the placebo-controlled and DBE periods. Start and stop day in the listing will be computed based on the placebo-controlled baseline. Please refer to the placebo-controlled SAP for definitions of concomitant therapies and PD symptomatic medication use at baseline.

#### 4.2.4 Protocol Deviations

Protocol deviations identified during site monitoring will be captured in a Protocol Deviation log and categorized as major or minor deviations. The major protocol deviations occurred in CONFIDENTIAL



V2.0

the DBE period will be summarized for subjects enrolled in DBE. The major protocol deviations for all ITT subjects in the combined placebo-controlled and DBE periods will also be summarized. Major and minor protocol deviations for all ITT subjects will be listed, respectively, across the placebo-controlled period and the DBE period. All summaries for protocol deviations will be presented by DBE treatment group. A separate Covid-19 related protocol deviation category will be shown in the protocol deviation listings.

#### 4.2.5 Study Drug Exposure and Study Drug Compliance

A summary table of study drug exposure and compliance in the DBE period will be provided. Number of infusions of BIIB054 received will be summarized as a continuous variable as well as a categorical variable (categories as 1-5, 6-10 and 11-15, 16-20, 20-25, >=26) as well as a continuous variable. Number of weeks on study treatment, calculated as (date of last dose – date of first dose +1)/7, will be summarized as a categorical variable (categories as <0.5 years, >=0.5 years, >=1 year, >=2 years, >=3 years) as well as a continuous variable. Percentage of study treatment taken up to the last dose, calculated as (the actual number of infusions / the number of infusions a subject is expected to take until the date of last infusion)\*100, will be summarized as a continuous variable. This table will be presented by DBE treatment group. A similar table will also be provided on the active treatment (placebocontrolled and DBE) period in order to summarize the exposure data while subjects are on BIIB054.

A listing of study drug administration records, including infusion start date and time, infusion stop date and time, total volume prepared, total volume administered, location of infusion, initial infusion rate, dose interruption or rate change or not, time of interruption or rate change, infusion rate after interruption or rate change, reason for interruption or rate change will be provided for the placebo-controlled and DBE period. A listing of subjects who received the wrong treatment compared to what they were randomized to will be provided for the placebo-controlled and DBE period.

#### 4.3 Efficacy analyses

#### 4.3.1 General Consideration

The analysis population for the efficacy analyses are defined in Section 4.2.1. The analysis period includes data from both placebo-controlled and DBE period combined. That is, data from both the placebo-controlled and DBE periods will be included in the analysis.

The following three comparisons will be evaluated for the long-term efficacy analyses of BIIB054:

- The early start 250 mg compared with the pooled delayed start group;
- The early start 1250 mg compared with the pooled delayed start group;
- The early start 3500 mg compared with the pooled delayed start group

The following comparisons may also be evaluated:

• The early start 250 mg compared with the delayed start 250 mg;



V2.0

- The early start 1250 mg compared with the delayed start 1250 mg.
- The early start 3500 mg compared with the delayed start 3500 mg.

The pooled delayed start group contains all the subjects who were randomized to placebo treatment in the placebo-controlled period including those who did and who did not enter into the DBE period. There will be no multiple comparison adjustments. Data after subjects start PD symptomatic treatment will be included in the analyses, since the majority of subjects are expected to take PD medication after Week 52.

Subjects who were randomized to placebo group but accidentally received one or more doses of the active treatment during the placebo-controlled period will be classified as delayed start for all the efficacy, pharmacodynamic, and analyses.

#### Visit Windows for by visit analyses

For the by visit summaries and MMRM models, the analysis visit should be defined using visit windows (see Tables 6-16 in the Appendix). If there is more than 1 value in the same analysis visit window (>1 value for the same analysis visit) for a certain parameter for a subject, then the closest record to the target visit day will be used for the by visit analysis. If they are with the same distance from the target visit day, then the record with the later time will be used for the by visit analysis.

#### Handling of missing items for scales

Please refer to the placebo-controlled SAP for the imputation method. The same method will be applied to efficacy endpoints collected in the DBE period.

#### 4.3.2 Primary efficacy endpoint analysis

The estimand of the primary analysis for MDS-UPDRS Part I+II+III total score at Week 72 is the mean difference of the change from baseline at Week 72 between treatment groups in the ITT population regardless of whether start of PD medication had occurred or not. Specifically, the estimand takes the following into consideration:

- A. Population: ITT population as defined in Section 4.1.1;
- B. Variable: change from baseline to Week 72 in the MDS-UPDRS Part I+II+III total score:
- C. Intercurrent events: regardless of whether start of PD medication had occurred or not;
- D. Population-level summary: difference in variable means between each early start group and delayed start group

Change from baseline in the MDS-UPDRS Part I+II+III total score at Week 72 will be analyzed using an MMRM model for all the visits in the placebo-controlled and DBE period.

Data after subjects start PD medication will be included in the primary analyses.

For details on the model to be used please refer back to the Year 1 SAP, for the analyses of MDS-UPDRS including data after PD medication. Adjusted means for each treatment group, CONFIDENTIAL



V2.0

pairwise adjusted differences for the comparisons, 95% confidence intervals for the differences will be presented at each visit, and p-values will be presented for the key visits of week 24, 52, and 72. Dose-response testing will be done using the adjusted mean with the pre-specified MCP-MOD procedure with pre-specified candidate models (refer to Year 1 SAP Sample Size Consideration section). If the distribution of the outcome is highly skewed, p-value will be generated from the MMRM model based on the rank data. Missing data are assumed to be missing at random behind the MMRM model.

A multiple comparison adjustment method (graphical procedure) will be applied to control the overall type I error at 0.05 in the study, due to the primary endpoint of MDS-UPDRS total score being analyzed at Week 52 and Week 72, and superiority against placebo is considered reached in study if statistically significant result is achieved at either timepoint. Please refer to the "Interim Analysis" section for this method. Pairwise comparison of each active group versus delayed-start group(s) will also be conducted, however, no additional multiplicity adjustment will be made, and nominal p-values will be reported. The primary comparison is between each of the early-start BIIB054 dose group, with the pooled delayed-start BIIB054 group.

The following three comparisons will be evaluated for the long-term efficacy analyses of BIIB054:

- The early start 250 mg compared with the pooled delayed start group;
- The early start 1250 mg compared with the pooled delayed start group;
- The early start 3500 mg compared with the pooled delayed start group

The following comparisons may also be evaluated:

- The early start 250 mg compared with the delayed start 250 mg;
- The early start 1250 mg compared with the delayed start 1250 mg.
- The early start 3500 mg compared with the delayed start 3500 mg.

Per design, a subset of subjects will enter year 3 and 4 for a limited time. There will be some visits with too few data in year 3 and 4. If this is the case, the visits with too few data will be excluded from the MMRM analyses, Otherwise, the MMRM model will not converge. In addition, since most patients will start PD medication by year 1, most data in year 2-4 will be after PD medication. Therefore, data after subject start PD medication will be included in the MMRM analyses. Otherwise, the MMRM model will not converge.

Data at the common visits of cohort A and cohort B will be included in the by visit summary and MMRM model. Data at all visits will be listed.



V2.0

#### 4.3.3 Secondary efficacy endpoints and additional endpoints analysis

Secondary endpoints, e.g., change from baseline in the MDS-UPDRS subscores (e.g., Part I, II, or III score, Part II and III total score) will be analyzed in a similar model, but no additional multiplicity adjustment will be made or for other secondary endpoints.

#### 4.3.3.1 MDS-UPDRS based endpoints

The analysis approaches and the MMRM model described will be performed for additional MDS-UPDRS based endpoints as listed below, except that, 1) the baseline MDS-UPDRS total score term in the model will be replaced by the corresponding baseline value of MDS-UPDRS total or sub-part score being analyzed, 2) MCP-MOD dose-response may be performed, 3) no additional multiple comparison adjustment will be applied for secondary efficacy and exploratory efficacy endpoints

- MDS-UPDRS Parts I, II, III (Secondary Efficacy Endpoints),
- MDS-UPDRS Total Score (I+II+III) at the end of the study
- MDS-UPDRS Parts II+III, Ib+II+III
- MDS-UPDRS Part IV
- Postural Instability -Gait Difficulty (PIGD) score (mean score of MDS-UPDRS items 2.12+2.13+3.10+3.11+3.12),
- Lower Extremity (LE) score (mean score of MDS-UPDRS items 3.10+3.11+3.12+3.13+3.3d+3.3e+3.7a+3.7b +3.8a+3.8b+3.17c+3.17d+2.12+2.13), and Tremor score (mean score of MDS-UPDRS items 2.10+3.15a+3.15b+3.16a+3.16b+3.17a+3.17b+3.17c+3.17d+3.17e+3.18).

#### 4.3.3.2 Other clinical efficacy measures





V2.0



#### 4.4 Pharmacodynamics analyses

There are three types of imaging outcomes in the study: DaT/SPECT imaging,

Please refer to the placebo-controlled SAP for details.

The analysis population for pharmacodynamic analyses is defined in Section 3.1.1. The analysis period is placebo-controlled and DBE period combined. That is, data from both the placebo-controlled and DBE periods will be included in the analyses.

Similar analyses will be conducted for the pharmacodynamic analyses as for the clinical outcome analysis. The main comparison will be between the early and delayed-start groups. The pooled delayed start group contains all the subjects who were randomized to placebo treatment in the placebo-controlled period including those who did and who did not enter to the DBE period. There will be no multiple comparison adjustments. Data after subjects start PD symptomatic treatment will be included in the analyses.

Visit Windows for by visit analyses



V2.0

For the by visit summaries and MMRM models, the analysis visit should be defined using visit windows (see Table 3 in the Appendix). If there is more than 1 value in the same analysis visit window (>1 value for the same analysis visit) for a certain parameter for a subject, then the closest record to the target visit day will be used for the by visit analysis. If they are with the same distance from the target visit day, then the record with the later time will be used for the by visit analysis.

A prespecified set of imaging measures as well as the change from baseline will be summarized by DBE treatment groups by visit for all the visits in the placebo-controlled and DBE period.

#### MMRM model analyses:

Similar MMRM model will be used to conduct the pharmacodynamic analyses as for the clinical outcome analysis, with the same terms included in the model.

#### 4.5 Safety Analyses

#### 4.5.1 General Considerations

#### Analysis population

Safety population will be used for safety analyses of AEs, clinical laboratory data, vital sign data, ECG data, physical and neurological examination findings, Columbia Suicide Severity Rating Scale (C-SSRS) data and MRI safety data.

#### DBE safety treatment groups

Please refer to Section 3.1 for the safety treatment groups. Subjects who were randomized to placebo group but accidentally received one or more doses of BIIB054 during the placebo-controlled period will be classified as early start for all the safety analyses that involves DBE, and their applicable safety data in the placebo-controlled period will be included in the analysis for active treatment (placebo-controlled and DBE) period.

#### Safety analysis period

Analysis period will be specified for each output. Analyses periods in this SAP are

- Long-term extension period for AE analyses
- Active treatment (placebo-controlled and DBE) period for AE analyses and analyses of hematology/blood chemistry/urinalysis, hepatotoxicity, vital sign, ECG, MRI.

Safety data in the specified analysis period will be included in the analysis. Listings will include all data in the placebo-controlled and DBE period, unless otherwise specified.

#### Incidence, incidence proportion and incidence rate

• Incidence and incidence proportion will be provided in incidence tables. Incidence is defined as the number of subjects who experienced an event. Incidence proportion is CONFIDENTIAL



V2.0

defined as the number of subjects who experienced an event divided by the total number of subjects in the analysis population, i.e., percentage. Each subject will be counted only once within each category.

• Incidence and incidence rate will be provided in incidence rate tables. Incidence rate is defined as the number of subjects who experienced an event divided by the total follow-up time among the subjects in the analysis population (e.g., incidence rate per 100 subject-years). The total follow-up time is the sum of all subjects' follow-up time. The follow-up time for a subject is defined as the number of days (inclusive) from the first dose of treatment until the last day on study divided by 365.25. For active treatment (placebo-controlled and DBE) period analyses, the first dose of treatment is considered as the first dose received in the study period (PC or OLE) in which a subject first receives BIIB054. Each subject will be counted only once within each category.

#### 4.5.2 Clinical Adverse Events

Treatment emergent AEs (TEAEs)

All AEs will be coded using the MedDRA dictionary version 23.0 or higher.

All AEs will be analyzed based on the principle of treatment emergence. A treatment emergent AE is defined as an AE that started or worsened after the start of first infusion of study treatment.

To define treatment emergence for AEs with missing start or stop date or time the following additional criteria will be used:

- if both the start and stop dates for a particular AE are missing, then that AE is considered treatment emergent.
- if the start date for a particular AE is missing and the stop date/time falls after the first dose date/time, then that AE is considered treatment emergent.
- if the start date for a particular AE was the same as the first dose date, and the start time was missing, then that event is considered treatment emergent.

For AEs with a partial start date, the year/month of the event date will be compared to that of the first dosing date to determine whether the event is treatment emergent.

In addition, SAEs that occurred since a subject was screened in the study and prior to the first infusion of study treatment, which by definition are not treatment emergent, will be analyzed separately.

Only TEAEs will be included in the AE tables, unless otherwise specified. Listings of AEs will include all events, whether treatment emergent or not.

#### 4.5.2.1 Summary and incidence analysis

Overall summary of AE table will be done for the following periods, by DBE treatment groups:

• DBE period, and,



V2.0

• the active treatment (placebo-controlled and DBE) period

The following information will be summarized: the number of subjects with any AE, with any AE by maximum severity, with any related AE (related to study drug as assessed by investigator), with radioligand rated AE, with SAE, with related SAE, with radioligand rated SAE, with AE leading to study drug discontinuation, with AE leading to study withdrawal and the number of deaths.

The sorting order of AE incidence tables, unless otherwise specified, will be by decreasing frequency order of "BIIB054 total" column within each category in the tables presented by DBE treatment group. A subject is counted only once within each category in each table. For example, for the table of AEs by system organ class and preferred terms sorted by decreasing frequency presented by DBE treatment group, system organ class will be presented in decreasing frequency order of BIIB054 total column, and within each system organ class, preferred terms will be presented in decreasing frequency order of BIIB054 total column. A subject is counted only once within each system organ class and preferred term.

The severity of AEs and SAEs is graded using the CTCAE grade, version 5.0. The categorisation of severity is as follows: grade 1 (mild), 2 (moderate), 3 (severe or medically significant), 4 (life-threatening) and 5 (death), Severe AEs and SAEs are classed as CTCAE grade >=3.

The following AE incidence tables will be provided for the DBE period:

- 1. AEs by system organ class and preferred term sorted by decreasing frequency
- 2. AEs by preferred term
- 3. Severe AEs by system organ class and preferred term
- 4. Severe AEs by preferred term
- 5. Study drug related AEs by system organ class and preferred term
- 6. SAEs by system organ class and preferred term sorted by decreasing frequency
- 7. SAEs by preferred term
- 8. Study drug related SAEs by system organ class and preferred term
- 9. AEs that led to discontinuation of study treatment by system organ class and preferred term
- 10. AEs that led to withdrawal from study by system organ class and preferred term

# 4.5.2.2 Incidence and incidence rate analysis for active treatment (placebo-controlled and DBE) period

Due to the different length of active treatment (placebo-controlled and DBE) period in early start versus delayed start subjects, both incidence (proportion) tables and incidence rate tables will be used for AE analyses in this period. The entire follow-up time is from the first dose in



V2.0

active treatment period (first dose in placebo-controlled period for early start subjects and first dose in DBE period for delayed start subjects) until the last day in the study.

The following incidence (proportion) will be provided for the active treatment (placebo-controlled and DBE) period. The follow-up adjusted incidence rate table will be provided for 1, 10, 12, 14, 16 and 17.

- 1. AEs by system organ class and preferred term sorted by decreasing frequency
- 2. AEs by system organ class and preferred term sorted by alphabetical order analysis
- 3. AEs by system organ class
- 4. AEs by preferred term
- 5. AEs with an incidence of 5% or more in any treatment group by preferred term
- 6. Severe AEs by system organ class and preferred term
- 7. Severe AEs by preferred term
- 8. AEs by maximum severity by system organ class and preferred term (System organ class will be presented alphabetically. Preferred term will be presented in decreasing frequency order.
- 9. AEs by maximum severity by preferred term (Preferred term will be presented in decreasing frequency order)
- 10. Study drug related AEs by system organ class and preferred term
- 11. Radioligand related AEs by system organ class and preferred term
- 12. SAEs by system organ class and preferred term
- 13. SAEs by preferred term
- 14. Study drug related SAEs by system organ class and preferred term
- 15. Radioligand related SAEs by system organ class and preferred term
- 16. AEs that led to discontinuation of study treatment by system organ class and preferred term
- 17. AEs that led to withdrawal from study by system organ class and preferred term
- 18. AEs that occurred within 2 hours from infusion start by system organ class and preferred term

The following listings will be provided for the placebo-controlled and DBE period:

- 1. Listing of AEs
- 2. Listing of SAEs
- 3. Listing of AEs that led to discontinuation of study treatment
- 4. Listing of AEs that led to withdrawal from study
- 5. Listing of AEs that occurred within 2 hours from infusion start
- 6. Listing of study drug related AEs
- 7. Listing of radioligand related AEs

#### CONFIDENTIAL



V2.0

8. Listing of deaths

#### 4.5.3 Clinical Laboratory Data

The following laboratory assessments will be performed in Year 2-4 to evaluate the safety profile of BIIB054:

- Hematology: Complete blood count with differential and platelet count, INR, PT, and APTT
- Blood chemistry: total protein, albumin, creatinine, blood urea nitrogen, uric acid, bilirubin (total and direct), alkaline phosphatase, alanine aminotransferase, aspartate aminotransferase, gamma-glutamyl transferase, glucose, calcium, phosphorus, bicarbonate, chloride, sodium, and potassium
- Urinalysis: dipstick for blood, protein, and glucose (microscopic examination may also be performed)

#### 4.5.3.1 Quantitative analyses

For quantitative analyses, analysis period is active treatment (placebo-controlled and DBE) period. For numeric laboratory parameters, actual values will be summarized by visit for all the common visits in both Cohort A and B in the active treatment (placebo-controlled and DBE) period. Number of evaluable subjects, mean, standard deviation, median, 25% and 75% quartiles, minimum and maximum values will be presented at each visit. Plots of mean actual values (with standard error) for key numeric laboratory parameters at each visit for all the visits in the active treatment (placebo-controlled and DBE) period will be provided.

Plots of mean actual values (with standard error) for numeric laboratory parameters at each visit for all the visits in the active treatment (placebo-controlled and DBE) period may be provided.

Change from baseline and percent change from baseline for numeric laboratory parameters will be summarized in the active treatment (placebo-controlled and DBE) period. Placebo-controlled baseline will be used for early start subjects and DBE baseline will be used for delayed start subjects. Change and percent change from baseline will be calculated based on the DBE baseline for delayed start subjects. Number of evaluable subjects, mean, standard deviation, median, 25% and 75% quartiles, minimum and maximum values will be presented at each visit.

Listings of individual laboratory measurements by patients for all the parameters will be provided for placebo-controlled and DBE period.



V2.0

Visit windows for by visit summaries

For laboratory by visit summaries, the analysis visit should be defined using visit windows (see Table 1 in the Appendix). Visit windows are generally from mid-points between the visit before to the current, and the midpoint from the current visit to the next visit. If there is more than 1 value in the same analysis visit window for a certain parameter for a subject, then the closest record to the target visit day will be used for the by visit analysis. If there are 2 values in the same analysis visit window with the same distance from the target visit day for a certain parameter for a subject, then the record with the later date will be used for the by visit analysis. If there are 2 values on the same day for a certain parameter for a subject, then the record with the later time will be used for the by visit analysis.

#### 4.5.3.2 Qualitative analyses

For qualitative analyses, all available values will be included (not just the "analyzed record" within each visit window in the quantitative analyses). Analysis period is active treatment (placebo-controlled and DBE) period.

#### Shift analyses

Laboratory data will be summarized using shift tables where appropriate for the active treatment (placebo-controlled and DBE) period. Each subject's hematology, blood chemistry and urinalysis numeric values will be flagged as "low", "normal", or "high" relative to the normal ranges of the central laboratory or as "unknown" if no result is available. Each subject's urinalysis categorical values will be flagged as "positive" or "negative", or "unknown" if no value is available.

Shifts from baseline to high/low status will be presented for hematology, blood chemistry and urinalysis numeric parameters, and shifts from baseline to abnormal (positive) will be presented for urinalysis categorical parameters. Shift to low includes normal to low, high to low, and unknown to low; Shift to high includes normal to high, low to high, and unknown to high. Subjects need to have at least one post-baseline evaluation and a baseline value not low or high or positive (including missing) in order to be included in the analysis.

For early start subjects, the placebo-controlled baseline will be used and shifts that occurred in either placebo-controlled or DBE period will be included. For delayed start subjects, the DBE baseline will be used and shifts that occurred in the DBE period based on DBE baseline will be included.

Potentially Clinically Significant (PCS) laboratory abnormalities analyses

Please refer to the placebo-controlled SAP for the parameters and criteria for potentially clinically significant laboratory abnormalities analyses.

The number of subjects with potentially clinically significant laboratory abnormalities post-baseline will be summarized for the active treatment (placebo-controlled and DBE) period.



V2.0

Subjects need to have at least one post-baseline evaluation in the active treatment period in order to be included in the analysis. For early start subjects, the placebo-controlled baseline will be used and abnormalities that occurred in either placebo-controlled or DBE period will be included. For delayed start subjects, the DBE baseline will be used and PCS abnormalities that occurred in the DBE period based on DBE baseline will be included.

A listing of subjects with PCS laboratory abnormalities in the active treatment (placebo-controlled and DBE) period will also be provided, with all the data in the placebo-controlled and DBE period will be listed.

#### Potential serious hepatotoxicity

Potential serious hepatotoxicity is defined as ALT or AST > 3x ULN and total bilirubin > 2x ULN at any time post-baseline, not necessarily concurrent, in the active treatment (placebo-controlled and DBE) period. A scatterplot of the maximum post-baseline ALT or AST value relative to ULN and maximum post-baseline total bilirubin value relative to ULN (not necessarily concurrent) will be provided. In addition, a line plot of ALT, AST, ALP and total bilirubin values over time for each subject with potential serious hepatotoxicity will be provided.

A listing of subjects with potential serious hepatotoxicity in the active treatment (placebo-controlled and DBE) period will be provided with the concurrent records labeled. All the data in the placebo-controlled and DBE period will be listed. Concurrent is defined as on the same day. Subjects with ALT > 1x ULN, > 3x ULN, > 5x ULN, > 10x ULN or > 20x ULN, subjects with AST > 1x ULN, > 3x ULN, > 5x ULN, > 10x ULN or > 20x ULN, subjects with total bilirubin > 1x ULN, > 1.5x ULN or > 2x ULN, subjects with ALP > 1x ULN or > 1.5x ULN and subjects with AST or ALT > 3x ULN post-baseline accompanied by concurrently elevated total bilirubin > 1.5x ULN or > 2x ULN will be labeled.

#### 4.5.4 Vital Sign Data

For vital sign data analyses, the analysis period is active treatment (placebo-controlled and DBE) period. Vital sign parameters include body temperature, systolic blood pressure, diastolic blood pressure, heart rate, respiration rate and weight. Vital signs will be measured with the subject supine and after the subject has been resting for at least 10 minutes. The descriptive statistics for actual values will be summarized at each visit in the active treatment (placebo-controlled and DBE) period. Plot of mean vital sign values in the active treatment (placebo-controlled and DBE period) may be provided.

Summary of change from baseline including number of evaluable subjects, mean, standard deviation, median, 25% and 75% quartiles, minimum, and maximum values will be summarized at each visit in the active treatment (placebo-controlled and DBE) period. Placebo-controlled baseline will be used for early start subjects and DBE baseline will be used for delayed start analysis.

The analysis of vital signs will also focus on the incidence of clinically relevant abnormalities at any post-baseline visit in the active treatment (placebo-controlled and DBE) period. Please refer to the placebo-controlled SAP for the criteria to assess potential clinically relevant abnormalities in vital sign. The incidence and percentage of clinically relevant abnormalities



V2.0

determined by each criterion will be summarized in the active treatment (placebo-controlled and DBE) period.

A listing of subjects with clinically relevant abnormalities at any post-baseline visit in the active treatment (placebo-controlled and DBE) period will also be provided. All the data in the placebo-controlled and DBE period will be listed.

Visit windows for by visit summaries

For vital sign by visit summaries, the analysis visit should be defined using windows (see Table 2 in the Appendix). For the same parameter for a subject, if there is more than 1 record in the same analysis visit window, then select the record closest to the target visit day. If there are 2 records in the same analysis visit window with the same distance from the target visit day, then select the record with the later date.

#### **4.5.5** ECG Data

For ECG data analyses, the analysis period is active treatment (placebo-controlled and DBE) period. The descriptive statistics for actual values will be summarized at each visit in the active treatment (placebo-controlled and DBE) period. Plot of mean ECG values in the active treatment (placebo-controlled and DBE) period may be provided.

Shift from normal or unknown ECG at baseline to abnormal post-baseline ECG, will be summarized in the active treatment (placebo-controlled and DBE) group. The number of subjects with potential QTcF interval outlier post-baseline will also be summarized in the active treatment (placebo-controlled and DBE) period. The criteria of defining QTcF interval outliers is specified in the placebo-controlled SAP. For early start subjects, the placebo-controlled baseline will be used. For delayed start subjects, the DBE baseline will be used.

A listing of subjects with abnormal ECG status post-baseline in the active treatment (placebo-controlled and DBE) period will be provided. All data in the placebo-controlled and DBE period will be listed.

#### 4.5.6 Physical and Neurological Examination

Abnormal findings during physical and neurological examinations are captured as adverse events and will be reflected in the summary of AEs.

#### 4.5.7 C-SSRS Data

The Columbia Suicide Severity Rating Scale (C-SSRS) is an assessment that evaluates suicidal ideation and behavior. There are 5 "Yes/No" questions on suicidal ideation following the increasing severity order: (1) Wish to be dead, (2) Non-specific active suicidal thoughts, (3) Active suicidal ideation with any methods (not plan) without intent to act, (4) Active suicidal ideation with some intent to act, without specific plan, (5) Active suicidal ideation with specific plan and intent, and 6 "Yes/No" questions on suicidal behavior



V2.0

following the increasing severity order: (6) Preparatory acts or behavior, (7) Aborted attempt, (8) Interrupted attempt, (9) Actual attempt, (10) Suicidal behavior, (11) Suicide (only at post-baseline visits). Another "Yes/No" question of whether the subject has engaged in non-suicidal self-injurious behavior is also collected.

The summary table for C-SSRS will be conducted for the active treatment (placebo-controlled and DBE) period. Number of subjects who answered "Yes" to each of the 11 questions post-baseline, subjects who answered "Yes" to at least one question for suicidal ideation, subjects who answered "Yes" to at least one question for suicidal behavior, and subjects who have engaged in non-suicidal self-injurious behavior will be presented.

A listing of subjects with any suicidal ideation or behavior at baseline or post-baseline will be provided for the placebo-controlled and DBE period.

#### 4.5.8 MRI Safety Data

Brain MRI safety finding are assessed at Screening visit, Week 24, 52, 96, 148 and 4 weeks after last dose/ET visits.

The MRI safety result is classified as normal or abnormal. Shift table from normal or unknown MRI at baseline to abnormal post-baseline MRI will be summarized in the active treatment (placebo-controlled and DBE) period. The worst post-baseline record of each subject is selected. A listing of details for abnormal brain MRI findings will be presented for placebo-controlled and DBE period.

#### 4.6 Pharmacodynamic - Imaging analysis

#### 4.6.1 General Consideration

There are three types of imaging outcomes in the study: DaT/SPECT imaging, Neuromelanin MRI imaging and Structural MRI imaging. Please refer to the placebo-controlled SAP for details.

The analysis population for pharmacodynamic analysis is defined in Section 3.1.1. The analysis period is placebo-controlled and DBE period. That is, data from both the placebo-controlled and DBE periods will be included in the analysis. All pharmacodynamic analyses will be presented by DBE treatment group.

The following three comparisons will be evaluated for the long-term pharmacodynamic analyses of BIIB054:

- The early start 250 mg compared with the delayed start 250 mg;
- The early start 1250 mg compared with the delayed start 1250 mg.
- The early start 3500 mg compared with the delayed start 3500 mg.

The following comparisons may also be evaluated:

• The early start 250 mg compared with the pooled delayed start group;



V2.0

- The early start 1250 mg compared with the pooled delayed start group;
- The early start 3500 mg compared with the pooled delayed start group

The pooled delayed start group contains all the subjects who were randomized to placebo treatment in the placebo-controlled period including those who did and who did not enter to the DBE period. There will be no multiple comparison adjustments. Data after subjects start PD symptomatic treatment will be included in the analyses.

#### Visit Windows for by visit analyses

For the by visit summaries and MMRM models, the analysis visit should be defined using visit windows (see Table 3 in the Appendix). If there is more than 1 value in the same analysis visit window (>1 value for the same analysis visit) for a certain parameter for a subject, then the closest record to the target visit day will be used for the by visit analysis. If they are with the same distance from the target visit day, then the record with the later time will be used for the by visit analysis.

#### 4.6.2 By Visit Summary and MMRM Model

A prespecified set of imaging measures as well as the change from baseline will be summarized by DBE treatment groups by visit for all the visits in the placebo-controlled and DBE period.

Change or percent change from baseline in the imaging measures will be analyzed using an MMRM model for all the visits in the placebo-controlled and DBE period. For details of the model to be used please see the 1 year SAP. Adjusted means for each treatment group, pairwise adjusted differences for the comparisons, 95% confidence intervals for the differences will be presented at each visit, and p-values will be presented for the key visits of week 24, 52, 96 and 148. If the distribution of the outcome is highly skewed, p-value will be generated from the MMRM model based on the rank data. Missing data are assumed to be missing at random behind the MMRM model.

Per design, a subset of subjects will enter year 3 and 4 for a limited time. There will be some visits with too few data in year 3 and 4. If this is the case, the visits with too few data will be excluded from the MMRM analyses, Otherwise, the MMRM model will not converge. In addition, since most patients will start PD medication by year 1, most data in year 2-4 will be after PD medication. Therefore, data after subject start PD medication will be included in the MMRM analyses. Otherwise, the MMRM model will not converge.

Data at the common visits of cohort A and cohort B will be included in the by visit summary and MMRM model. Data at all visits will be listed.

#### 4.6.3 Additional analyses of placebo-controlled period due to COVID-19

Due to COVID-19 public health emergency, considerations were made to allow week 52 assessments to be delayed up to 4 weeks. If this occurs, some of the data may not be included in the all patient week 52 analyses, as they may miss the timeline of the corresponding CONFIDENTIAL



V2.0

interim database lock. However, these data are still considered in the placebo-controlled period because they are before the first dose of DBE period. Depending how much data are missing in the all patient week 52 analyses database lock, the MMRM analyses in the placebo-controlled period may be repeated by including all the available data in the placebo-controlled period.



#### 4.8 Pharmacokinetics Analysis

Per protocol, sparse PK data are collected in the DBE period. Therefore, the PK analyses will be focused on summarizing the PK concentration over time. The PK analysis population as defined in Section 3.1.1 and data from both placebo-controlled and DBE periods will be included. All the PK analyses will be presented by DBE treatment group. In addition, an exposure-response (ER) analysis from both placebo-controlled and DBE periods will be conducted, to detect any ER relationship trend and potential covariate using any primary or secondary endpoint and BIIB054 exposure metrics as deemed appropriate. Other tables and figures based on the population PK and ER analyses will be generated by Clinical Pharmacology and Pharmacometrics (CPP) team and will be included in a separate report from CPP.

#### 4.9 Immunogenicity Analysis

#### 4.9.1 Analysis population

All immunogenicity data will be analyzed based on the immunogenicity population, which is same as the safety population as defined in Section 3.1.1.



V2.0

#### 4.9.2 Method of analysis

A summary table of subjects with treatment-emergent positive anti-BIB054 antibody responses in the placebo-controlled and DBE active treatment period will be displayed by DBE treatment group and by visit. Please refer to the placebo-controlled SAP for the definition of treatment-emergent positive anti-BIB054 antibody responses. In this summary, DBE baseline will be used for delayed start subjects who are assigned to receiving BIB054 in the DBE period. A listing of immunogenicity data in the placebo-controlled and DBE period for subjects with anti-BIB054 antibody positive responses will be provided.

#### Visit Windows for by visit analyses

For immunogenicity by visit summaries, the analysis visit should be defined using visit windows (see Table 12 in the Appendix). If there is more than 1 value in the same analysis visit window for a subject, then the closest record to the target visit day will be used for the by visit analysis. If there are 2 values in the same analysis visit window with the same distance from the target visit day for a certain parameter for a subject, then the record with the later date will be used for the by visit analysis. If there are 2 values on the same day for a certain parameter for a subject, then the record with the later time will be used for the by visit analysis.

#### 4.10 Interim Analyses

Safety and PK data only will be reviewed by the IDMC after subjects in Cohort A have completed Week 12 Visit assessments, and before dosing any subjects in Cohort B.

After subjects in Cohort A complete the Week 24 Visit, all available serum PK, and biomarker data (specifically the α-syn levels and complex formation data, if available) from Cohort A will be analyzed by a statistical/PK team independent of the study. The grouped level summary statistics will be reviewed only by a limited number of individuals at Biogen who are not involved in the management of the subjects or subject-level data for the study. No changes to the study design are expected based on this review.

For the purpose of planning for future studies, an administrative interim analysis may be

For the purpose of planning for future studies, an administrative interim analysis may be performed when approximately 60% of the subjects have completed the Week 52 Visit. A small unblinded team from Biogen, separate from the study management team, will have access to the unblinded interim analysis results. As of the finalization of protocol Version 8 and all subjects have completed Week 52 visits, this analyses was not conducted.

A full analysis of the 1-year data will be performed after all subjects have completed the Week 52 Visit. A small unblinded team from Biogen, separate from the study management team, will have access to the unblinded 1-year analysis results.

An interim analysis when all subjects have completed the Week 72 Visit is planned to be conducted. A small unblinded team from Biogen, separate from the study management team, will have access to the unblinded interim analysis results. All efficacy endpoints will be analyzed at the Week 72 analyses. Selected key safety data (e.g. summary of AE and SAE, summary of MRI safety findings and incidence of anti-drug antibodies) will be summarized, as this is only a snapshort of the safety profile at the time of CONFIDENTIAL



V2.0

the Week 72 interim analysis, and the comprehensive safety profile will be presented at the End of Study

A multiple comparison adjustment method will be applied to control the overall type I error at 0.05 in the study, due to the primary endpoint of change from baseline in MDS-UPDRS total score being analyzed at Week 52 and Week 72, and superiority against placebo is considered reached in the study if statistically significant result is achieved at either timepoint at the respective adjusted alpha-level.

A graphical procedure will be used to control the overall type I error at 0.05 level due to multiple-testing. An alpha of 0.04 will be allocated to the Week 52 primary endpoint analyses and an alpha of 0.01 will be allocated to the Week 72 primary endpoint analysis.

- If the Week 52 analysis is statistically significant at the 0.04 level (i.e. p-value ≤ 0.04), the alpha of 0.04 will be transferred (recycled) to the Week 72 analysis, and Week 72 will have alpha=0.05.
- If the Week 52 analysis is not statistically significant at the 0.04 level, alpha of 0.01 will be used for the Week 72 analysis. Statistically significance is considered achieved if the p-value is ≤0.01 at Week 72.
- If statistical significance is achieved at the Week 72, in either scenarios above, then the alpha of 0.01 will be transferred (recycled) back to Week 52, and the Week 52 primary analysis will be re-evaluated for statistically signifiance at the 0.05 level. This will only change the conclusion of the Week 52 results if the initial p-value is greater than 0.04 and ≤0.05.

No additional multiplicity adjustments will be made for secondary or exploratory endpoint analyses.

A blinded sample size re-estimation may be conducted when approximately 10% of subjects have completed the Week 52 Visit or approximately 1 month before enrollment is projected to be completed, whichever is earlier. The study sample size may be increased based on this blinded data review. There may be small adjustments to the percentage depending on actual enrollment rate. As of the finalization of protocol Version 8 and all subjects have completed Week 52 visits, this analyses was not conducted.

#### 5 Assessment of the impact of Covid-19 on statistical analyses

As this study is on-going when the Covid-19 public health emergency (PHE) occurred, subject visits and data collection were impacted, including missing visits, delayed visits, missed assessments and/or some visits were performed via remote assessments, e.g. telephone/video visits. Every effort was made to document these impacted study activities systematically on the eCRF and other electronic source data.



V2.0

A complete listing of all visits impacted (e.g. missed visits, delayed or assessment done via remote visits) will be listed in the clinical study report. Missing data due to Covid-19 is considered as missing at random.

#### Impact of COVID-19 on the clinical outcome analyses

In addition, subgroup analyses of the selected key clinical outcome MDS-UPDRS will be performed on a subset of subjects who did not have >=3 consecutive missing doses throughout the study to further evaluate the impact of Covid-19 on the study. The same MMRM model for the primary analyses will be used for the subgroup analyses.

In addition, due to Covid-19, some visits were delayed. A few subjects will have their Week 52 imaging done at later visits up to Week 72 and these will still be considered as Week 52 visit data in the analyses for Week 52. These data were not included in the Week 52 database lock in time, but will be included in the Week 72 database, and the related Week 52 imaging analyses will be updated at the time of the Week 72 interim analyses.

#### Impact of COVID-19 on the safety analyses

During the COVID-19 pandemic period, subjects may be prone to a high risk of getting depressed or anxiety. As a result, the analyses below will be performed to evaluate the impact of the COVID-19 pandemic on the safety analyses.

- 1. An overall summary of AE in DBE period based on data after March 7<sup>th</sup>, 2020, the start date when subjects in SPARK get impacted by COVID-19
- 2. An overall summary of AE in the active treatment (placebo-controlled and DBE) period based on data after March 7<sup>th</sup>, 2020, the start date when subjects in SPARK get impacted by COVID-19
- 3. AEs by system organ class and preferred term sorted by decreasing frequency in DBE period based on data after March 7<sup>th</sup>, 2020, the start date when subjects in SPARK get impacted by COVID-19
- 4. AEs by system organ class and preferred term sorted by decreasing frequency in active treatment (placebo-controlled and DBE) period based on data after March 7<sup>th</sup>, 2020, the start date when subjects in SPARK get impacted by COVID-19
- 5. C-SSRS data summary based on data after March 7<sup>th</sup>, 2020, the start date when subjects in SPARK get impacted by COVID-19

#### **Certificate Of Completion**

Envelope Id: ECF3A588273348DCBA7D0E61E7899330

Subject: Please DocuSign: 228PD201\_SAP\_DBE\_final\_v2.0\_clean\_23June2021.docx

Vendor Name: Source Envelope:

Document Pages: 41 Certificate Pages: 5

AutoNav: Enabled

**Envelopeld Stamping: Enabled** 

Time Zone: (UTC-05:00) Eastern Time (US & Canada)

Status: Completed

**Envelope Originator:** 



#### Record Tracking

Status: Original

6/23/2021 1:48:56 PM

Location: DocuSign

#### Signer Events

Biogen

Security Level: Email, Account Authentication

(None)

#### Signature

Signatures: 5

Initials: 0



Signature Adoption: Pre-selected Style Using IP Address:

#### **Timestamp**

Sent: 6/23/2021 1:51:14 PM Viewed: 6/23/2021 2:42:37 PM Signed: 6/23/2021 2:42:55 PM

#### **Electronic Record and Signature Disclosure:**

Not Offered via DocuSign



Biogen

Security Level: Email, Account Authentication (None)

Signature Adoption: Pre-selected Style Using IP Address:

Sent: 6/23/2021 1:51:14 PM Viewed: 6/23/2021 2:05:35 PM Signed: 6/23/2021 2:05:49 PM

#### **Electronic Record and Signature Disclosure:**

Not Offered via DocuSign



Security Level: Email, Account Authentication (None)



Signature Adoption: Pre-selected Style Using IP Address:

Sent: 6/23/2021 1:51:15 PM Viewed: 6/23/2021 2:08:11 PM Signed: 6/23/2021 2:08:17 PM

#### **Electronic Record and Signature Disclosure:**

Accepted: 6/23/2021 2:08:11 PM

ID: 520189fa-b9b6-4e49-9c27-538c44833496



Biogen

Security Level: Email, Account Authentication (None)

**Electronic Record and Signature Disclosure:** 

Not Offered via DocuSign



Signature Adoption: Pre-selected Style Using IP Address:

Sent: 6/23/2021 1:51:14 PM Viewed: 6/23/2021 2:54:33 PM Signed: 6/23/2021 2:54:52 PM

### Signer Events

Biogen

Security Level: Email, Account Authentication

#### Signature



Signature Adoption: Pre-selected Style Using IP Address:

#### **Timestamp**

Sent: 6/23/2021 1:51:14 PM Viewed: 6/23/2021 1:51:32 PM Signed: 6/23/2021 1:51:42 PM

# Electronic Record and Signature Disclosure: Not Offered via DocuSign

| In Person Signer Events | Signature | Timestamp |
|---|---|---|
| Editor Delivery Events | Status | Timestamp |
| Agent Delivery Events | Status | Timestamp |
| Intermediary Delivery Events | Status | Timestamp |
| Certified Delivery Events | Status | Timestamp |
| Carbon Copy Events | Status | Timestamp |
| Witness Events | Signature | Timestamp |
| Notary Events | Signature | Timestamp |
| Envelope Summary Events | Status | Timestamps |
| Envelope Sent Certified Delivered Signing Complete Completed | Hashed/Encrypted Security Checked Security Checked Security Checked | 6/23/2021 1:51:15 PM<br>6/23/2021 1:51:32 PM<br>6/23/2021 1:51:42 PM<br>6/23/2021 2:54:52 PM |
| Payment Events | Status | Timestamps |
| Electronic Record and Signature Disclosure | | |

#### ELECTRONIC RECORD AND SIGNATURE DISCLOSURE

From time to time, Biogen (we, us or Company) may be required by law to provide to you certain written notices or disclosures. Described below are the terms and conditions for providing to you such notices and disclosures electronically through your DocuSign, Inc. (DocuSign) Express user account. Please read the information below carefully and thoroughly, and if you can access this information electronically to your satisfaction and agree to these terms and conditions, please confirm your agreement by clicking the 'I agree' button at the bottom of this document.

#### Getting paper copies

At any time, you may request from us a paper copy of any record provided or made available electronically to you by us. For such copies, as long as you are an authorized user of the DocuSign system you will have the ability to download and print any documents we send to you through your DocuSign user account for a limited period of time (usually 30 days) after such documents are first sent to you. After such time, if you wish for us to send you paper copies of any such documents from our office to you, you will be charged a \$0.00 per-page fee. You may request delivery of such paper copies from us by following the procedure described below.

#### Withdrawing your consent

If you decide to receive notices and disclosures from us electronically, you may at any time change your mind and tell us that thereafter you want to receive required notices and disclosures only in paper format. How you must inform us of your decision to receive future notices and disclosure in paper format and withdraw your consent to receive notices and disclosures electronically is described below.

### Consequences of changing your mind

If you elect to receive required notices and disclosures only in paper format, it will slow the speed at which we can complete certain steps in transactions with you and delivering services to you because we will need first to send the required notices or disclosures to you in paper format, and then wait until we receive back from you your acknowledgment of your receipt of such paper notices or disclosures. To indicate to us that you are changing your mind, you must withdraw your consent using the DocuSign 'Withdraw Consent' form on the signing page of your DocuSign account. This will indicate to us that you have withdrawn your consent to receive required notices and disclosures electronically from us and you will no longer be able to use your DocuSign Express user account to receive required notices and consents electronically from us or to sign electronically documents from us.

#### All notices and disclosures will be sent to you electronically

Unless you tell us otherwise in accordance with the procedures described herein, we will provide electronically to you through your DocuSign user account all required notices, disclosures, authorizations, acknowledgements, and other documents that are required to be provided or made available to you during the course of our relationship with you. To reduce the chance of you inadvertently not receiving any notice or disclosure, we prefer to provide all of the required notices and disclosures to you by the same method and to the same address that you have given us. Thus, you can receive all the disclosures and notices electronically or in paper format through the paper mail delivery system. If you do not agree with this process, please let us know as described below. Please also see the paragraph immediately above that describes the consequences of your electing not to receive delivery of the notices and disclosures electronically from us.

#### How to contact Biogen:

You may contact us to let us know of your changes as to how we may contact you electronically, to request paper copies of certain information from us, and to withdraw your prior consent to receive notices and disclosures electronically as follows:

To contact us by email send messages to: DL-eSignature@biogen.com

#### To advise Biogen of your new e-mail address

To let us know of a change in your e-mail address where we should send notices and disclosures electronically to you, you must send an email message to us at DL-eSignature@biogen.com and in the body of such request you must state: your previous e-mail address, your new e-mail address. We do not require any other information from you to change your email address.. In addition, you must notify DocuSign, Inc to arrange for your new email address to be reflected in your DocuSign account by following the process for changing e-mail in DocuSign.

#### To request paper copies from Biogen

To request delivery from us of paper copies of the notices and disclosures previously provided by us to you electronically, you must send us an e-mail to DL-eSignature@biogen.com and in the body of such request you must state your e-mail address, full name, Postal address, and telephone number. We will bill you for any fees at that time, if any.

#### To withdraw your consent with Biogen

To inform us that you no longer want to receive future notices and disclosures in electronic format you may:

i. decline to sign a document from within your DocuSign account, and on the subsequent page, select the check-box indicating you wish to withdraw your consent, or you may; ii. send us an e-mail to DL-eSignature@biogen.com and in the body of such request you must state your e-mail, full name, IS Postal Address, telephone number, and account number. We do not need any other information from you to withdraw consent.. The consequences of your withdrawing consent for online documents will be that transactions may take a longer time to process..

#### Required hardware and software

| Operating Systems: | Windows2000? or WindowsXP? |
|---|---|
| Browsers (for SENDERS): | Internet Explorer 6.0? or above |
| Browsers (for SIGNERS): | Internet Explorer 6.0?, Mozilla FireFox 1.0, |
| | NetScape 7.2 (or above) |
| Email: | Access to a valid email account |
| Screen Resolution: | 800 x 600 minimum |
| Enabled Security Settings: | •Allow per session cookies |
| | •Users accessing the internet behind a Proxy<br>Server must enable HTTP 1.1 settings via<br>proxy connection |

<sup>\*\*</sup> These minimum requirements are subject to change. If these requirements change, we will provide you with an email message at the email address we have on file for you at that time providing you with the revised hardware and software requirements, at which time you will have the right to withdraw your consent.

#### Acknowledging your access and consent to receive materials electronically

To confirm to us that you can access this information electronically, which will be similar to other electronic notices and disclosures that we will provide to you, please verify that you were able to read this electronic disclosure and that you also were able to print on paper or electronically save this page for your future reference and access or that you were able to e-mail this disclosure and consent to an address where you will be able to print on paper or save it for your future reference and access. Further, if you consent to receiving notices and disclosures exclusively in electronic format on the terms and conditions described above, please let us know by clicking the 'I agree' button below.

By checking the 'I Agree' box, I confirm that:

- I can access and read this Electronic CONSENT TO ELECTRONIC RECEIPT OF ELECTRONIC RECORD AND SIGNATURE DISCLOSURES document; and
- I can print on paper the disclosure or save or send the disclosure to a place where I can print it, for future reference and access; and
- Until or unless I notify Biogen as described above, I consent to receive from exclusively through electronic means all notices, disclosures, authorizations, acknowledgements, and other documents that are required to be provided or made available to me by Biogen during the course of my relationship with you.